QSC207031(MMV\_MMV367\_21\_01) - Reporting and Amalysis Plant Sciences

#### **Quotient Confidential**

Doc No: DOC-101489 Version: 2.0 Status: Ready for Approval

Doc Name: QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan

Project Number: 207031

## REPORTING AND ANALYSIS PLAN

A First-in-Human, Single-Centre, Single Ascending Dose, Multiple Dose and Pilot Food Effect Study to Assess the Safety, Tolerability and Pharmacokinetics of MMV367 in Healthy Participants

Quotient Study Number: QSC207031

Sponsor Study Number: MMV\_MMV367\_21\_01

**Sponsor:** Medicines for Malaria Venture

ICC - Block 3, 3rd Floor 20 Route de Pré-Bois

PO Box 1826 1215 Geneva 15

Switzerland

**Date of RAP:** 15 Dec 2022

Status of RAP: Final v2.0

**Document Version History** 

| Version<br>Number | Reason for Update | Updated By: | Date |
|---|---|---|---|
| v1.0 | Initial version | Claire Wilson | 11 Jul 2022 |
| v2.0 | Amended to include protocol v3.0 updates | Claire Wilson | 15 Dec 2022 |


This Reporting and Analysis Plan may not be reproduced or communicated to a third party without the written permission of Medicines for Malaria Venture (MMV).


Author

Medical Director (MMV)

See electronic signature at end of document 19 Dec 2022 Claire Wilson Date Lead Statistician (Quotient) **Approvers** See electronic signature at end of document 19 Dec 2022 **Ewan Thomson** Date Lead Statistical Programmer (Quotient) See electronic signature at end of document 19 Dec 2022 Tom Dove Date Lead Pharmacokineticist (Quotient) See electronic signature at end of document 19 Dec 2022 Gemma Bell Date Lead Medical Writer (Quotient) See electronic signature at end of document 19 Dec 2022 Nand Singh Date Principal Investigator (Quotient) 15 DEC 2022 Denis Gossen Clinical Scientist Consultant (MMV) Stephan Chalon 19 Dec 2022 Stephan Chalon Date

Number: DOC-101489 Version: 2.0 Status: Approved Approved Date: 19 Dec 2022 QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


# I Table of Contents

| 1 | | Table of Contents | 3 |
|---|---|---|---|
| 2 | | List of Abbreviations | 6 |
| 3 | | Introduction | 9 |
| 3.1 | | Responsibilities | 9 |
| 3.2 | | Definitions | 9 |
| | 3.2.1<br>3.2.2<br>3.2.3 | Subject Definitions Definition of Treatments Definition of Visits | 10 |
| 4 | | Objectives and Endpoints | 11 |
| 5 | | Study Design | 12 |
| 5.1 | | Brief Description | 12 |
| 5.2 | 5.1.1<br>5.1.2<br>5.1.3 | Part 1 – Single Ascending Dose Cohorts Part 2 – Food Effect Cohort Part 3 – Multiple Dose Cohort(s) Criteria for In-Study Decisions | 13 |
| 5.3 | 5.2.1<br>5.2.2 | Decision Points | 15 |
| 5.4 | | Randomisation (including Replacement Subjects) | 17 |
| 5.5 | 5.4.1 | Participant Numbers | |
| 5.6 | | Unblinding procedures | |
| 5.7 | | Maintaining the Blind During Interim PK Analyses | |
| 6 | | Populations and Analysis Sets | 20 |
| 6.1 | | Safety Population and Safety Analysis Set | 20 |
| 6.2 | | Taste Population and Taste Analysis Set | 20 |
| 6.3 | | Pharmacokinetic Population and Pharmacokinetic Analysis | Set(s)21 |
| 7 | | Participant Disposition, Demographics and Baseline Cha 22 | racteristics |
| 7.1 | | Screening Failures | 22 |
| 7.2 | | Participant Disposition and Withdrawals | 22 |
| 7.3 | | Analysis Populations | 22 |
| 7.4 | | Analysis Sets and Subsets | 23 |
| 7.5 | | Demographic Characteristics and Lifestyle Details | 23 |
| 7.6 | | Medical History | 23 |

Number: DOC-101489 Version: 2.0 Status: Approved Approved Date: 19 Dec 2022 QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


| 7.7 | | Prior and Concomitant Medication | 23 |
|---|---|---|---|
| 7.8 | | Other Baseline Characteristics | 24 |
| 8 | | Efficacy | 24 |
| 9 | | Pharmacokinetics | 24 |
| 9.1 | | Plasma PK Parameter Estimation | 24 |
| | 9.1.1 | Definition of Plasma PK Parameters | 24 |
| 0.2 | 9.1.2<br>9.1.3 | Rules for Plasma PK Parameter Estimation using WinNonlin Plasma PK Parameter Reporting Specifications Urine PK Parameter Estimation | 28 |
| 9.2 | 0.0.4 | Definition of Urine PK Parameters | |
| 9.3 | 9.2.1 | Concentration and PK Parameter Summary Tables | |
| 9.4 | | Concentration and PK Figures | 31 |
| 9.5 | | Concentration and PK Listings | 32 |
| 9.6 | | Statistical Analysis of PK Parameters | 32 |
| | 9.6.1<br>9.6.2 | Part 1 and Part 3: Assessment of Dose Proportionality Part 2: Assessment of Food Effect | |
| 9.7 | 9.6.3 | Statistical Figures for Analysis of Pharmacokinetic Data Interim Pharmacokinetic Analysis | 35 |
| 10 | | Taste Assessment | 36 |
| 10.1 | | Summary Tables for Taste Questionnaire Assessments | 36 |
| 10.2 | | Listings for Taste Questionnaire Assessments | 36 |
| 10.3 | | Statistical Figures for Analysis of Taste Questionnaire Data | 36 |
| 11 | | Safety Assessments | 36 |
| 11.1 | | Extent of Exposure and Treatment Compliance | 36 |
| 11.2 | | Meal Details | |
| 11.3 | | Adverse Events | 37 |
| | 11.3.1 | Summary Tables for Adverse Events | |
| | | Listings for Adverse Events | 40 |
| 11.4 | | Laboratory Evaluations | |
| | 11.4.1 | Summary Tables for Laboratory Evaluations | |
| 11.5 | 11.4.2 | Listings for Laboratory Evaluations | |
| | 11.5.1 | Summary Tables for Vital Signs | |
| | 11.5.2 | Listings for Vital Signs | 42 |
| 11.6 | | ECGs. | |
| | 11.6.1<br>11.6.2 | Summary Tables for ECGs | |
| 11.7 | 11.0.2 | Body Weight | |
| 11.8 | | Physical Examination | |
| | | · | |

01489 Version: 2.0 Status: Approved Approved Date: 19 Dec 2022 QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan Number: DOC-101489


| 12 | Interim Statistical Analyses | 45 |
|---|---|---|
| 13 | Changes in the Conduct of the Study or Planned Analysis | 45 |
| 13.1 | Changes in the Conduct of the Study | 45 |
| 13.2 | Changes to the Planned Analyses | 45 |
| 13.3 | Any Other Relevant Changes | 45 |
| 14 | Overall Considerations | 45 |
| 14.1 | Statistical Programming and Analysis | 45 |
| 14.2<br>Statistical Ana | Quality Control of Summary Tables, Figures and Listings lysis | |
| 14.2.1 | Quality Control - Summary Tables | |
| 14.2.2<br>14.2.3 | Quality Control - Figures | |
| 14.2.4 | Quality Control - Data Listings | |
| 15 | SAS Data Transfer | 48 |
| 16 | Programming Conventions | 49 |
| 17 | Reference List | 49 |
| 18 | Index of Tables | 50 |
| 19 | Index of Figures | 58 |
| 20 | Index of Listings | 62 |
| 21 | Mock Tables | 73 |
| Appendix 1 | Schedule of Assessments: Part 1 (Cohorts 1A to 1E) | 115 |
| Appendix 2 | Schedule of Assessments: Part 2 | 117 |
| Appendix 3 | Schedule of Assessments: Part 3 (Cohorts 3A to 3C) | 119 |
| Appendix 4 Pa<br>(Days 1 to 7) | art 1 (All Cohorts) Safety and Pharmacokinetic Assessment Time Po<br>121 | oints |
| Appendix 5 to 14) | Part 2 Safety and Pharmacokinetic Assessment Time Points (Da 122 | ys 1 |
| Appendix 6 to 9) | Part 3 Safety and Pharmacokinetic Assessment Time Points (Da 124 | ys 1 |
| Appendix 7 | Example Taste/Palatability Questionnaire | 127 |

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


## 2 List of Abbreviations

ADaM analysis data model

AE adverse event

ATC anatomical therapeutic chemical

AUC area under the curve

BLQ below the limit of quantification

BMI body mass index

BP blood pressure

CDISC Clinical Data Interchange Standards Consortium

CHMP Committee for Medicinal Products for Human Use

CI confidence interval

COVID-19 Coronavirus disease 2019

CS clinically significant

CSR clinical study report

CV% coefficient of variation

D 'substantial' decrease from baseline for vital signs parameters

DP decimal place

ECG electrocardiogram

eCRF electronic case report form

F absolute bioavailability

Frel relative bioavailability

GMR geometric mean ratio

h hour

Ī

H flag used for value that is above normal reference range

HR heart rate

'substantial' increase from baseline for vital signs parameters /

increase in QTcF interval from baseline

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


ICH International Council for Harmonisation

IMP investigational medicinal product

ISF Investigator Site File

L flag used for value that is below normal reference range

LLOQ lower limit of quantification

LOCF last observation carried forward

Max maximum

MedDRA Medical Dictionary for Regulatory Activities

Min minimum

MPR metabolite to parent ratio

n number of subjects with an observation

N number of subjects in the dataset

NA not applicable

NC not calculated

NR not reportable/no result

NS no sample

PI principal investigator

PK pharmacokinetic

PT preferred term

QC quality control

QTcB QT interval corrected for heart rate using Bazett's correction

QTcF QT interval corrected for heart rate using Fridericia's correction

RAP reporting and analysis plan

SAC safety advisory committee

SAE serious adverse event

Check validity before use

Number: DOC-101489 Version: 2.0 Status: Approved Approved Date: 19 Dec 2022 QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


SD standard deviation

SDTM study data tabulation model

SF significant figure

SI substantial increase in QTcF interval from baseline

SOC system organ class

SOP standard operating procedure

TEAE treatment-emergent adverse event

TFL tables, figures and data listings

WHO World Health Organisation

Abbreviations used for pharmacokinetic parameters and associated flags are defined in Section 9.1.1, and Section 9.1.3 respectively.

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


#### 3 Introduction

This document details the following for Quotient Sciences (Quotient) Study QSC207031 (MMV\_MMV367\_21\_01):

- Criteria to be used for the definition of the populations and analysis sets relating to safety, taste and pharmacokinetic (PK) data
- · Handling of missing data
- Proposed tables, figures and data listings (TFLs) for demographic, dosing, safety and PK data
- Methods for PK parameter estimation and the formal statistical analysis

This document has been compiled according to the Quotient standard operating procedure (SOP) "Production of Reporting and Analysis Plans" and has been written based on information contained in the final study protocol (v3.0) dated 08 Sep 2022.

The v1.0 RAP was amended to incorporate updates from the v3.0 protocol, which included increasing the window of the end of study visit in each study part, from  $\pm$  1 h to  $\pm$  1 day. Thus, ensuring sufficient time to complete all agreed procedures. Furthermore, additional clarification relating to the collection of urine for PK assessments has also been included.

#### 3.1 Responsibilities

The Data Sciences Department at Quotient will be responsible for the production of the following items using Quotient SOPs: Clinical Data Interchange Standards Consortium (CDISC) study data tabulation model (SDTM) and analysis data model (ADaM) datasets, safety and PK outputs; including all TFLs, and formal statistical analysis; and the clinical study report (CSR).

Quotient will provide two sets of TFLs during the study:

- Post database lock TFLs (draft) for MMV review
- Post-review TFLs (final) for inclusion into the CSR

Quotient will be responsible for the quality control (QC) of all deliverables prior to the client review (Section 14.2).

All Holter ECGs will be collected electronically using a Mortara H12+ Holter Recorder and analysed by Banook. The reporting of the ECG Holter data is not the responsibility of Quotient and will be subject of a separate analysis plan and will not be part of the final study CSR.

If required, metabolite profiling and genetic testing will the responsibility of The Doctors Laboratory and will be the subject of a separate analytical work plan should the analysis be required. Metabolite profiling may be included in the CSR as an addendum, however genetic testing will be reported separately.

#### 3.2 Definitions

#### 3.2.1 Subject Definitions

During the clinical phase of the study, an evaluable participant in Part 1 and Part 3 is defined as a participant who received the study drug and completed safety and PK

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


assessments up to 96 h post-dose (Part 1)/post-final dose (Part 3). In Part 2, a participant will be considered evaluable if they have received the study drug and completed safety and PK assessments up to 96 h post-dose in both periods. This will be monitored during the clinical phase to identify any requirement for replacement subjects. This definition will not be used during the reporting phase including the identification of analysis populations and datasets which are defined in Section 5.7.

In all study parts, an enrolled participant is defined as a participant who signed the informed consent, qualified per the inclusion/exclusion criteria, and was randomised.

#### 3.2.2 Definition of Treatments

Throughout the reporting of the study, the test product will be referred to as MMV367 and the investigational medicinal products (IMPs) relating to each study part are presented in Table 1, Table 2 and Table 3, respectively.

Table 1 Description of Regimens: Part 1

| SAD<br>Cohort | Regimen | IMP | Dose | Route of Administration | TFL Label |
|---|---|---|---|---|---|
| 1A | 1 | MMV367 or placebo | 100 mg | Oral, Fasted | 100 mg |
| 1B | 2 | MMV367 or placebo | 300 mg <sup>a</sup> | Oral, Fasted | 300 mg |
| 1C | 3 | MMV367 or placebo | 750 mg <sup>a</sup> | Oral, Fasted | 750 mg |
| 1D | 4 | MMV367 or placebo | 1500 mg <sup>a</sup> | Oral, Fasted | 1500 mg |
| 1E<br>Optional | 5 | MMV367 or placebo | 2000 mg <sup>a</sup> | Oral, Fasted | 2000 mg |

<sup>&</sup>lt;sup>a</sup> Predicted dose

Table 2 Description of Regimens: Part 2

| Food Effect<br>Cohort | Period | Regimen | IMP | Dose <sup>a</sup> | Route of Administration | TFL Label |
|---|---|---|---|---|---|---|
| 24 | 1 and 2<br>(randomised) | 6 | MMV367 | XX mg | Oral, Fasted | XX mg Fast |
| 2A | | 7 | MMV367 | XX mg | Oral, Fed | XX mg Fed |

<sup>&</sup>lt;sup>a</sup> The dose administered in Part 2 will be determined once predicted human therapeutic concentrations of MMV367 and a safe exposure window has been established in Part 1. The dose for Regimens 6 and 7 will be the same.

Table 3 Description of Regimens: Part 3

| Multiple Dose<br>Cohort | Regimen | IMP | Doseª | Route of Administration | TFL Label |
|---|---|---|---|---|---|
| 3A | 8 | MMV367 or placebo | XX mg for 3 days | Oral, Fasted | XX mg |
| 3B<br>Optional | 9 | MMV367 or placebo | XX mg for<br>3 days | Oral, Fasted | XX mg |
| 3C<br>Optional | 10 | MMV367 or placebo | XX mg for<br>3 days | Oral, Fasted | XX mg |

<sup>&</sup>lt;sup>a</sup> The dose(s) administered in Part 3 will be determined after review of the data from Part 1.

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Where pooling of active or placebo subjects is required within a study part (i.e., safety summaries in Part 1 and Part 3) these will be presented as All Active and All Placebo respectively.

#### 3.2.3 Definition of Visits

For clinical data, visits will be referred to as Day throughout this document, and each Day will be stated as screening, Day -1 (Admission), with the following duration based on study Part:

- Part 1: Day 1 through to Day 5, with a return visit on Day 7 and an end of study visit on Day 15
- Part 2: Day 1 through to Day 7 Period 1, and Day 8 through to Day 12 in Period 2, with an end of study visit on Day 14 (The actual dosing days within Period 2 may change if the washout period is extended – see Section 8.1.2 of the study protocol)
- Part 3: Day 1 through to Day 7, with a return visit on Day 9 and an end of study visit on Day 17.

Time points within these days are detailed in the schedule of assessments for each study part Appendix 4 (Part 1), Appendix 5 (Part 2) and Appendix 6 (Part 3).

Baseline is defined as nominally the last measurement recorded prior to the first dose of IMP, for each dosing period.

4 Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary To assess the safety and tolerability of single and multiple oral doses of MMV367 in healthy participants | Incidence of adverse events (AEs), physical examination findings, and change from baseline for vital signs, electrocardiograms (ECGs) and laboratory safety tests. |
| Secondary To assess the pharmacokinetics (PK) of single and multiple doses of MMV367 in plasma (Parts 1, 2 and 3) | PK parameters such as AUC, Tmax, Cmax, CL/F, Vz/F, T1/2 and AR, when applicable |
| To assess the effect of a high-fat meal on the PK of a single dose of MMV367 in healthy participants (Part 2 only) | PK parameters such as AUC, Tmax, Cmax and Frel, as appropriate, under fed and fasted conditions |
| Exploratory To assess the PK of single dose of MMV367 in urine (Part 1 only) of healthy participants (optional) <sup>a</sup> | Urine PK parameters such as Ae, and derived plasma PK parameters such as CLr, when applicable |
| To assess exposure response relationship for potential effects of MMV367 on ECG intervals (QT, QTcF, QTcB, PR, QRS) <sup>b</sup> | ECG intervals, MMV367 plasma concentrations (time-matched) |
| To investigate metabolite(s) of MMV367 in healthy participants <sup>a</sup> | Metabolite characterisation for MMV367 in plasma and urine, when applicable |
| To evaluate the taste attributes (smell, sweetness, bitterness, flavour, mouthfeel/texture, grittiness and aftertaste) and overall acceptability of the IMP (Part 1 only) | Taste questionnaire score, based on a 9-point Likert scale assessing the acceptability for each taste attribute (smell, sweetness, bitterness, flavour, mouthfeel/texture, grittiness, and aftertaste) and overall acceptability for each dose level of MMV367 |

<sup>&</sup>lt;sup>a</sup> Depending on availability of the data, these objectives may be reported in an addendum to the final study Clinical Study Report (CSR) or in a separate report.

Check validity before use

<sup>&</sup>lt;sup>b</sup> This objective will be reported in a separate cardiac safety report and will not be part of the final study CSR

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


# 5 Study Design

## 5.1 Brief Description

The study is divided into Parts 1, 2 and 3. For each of the three parts, participants will be screened within 28 days prior to first admission to the clinical unit on the morning of Day -1. Each participant will receive verbal and written information followed by signing of the informed consent form (ICF) prior to any screening procedures taking place.

#### 5.1.1 Part 1 - Single Ascending Dose Cohorts

Part 1 will be a double-blinded, randomised, placebo-controlled, SAD study, which will comprise up to 5 fasted cohorts (Cohorts 1A to 1E; Cohort 1E will be optional), with 8 participants in each cohort. Participants will be randomly assigned to receive a single oral dose of either active IMP (6 participants) or placebo (2 participants) to assess its safety, tolerability and PK profile. Each participant will take part in one cohort. The data obtained from each cohort (safety, tolerability and PK) will undergo a formal review by the safety advisory committee (SAC). The SAC will determine if it is safe and appropriate to proceed with the next dose/cohort. Following review of the emerging PK data from each preceding cohort, if results suggest that the exposure plateau has been reached, the next planned cohort will not be conducted. Similarly, if PK predictions suggest that this exposure plateau would be exceeded at the next cohort/dose level, a lower dose than originally anticipated will be proposed.

It is planned to enrol 8 healthy male and female participants per cohort to ensure data in a minimum of 4 participants (per cohort) on active IMP. In each cohort, participants will be dosed on Day 1 and will remain resident in the clinical unit until discharge on Day 5. They will attend the clinical unit for a return visit on Day 7 and again on Day 15 (±1 day) for end of study assessments. Blood samples will be collected at regular intervals for PK analysis and safety from Day 1 to discharge from the study on Day 15 (±1 day), as detailed in Appendix 2. Each cohort will follow the same study design (Figure 1).

Figure 1 Study Sequence: Part 1 (Cohorts 1A to 1E)



Each participant will take part in one cohort and will receive one of the regimens presented in Table 1, according to the randomisation schedule.

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


There will be a blinded interim review of the safety, tolerability and PK data after each cohort prior to the dose decision for subsequent cohorts. Full details of the interim data reviews are provided in Section 5.2.

Participants will also complete a written taste/palatability questionnaire individually and privately following administration of the IMP. In the evening of Day -1, participants will be trained to respond to a sample questionnaire using a suitable example fluid (e.g., orange juice/squash). On the morning of Day 1, participants will brush their teeth using tap water (toothpaste not permitted). In order to evaluate taste, participants will hold the IMP in their mouth and swirl it around for 10 to 15 sec before swallowing. Immediately after swallowing, they will complete a taste questionnaire individually and privately.

#### 5.1.2 Part 2 – Food Effect Cohort

Part 2 will be an open-label, randomised, balanced two-period crossover, food effect evaluation. The effect of food on the PK of MMV367 will be explored in Part 2 by administering a single dose of MMV367 after a high-fat breakfast, as per FDA guidance, and a single dose of MMV367 in the fasted state.

Each participant will receive 2 single doses of MMV367. In Period 1, participants will be randomised to 1 of 2 treatment sequences (Regimen 6/Regimen 7 or Regimen 7/Regimen 6). If a participant is randomised to receive MMV367 in the fasted state (Regimen 6) in Period 1, they will receive MMV367 in the fed state (Regimen 7) in Period 2 and vice versa. It is planned to enrol 8 healthy male and female participants to ensure data in a minimum of 6 participants.

Participants will be dosed on Day 1 (Period 1 dose) and on Day 8 (Period 2 dose) and will remain resident in the clinical unit until discharge on Day 12. They will attend the clinical unit on Day 14 (±1 day) for end of study assessments. Based on emerging PK data from Part 1, the washout period between the Period 1 and Period 2 doses may be extended. Blood samples will be collected at regular intervals for PK analysis and safety from Day 1 to the end of study visit on Day 14 (±1 day), as detailed in Appendix 3. The study design for Part 2 is presented in Figure 2.

Figure 2 Study Sequence: Part 2



QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Each participant will receive Regimens 6 and 7, presented in Table 2.

## 5.1.3 Part 3 – Multiple Dose Cohort(s)

Part 3 will be a double-blinded, randomised, placebo-controlled, multiple-dose study. A total of 8 participants per cohort will receive once-daily doses of MMV367 (6 participants) or placebo (2 participants) for 3 days, in the fasted state, to assess safety, tolerability and PK profile of multiple dosing.

It is planned to enrol 8 healthy male and female participants to ensure data in a minimum of 4 participants on active IMP.

Participants will receive a single dose on Days 1, 2 and 3 and will remain resident in the clinical unit until discharge on Day 7. They will attend the clinical unit for a return visit on Day 9 and again on Day 17 (±1 day) for end of study assessments. Blood samples will be collected at regular intervals for PK analysis and safety from Day 1 to discharge from the study on Day 17 (±1 day), as detailed in Appendix 4. Each cohort will follow the same study design (Figure 3).

Figure 3 Study Sequence: Part 3 (Cohorts 3A to 3C)



Each participant will receive one of the regimen(s) presented in Table 3 according to the randomisation schedule.

During the interim review of each cohort within Part 1, if it is determined that the optimal dose has been identified for the assessment of food effect, Part 2, may commence prior to the completion of Part 1, provided that this is justified by PK and safety data obtained from completed cohorts in Part 1. Similarly, Part 3 may commence prior to the completion of Part 1 if the required dose level is identified during interim review. However, the total amount of active IMP administered as multiple doses (i.e., cumulative 3-day dose) in Part 3 will be no greater than the maximum safe and well tolerated dose identified Part 1, dosed at a single dose level. Parts 2 and 3 may be conducted in parallel.

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


The data obtained (safety and PK) from the multiple dose administration will undergo a formal review by the SAC after all 8 participants have completed the study. Consequently, Part 3 may be extended to evaluate a second and/or third dose level in a 3-day QD regimen.

Parts 1 and 3 will follow a sentinel dosing design. On the first day of dosing in each cohort in Part 1 and in Part 3, only 2 (sentinel) participants will be dosed. The randomisation schedule will be constructed such that 1 of the participants dosed on the first day will receive MMV367 and 1 will receive placebo. After review of the safety data up to 96 h post-dose for SAD cohorts in Part 1 and up to 96 h post-final dose in Part 3, the investigator, or medically qualified designee who is familiar with the study protocol and IB, and medical monitor or delegate (with approval from the sponsor's medical director or delegate) will decide whether to proceed with dosing the remaining participants in the cohort.

#### 5.2 Criteria for In-Study Decisions

In-study decisions will be made by the safety advisory committee (SAC), which will always comprise the investigator, the medical monitor, the sponsor's medical director, and PK, together with appropriate representation from the partner organisation (GlaxoSmithKline plc [GSK]) where appropriate.

#### 5.2.1 Decision Points

The following in-study decisions will be made during this study:

- Dose selection for Cohorts 1B to 1E in Part 1
- Progression from Cohort 1D to 1E in Part 1
- Washout period duration between periods in Part 2
- Dose selection for Parts 2 and 3
- Changes to safety and/or PK time points, if there is reason to believe that the change might improve the quality of the data as a consequence of review of emerging data
- Progression from Cohort 3A to further multiple dose levels in Part 3

#### 5.2.2 Criteria for Dose Decision

Part 1: Single Ascending Dose Cohorts 1A to 1E

Progression to the next dose cohort will be permitted after review of safety, tolerability and PK data suggests that it is safe to do so. Quotient will provide data to the SAC in accordance with Quotient's standard operating procedure (SOP) on interim dose decision making and dose escalation. The decision will be documented and signed by the investigator as per Quotient's current SOP. Evidence of the decision will be retained in the ISF and Trial Master File.

For dose escalation to proceed, data must be available from a minimum of 6 participants who have completed the planned safety assessments up to 7 days after dosing and planned PK assessments up to 144 h after dosing to ensure at least 4 participants had received active IMP. Dose increases will only be made after a complete review of all data collected from the previous dose group by the SAC.

It is planned that the dose will be escalated for each subsequent cohort; however, the SAC may also agree to enrol additional participants for an intermediate dose level if

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


warranted or may agree to reduce the dose with no limit on the possible extent of reduction. Any decision to investigate an intermediate or reduced dose level will be fully documented.

The decision to proceed to the next dose level will be based on safety, tolerability and available PK data. The following data are required:

- AEs
- Vital signs
- Safety laboratory results
- ECGs
- Physical examination findings
- Plasma concentrations of MMV367
- Interim PK parameter estimations (Tmax, Cmax, AUC(0-24), AUC(0-48), AUC(0last), AUC(0-inf), T1/2, where possible and appropriate)

Rules for dose decision are as follows:

- Dose increments between SAD cohorts will be a maximum of 3-fold and dose escalation may be halted in the SAD cohorts if an exposure plateau appears to have been reached
- Dose increments between multiple dose optional cohorts will be no more than 3fold
- No dose selected for SAD or MAD will be expected to result in a mean group exposure at the next dose level (based on predicted human PK and assuming dose linearity) greater than AUC(0-inf) 376 μg.h/mL, and Cmax 23.8 μg/mL based on the NOAEL in dogs and the corresponding human therapeutic exposure
- The predicted exposure (AUC(0-inf)) of the cumulative dose after a 3-day treatment will not exceed that of a single dose evaluated in Part 1 which is safe and well tolerated
- The study will be halted (see Section 8.5 of the study protocol) and thus a further dose decision will not be made if:
  - One or more participants experience an IMP-related serious AEs (SAE)
  - Two or more participants experience an IMP-related severe or clinically significant non-serious AE at the same dose level/same cohort

If, following review by the SAC it is deemed acceptable to continue dose escalation above the defined maximal dose or exposure limit, a substantial amendment with relevant data will be submitted for approval to the Medicines and Healthcare products Regulatory Agency (MHRA) and ethics committee (EC).

Progression from Part 1 (SAD) to Part 2 (Food Effect).

For the dose level decision to be made for Part 2, data must be available from a minimum of 6 participants who have completed the planned safety assessments up to 7 days after dosing and planned PK assessments up to 144 h after dosing (to ensure at least 4 participants had received active IMP), at a relevant dose level in Part 1. A "relevant dose level" is defined as a dose that demonstrated acceptable safety/tolerability (i.e., exposure levels at which no study specific criteria stopping dose progression and/or escalation were met) at a mean exposure that is not anticipated to be exceeded by the

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


dosing regimen in Part 2, taking into account a potential bioavailability increase to 100% after a high-fat breakfast.

Progression from Part 1 (SAD) to Part 3 (Multiple Dose).

For the dose level decision to be made for Part 3, data must be available from a minimum of 6 participants who have completed the planned safety assessments up to 7 days after dosing and planned PK assessments up to 144 h after the final dose (to ensure at least 4 participants had received active IMP), at a relevant dose level in Part 1. The total dose in Part 3 (3 × QD dose) will not exceed a dose of MMV367 administered and evaluated as a single dose in Part 1, and the predicted exposure will not exceed an exposure observed and determined to be safe in Part 1. If a less than dose-proportional increase in exposure is observed in Part 1 (SAD), the proposed dose(s) for Part 3 may be adjusted to ensure the equivalent exposures between SAD and MAD.

#### 8.2.1 Criteria for Sentinel Dosing Decisions

For all cohorts following a sentinel design (Parts 1 and 3) the decision to proceed with the main group will be made by the investigator, based on safety data until 96 h postdose (Part 1) or 96 h post-final dose (Part 3) in the sentinel participants. The investigator or medically qualified designee who is familiar with the study protocol and IB, and medical monitor or delegate (with approval from the sponsor's medical director or delegate) will decide whether to proceed with dosing the remaining participants in the cohort.

#### 5.3 Study Sample Size

For Parts 1 and 3, the primary objective is an initial assessment of safety and each treatment group is therefore limited to 6 participants receiving active IMP. Administration of MMV367 to 6 participants at each dose level provides a 47%, 62%, 74%, or 82% probability of observing at least 1 occurrence of any AE, with a true incidence rate for a given dose group of 10%, 15%, 20%, or 25%, respectively.

Furthermore, it is assumed that pooling the data for the 2 participants who receive placebo in each cohort will provide an adequately sized control group to assess a possible drug effect on safety laboratory tests, vitals and ECG parameters.

Part 2 is a pilot evaluation designed to determine whether MMV367 PK is impacted by high-fat food. Historically, 8 participants have proven sufficient to characterise the preliminary effects of food on safety and PK of a new chemical entity in healthy participants. Therefore, a sample size of 8 is considered adequate at this stage of drug development.

#### 5.4 Randomisation (including Replacement Subjects)

Parts 1 and 3 will be randomised (IMP/placebo) and double-blinded. Part 2 will be randomised (fed/fasted) and open-label. A randomisation schedule will be produced for each study part. Instructions to dispense and dose will be produced prior to dosing using the randomisation schedule and will be retained in the ISF.

For Part 2, the original randomisation schedule and proof of quality control procedures will be held by the Data Sciences department at Quotient until the study is archived, at which time the randomisation materials will be retained in the ISF.

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Using computer-generated randomisation schedules, participant numbers will be allocated to treatment regimens in a 6:2 ratio (MMV367:placebo) in each cohort (Part 1 or Part 3). In Part 2, the allocation will be balanced with 8 participants assigned to receive MMV367 in both the fed and fasted states. Participants will be randomised to 1 of 2 treatment sequences (Regimen 6/Regimen 7 or Regimen 7/Regimen 6) on Day 1 prior to dosing in the first period.

For participants in Parts 1 and 3, a sentinel group of 2 participants will be dosed ahead of the remaining participants in each cohort. For each cohort, using a computer-generated randomisation schedule, the first 2 participant numbers will be allocated to active or placebo in a 1:1 ratio (i.e., 1 participant will be randomly assigned to receive MMV367 and 1 participant will be randomly assigned to receive placebo). The remaining 6 participant numbers will be allocated to active or placebo in a 5:1 ratio (i.e., 5 participants will be randomly assigned to receive MMV367 and 1 participant will be randomly assigned to receive placebo).

Participants will be randomised immediately before administration of the first dose.

#### 5.4.1 Participant Numbers

Participant numbers will be allocated on the morning of dosing according to the code 101 to 140 in Part 1, 201 to 208 in Part 2, and 301 to 324 in Part 3 using the lowest number available. Replacement participants will be allocated participant numbers 901 to 940 in Part 1, 801 to 808 in Part 2 and 701 to 724 in Part 3, where the last two digits are the same as those of the original participant (e.g., if Participant 105 withdraws, the replacement will have Participant Number 905 and will receive the same regimen as Participant 105).

In Part 1, up to 2 replacement participants may be used per cohort. The maximum number of participants that may be dosed is 50 (8+2 per cohort). In Part 2, up to 4 replacement participants may be enrolled into the study. The maximum number of participants that may be dosed in Part 2 is 12 (8+4). In Part 3, up to 2 replacement participants per cohort (if optional cohorts are utilised) may be enrolled into the study. The maximum number of participants that may be dosed is 30 (8+2 per cohort).

Any participant withdrawn due to an IMP related AE will not be replaced.

Participants withdrawing for other reasons may be replaced as required by agreement between the investigator and sponsor to ensure sufficient evaluable participants. Participant numbering by study part and cohort is provided in Table 4.

**Table 4** Participant Numbers

| Study Part | Cohort | Participant Numbers |
|------------|---------------|---------------------|
| | 1A | 101–108 |
| | 1B | 109–116 |
| 1 | 1C | 117–124 |
| | 1D | 125–132 |
| | 1E (optional) | 133–140 |
| 2 | 2A | 201–208 |
| | 3A | 301–308 |
| 3 | 3B (optional) | 309–316 |
| | 3C (optional) | 317–324 |

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


#### 5.5 Blinding Issues

Parts 1 and 3 of the study are double-blinded. Treatment assignment will not be known to the participants, the sponsor or the staff who are involved in the clinical evaluation of the participants and the analysis of data. If appearance matching of the placebo is not possible then masking and/or unblinded dosing teams will be used to preserve the study blind. Further details of these steps will be contained in the study specific blinding plan, which will be approved prior to dosing. The randomisation schedules and disclosure envelopes will be generated by an unblinded statistician at Quotient according to Quotient's SOPs. The unblinded statistician will not be involved in any decisions relating to populations for analysis prior to unblinding. Prior to database lock and unblinding, all original randomisation materials, including the original final signed and dated randomisation schedule, will be held by the Quality Assurance (QA) department at Quotient. The Data Sciences department will not have access to the randomisation schedule before database lock and unblinding.

Interim PK parameter estimations will be performed using bioanalytical data applied with participant aliases in order to maintain the study blind.

There may be instances where interim PK data have the potential to be treatment revealing e.g., missed blood sampling occasions. In these cases, every effort will be made by the pharmacokineticist to maintain the study blind by appropriate presentation of data to the study team. Data demonstrating extremes of exposure will always be presented, regardless of the potential to reveal the study blind. To permit selection of the dose level, individual data may be made available in full if judged necessary by the investigator or sponsor regardless of the potential to reveal study blind.

The unblinded Qualified Person or designee at the clinical site will receive a copy of the final randomisation schedule for preparation of the study drug and preparation of the instructions to dispense and dose. A copy of the randomisation schedule will also be made available to the laboratory performing the bioanalysis to allow selective analysis of drug concentrations (for Parts 1 and 3) and to the pharmacovigilance provider for analysis of pharmacovigilance.

Two sets of disclosure envelopes (i.e., sealed envelopes containing individual participant randomisation details) will be provided. One set will be held in the clinical area and the other retained in the ISF. These may be used in the event of an emergency by the investigator or delegate. Any request for information on the randomisation schedule after initial issue must be made using a randomisation disclosure form, except in the case of emergency unblinding, which must be recorded on the emergency unblinding form. Access to study drug assignment will be immediately available if the investigator deems it necessary to break the study blind in the interest of a participant's medical safety, in case of a medical emergency, or if warranted during scheduled safety reviews. The medical monitor must be contacted within 24 h following disclosure of study drug assignment.

Details of any disclosure of the randomisation schedule will be documented and retained in the ISF. The sponsor will be notified if the study blind is broken.

Part 2 of the study is open-label and therefore blinding is not required.

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


#### 5.6 Unblinding procedures

The study blind will be broken after the study database has been locked and the safety population has been defined. Any subsequent request for issue of the randomisation schedule prior to unblinding must be made using a randomisation disclosure form.

#### 5.7 Maintaining the Blind During Interim PK Analyses

The interim PK analysis/analyses in Part 1 and Part 3 will be performed on QC checked concentration data for MMV367 in plasma using nominal sampling times and doses. Data will be received with participant aliases applied to the concentration data in order to maintain the study blind.

There may be instances where interim data has the potential to be treatment revealing eg missed blood sampling occasions. In this case every effort will be made by the pharmacokineticist to maintain the study blind by appropriate restriction/modification of data presented to the study team, such as only presenting the summary statistics e.g., mean, SD, minimum, median, maximum, geometric mean and geometric CV% for both PK parameters and concentration data.

Data demonstrating extremes of exposure will always be presented, regardless of the potential to reveal the study blind. Further details can be found in the blinding plan.

# 6 Populations and Analysis Sets

## 6.1 Safety Population and Safety Analysis Set

The safety population and safety analysis sets will be defined separately for each study part.

The safety population will include all subjects who have received any amount of IMP.

The safety analysis set will be defined on a treatment basis and will include all safety data from the subjects included in the safety population who have received that treatment.

The safety population will be confirmed by Quotient with approval from MMV after database lock (Part 2) and prior to unblinding (Part 1 and Part 3) and will be summarised for the populations table and to determine the subjects to be included in the safety analysis set.

The safety analysis set will be confirmed by Quotient with approval from MMV at the same time as the relevant safety population and will be summarised for the analysis of demographic and baseline characteristics, and all safety data.

#### 6.2 Taste Population and Taste Analysis Set

The taste population will include all subjects who have received at least one regimen (i.e., active dose or placebo), in Part 1, and held it in their mouth for approximately 10 to 15 seconds. Participants will have also completed the taste questionnaire for a regimen and have no relevant protocol deviations for any taste test or AEs which confound the taste assessment.

The taste population will be determined by Quotient with approval from MMV after database lock and will be used for the taste tables and to determine the participants to be included in the taste analysis set.

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


The taste analysis set will be defined on a regimen basis and will include all relevant data from the participants included in the taste population who have received that test product.

The taste analysis set will be determined by Quotient with approval from MMV at the same time as the taste population and will be used for all summary tables and formal statistical analysis of taste data.

#### 6.3 Pharmacokinetic Population and Pharmacokinetic Analysis Set(s)

The PK population will be defined separately for study Parts 1, 2 and 3 and will include all subjects who have received at least one dose of IMP and who satisfy the following criteria for at least one profile:

- No missing samples or invalid post-dose analytical results at critical time points e.g., around Cmax
- No relevant protocol deviations that may impact the study objectives with respect to the PK endpoints
- No relevant AEs such as vomiting that suggest that the whole dose was not available for absorption for a particular participant

Handling of the urine concentration data is not currently a planned analysis in the CSR; however, should a validated method be developed and the urine concentrations be required to be reported by Quotient in Part 1, then the following should apply to the processing of the urine data. Any protocol deviations or AEs specific to the analysis of urinary PK parameters will be documented as an update to the PK population when urine data are available for analysis. Subjects who received placebo in Part 1 and 3 will not be included in the PK population.

The PK analysis set will be defined on a per-treatment basis and will include all relevant data from the subjects included in the PK population who have received that treatment.

In Part 1, individual subjects will be excluded from the PK analysis set where deemed appropriate such as if the participant's data for the treatment affected did not meet the bullet point criteria above, or other study emergent point related to PK analysis or interpretation.

In Part 2, individual participant profiles (i.e., treatments) will be excluded from the PK analysis set where deemed appropriate such as if the participant's data for the treatment affected did not meet the bullet point criteria above, or other study emergent point related to PK analysis or interpretation.

In Part 3, individual subjects will be excluded from the PK analysis set where deemed appropriate such as if the participant's data for the treatment affected did not meet the bullet point criteria above for at least one individual profile (i.e., day), or other study emergent point related to PK analysis or interpretation.

Individual participant profiles in Part 3 (i.e., days) will be flagged and excluded from the PK summary statistics where deemed appropriate such as if the profile in the day affected did not meet the bullet point criteria above, or other study emergent point related to PK analysis or interpretation.

The PK population and analysis set will be confirmed by Quotient with approval from MMV following derivation of all PK parameter estimates.

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


If required, a PK analysis subset(s) will also be documented by Quotient, with approval from MMV, at the same time as the PK population and analysis set, if additional subjects are required to be excluded from the statistical analysis (i.e., to exclude subjects who have not received both the fed and fasted treatments in Part 2).

All enrolled subjects will be used for the PK data listings. The PK population will be used for the populations table. The PK analysis set and/or the PK analysis subset(s), if defined, will be used for the provision of PK summary tables and figures as well as the formal statistical analysis and will be documented as the same time as the PK population.

# 7 Participant Disposition, Demographics and Baseline Characteristics

No formal statistical testing will be performed on participant disposition, or on demographic or baseline data. Summaries of participant disposition and analyses populations will be based on all enrolled subjects and summaries of all other data described in this section will be based on the safety analysis set unless otherwise stated.

#### 7.1 Screening Failures

For each study part, data for subjects who have failed screening will be databased but will not be cleaned and therefore will not be included in the SDTM or ADaM datasets or any of the TFLs or the CSR.

#### 7.2 Participant Disposition and Withdrawals

For each study part, the number and percentage of subjects randomised, dosed, completed and discontinued will be presented by sequence and overall in Part 2, and by all placebo, all active and each dose level in Part 1 and Part 3. If any subjects discontinued from the study early then the number of subjects for each reason for discontinuation will be presented by sequence and overall in Part 2, and by all placebo, all active and each dose level in Part 1 and Part 3. However, if none of the subjects are discontinued from the study early, then the reasons for discontinuation will not be populated in the summary table. A participant may be discontinued from the study early for 1 reason only.

Participant disposition and withdrawal data will be listed including details of informed consent.

Protocol deviations and any violations of the inclusion/exclusion criteria will also be listed.

#### 7.3 Analysis Populations

A summary table will be produced detailing the number and percentage of subjects in each population (i.e., safety/taste/PK, as applicable) by sequence and overall in Part 2, and by all placebo, all active and each dose level in Part 1 and Part 3. The reasons for exclusion from each population will also be included in the summary table. However, if none of the subjects were excluded from a population, then the reasons for exclusion will not be populated in the summary table. A participant may be excluded from a population for more than 1 reason. The denominator for the percentage is the number of subjects enrolled in the respective sequence in Part 2, and the number of subjects enrolled in Part 1 and Part 3.

Details of subjects included and excluded in the different analysis populations will be listed.

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


#### 7.4 Analysis Sets and Subsets

A summary table will be produced detailing the number and percentage of subjects in each of the safety, taste and PK analysis sets and analysis subsets (if applicable) for each treatment and overall in Part 2, and by all placebo, all active and each dose level in Part 1 and Part 3. Separate tables will be presented for safety, taste and PK, analysis sets and each table will be based on the relevant population the analysis set is derived from. If analysis subsets are defined they will be included on the same table as the corresponding analysis set. The reasons for exclusion from each analysis set/subset will also be included in the summary. However, if none of the subjects were excluded from an analysis set, then the reasons for exclusion will not be populated in the summary table. A participant may be excluded from an analysis set for more than 1 reason. The denominator for the percentage is the number of subjects in each population.

Details of subjects included and excluded in the different analysis sets/subsets will be listed.

#### 7.5 Demographic Characteristics and Lifestyle Details

Demographic data (age, ethnicity, race, sex, height [cm], weight [kg] and body mass index [BMI; kg/m²]) will be recorded at screening.

Summary statistics (number of subjects with an observation [n], mean, standard deviation [SD], median, minimum and maximum) will be presented for age, height, weight and BMI at screening by sequence and overall in Part 2, and by all placebo, all active and each dose level in Part 1 and Part 3. The number and percentage of subjects will be presented by sequence and overall in Part 2, and by all placebo, all active and each dose level in Part 1 and Part 3 for ethnicity, race and sex. The denominator for the percentage is all subjects in the safety analysis set. If any values are missing, a "missing" row will be presented on the table.

Lifestyle details (i.e., smoking history [does the participant smoke, use e-cigarettes or use nicotine replacement products?] and alcohol consumption) will be summarised by sequence and overall in Part 2, and by all placebo, all active and each dose level in Part 1 and Part 3, as a categorical variable.

Demographic and lifestyle data for all enrolled subjects will be listed. For Part 2 only, separate columns will be provided in the demographic listing for body weight at screening and admission.

#### 7.6 Medical History

Medical history will be recorded for each participant at the screening visit and updated at admission. Medical histories will be coded using MedDRA v25.0 (or a more recent version) including Lowest Level Term, Preferred Term (PT), and System Organ Class (SOC).

All medical history data will be listed including coded terms.

## 7.7 Prior and Concomitant Medication

Medications (product name) will be coded using the World Health Organization (WHO) Drug Dictionary Global Drug Reference version 2022 March (or more recent version) using the following Anatomical Therapeutic Chemical (ATC) classification codes

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


- Product name
- Preferred name
- Drug code
- Therapeutic subgroup (ATC 2nd level code)
- Chemical subgroup (ATC 4th level code)

Prior medications are defined as medications that start and stop prior to the first dose of IMP. All other medications will be defined as concomitant medications including those that start prior to the first dose of IMP and continue thereafter. Any medications with an unknown start or stop date will be assumed to be concomitant medications unless a partial start or stop date indicates otherwise.

All medications, including coded terms, and the underlying indication for which the medication was given, will be listed. One combined data listing of prior and concomitant medications will be provided. All prior medications as defined above will be flagged with a "#" symbol. Within this flagged group medications that started after screening and stopped before dosing of IMP will also be flagged using a "\*" symbol.

#### 7.8 Other Baseline Characteristics

All other baseline characteristics, as listed below, at screening and on admission (unless otherwise stated) will be listed separately for each study part:

- Carbon monoxide breath test
- Urine drug screen
- Alcohol breath test
- Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) Antigen test
- Beck Depression Inventory (BDI-II) Questionnaire
- Virology (Screening only)
- Creatinine clearance (Admission only)
- Follicle stimulating hormone for female subjects (Screening only)
- Serum pregnancy test for female subjects (Screening only)
- Urine pregnancy test (Admission only)

## 8 Efficacy

Not applicable for this Phase I study.

#### 9 Pharmacokinetics

## 9.1 Plasma PK Parameter Estimation

The PK parameters (Table 5 [Part 1 and 2], Table 6 [Part 3]) for MMV367 in plasma will be estimated where possible and appropriate for each participant profile (i.e., treatment/day [where relevant]) by non-compartmental analysis methods using Phoenix WinNonlin software (v8.3 or a more recent version, Certara USA, Inc., USA). Additional parameters may be calculated if required, depending on the data.

#### 9.1.1 Definition of Plasma PK Parameters

Plasma PK parameter definitions are provided in Table 5 and Table 6.

# Table 5 Plasma PK Parameter Definitions and Rounding Specifications – Part 1 and 2

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


| Parameter | Definition | Unit | DP<br>or SF | No. of<br>DP/SF |
|---|---|---|---|---|
| Tmax | Time of maximum observed concentration | h | DP | 2 |
| Cmax | Maximum observed concentration | mass unit/mL | SF | 3 |
| AUC(0-24) | Area under the curve from time 0 to 24 h post dose | mass<br>unit.h/mL | SF | 3 |
| AUC(0-48) | Area under the curve from time 0 to 48 h post dose | mass<br>unit.h/mL | SF | 3 |
| AUC(0-72) | Area under the curve from time 0 to 72 h post dose | mass<br>unit.h/mL | SF | 3 |
| AUC(0-last) | Area under the curve from time 0 to the time of last measurable concentration | mass<br>unit.h/mL | SF | 3 |
| AUC(0-inf) | Area under the curve from time 0 extrapolated to infinity | mass<br>unit.h/mL | SF | 3 |
| AUCextrap | Area under the curve (AUC) from time of the last measurable concentration to infinity as a percentage of the area under the curve extrapolated to infinity | % | DP | 2 |
| T1/2 | Terminal elimination half-life | h | DP | 2 |
| lambda-z | First order rate constant associated with the terminal (log-linear) portion of the curve | 1/h | DP | 4 |
| CL/F | Total apparent body clearance calculated after a single extravascular administration where F (fraction of dose bioavailable) is unknown. | mL/min | SF | 3 |
| CLr <sup>a</sup> | Renal clearance calculated using plasma AUC – Part 1 only | mL/min | SF | 3 |
| Vz/F | Apparent volume of distribution based on the terminal phase calculated using AUC(0-inf) after a single extravascular administration where F (fraction of dose bioavailable) is unknown | L | SF | 3 |
| Frel Cmax | Relative bioavailability based on Cmax (Part 2 fed dosing only) | % | DP | 2 |
| Frel AUC(0-last) | Relative bioavailability based on AUC(0-last) (Part 2 fed dosing only) | % | DP | 2 |
| Frel AUC(0-inf) | Relative bioavailability based on AUC(0-inf) (Part 2 fed dosing only) | % | DP | 2 |
| lambda-z lower* | Lower limit on time for values to be included in the calculation of lambda-z | h | DP | 2 |
| lambda-z upper* | Upper limit on time for values to be included in the calculation of lambda-z | h | DP | 2 |

DP: decimal places; NA: not applicable; SF: significant figures

Table 6 Plasma PK Parameter Definitions and Rounding Specifications – Part 3

<sup>\*</sup> these values should be listed but omitted from the descriptive statistics

<sup>&</sup>lt;sup>a</sup> Renal clearance will only be calculated in Part 1 should a validated method be developed, and the urine concentrations be required to be reported by Quotient, as an addendum to the CSR

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


| Parameter | Definition | Unit | DP or<br>SF | No. of<br>DP/SF |
|---|---|---|---|---|
| Tmax | Time of maximum observed concentration | h | DP | 2 |
| Cmax | Maximum observed concentration | mass unit/mL | SF | 3 |
| AUC(0-tau) | Area under the curve for the defined interval between doses (tau) | mass unit.h/mL | SF | 3 |
| T1/2 | Terminal elimination half-life (Day 3 only) | h | DP | 2 |
| lambda-z | First order rate constant associated with the terminal (log-linear) portion of the curve (Day 3 only) | 1/h | DP | 4 |
| CL/Ftau | Total body clearance calculated using AUC(0-tau) after repeated extravascular administration, where F (fraction of dose bioavailable) is unknown (Day 3 only) | mL/min | SF | 3 |
| Vz/Ftau | Apparent volume of distribution based on the terminal phase calculated using AUC(0-tau) after extravascular administration where F (fraction of dose bioavailable) is unknown (Day 3 only) | L | SF | 3 |
| AR Cmax | Accumulation ratio based on Cmax repeated dose/Cmax single dose (Day 3 only) | NA | DP | 2 |
| AR AUC | Accumulation ratio based on AUC(0-tau) repeated dose/AUC(0-tau) single dose (Day 3 only) | NA | DP | 2 |
| lambda-z lower* | Lower limit on time for values to be included in the calculation of lambda-z (Day 3 only) | h | DP | 2 |
| lambda-z upper* | Upper limit on time for values to be included in the calculation of lambda-z (Day 3 only) | h | DP | 2 |

DP: decimal places; NA: not applicable; SF: significant figures

Dose will be used in the calculation of relevant PK parameters as per Table 7.

**Table 7** Dose Specifications

| Dose (nominal/actual) | Nominal |
|-----------------------|-----------------|
| Precision | As per protocol |

In Part 2, relative bioavailability (Frel) will be calculated as follows:

$$Frel = \left\{ \frac{AUC \text{ or Cmax (test)}}{AUC \text{ or Cmax (reference)}} \right\} \times 100$$

Frel will be calculated using Cmax, AUC(0-last) and AUC(0-inf). If for any reason the AUC(0-inf) is not calculable then an alternative or additional AUC over a partial area may be used to calculate Frel for all subjects.

The following comparisons will be made:

<sup>\*</sup> these values should be listed but omitted from the descriptive statistics

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


 XX mg MMV367 fed [Regimen 7] (test) vs XX mg MMV367 fasted [Regimen 6] (reference)

Renal clearance (CLr) is a plasma parameter and will be calculated as follows in Part 1, if applicable:

$$CLr = \frac{Ae}{AUC}$$

where both amount excreted (Ae) of parent in urine and AUC of parent in plasma are determined over co-incident time ranges after dosing. For example, if urinary Ae is calculated over 0-24 hours then the plasma AUC used will also be calculated over the same period. Details of methods for calculation of CumAe are included in Section 9.2.

## 9.1.2 Rules for Plasma PK Parameter Estimation using WinNonlin

The imputation of non-numerical (e.g., below the limit of quantification [BLQ]) or negative values (e.g., pre-dose sampling times) reported in the input data set will be performed as follows for calculation of PK parameters:

- Pre-dose sample times will be entered as zero
- Values that are BLQ obtained prior to Cmax will be entered as zero
- Values that are BLQ after Cmax will be treated as missing but where BLQ concentrations are defined as parameters these will be reported as BLQ
- Values that are BLQ after Cmax may be imputed as zero for the calculation of partial AUCs, in cases where lambda-z cannot be determined
- Values that are measurable after at least 2 consecutive BLQ values after Cmax will be treated as missing for the calculation of PK parameters
- Values that are reported as "No Result" or "Not Reportable" (NR), "Not Calculated" (NC) or "No Sample" (NS) etc. will be generally be considered missing

Missing or unusual concentration values in the input data may be queried to ascertain any underlying cause. Exclusion of missing or unusual concentration values, or repeat bioanalysis of samples, will only be performed if a definitive root cause can be established and approval from MMV has been obtained. Any exclusions of concentration values or repeat analysis of samples will be documented appropriately.

Check validity before use

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Plasma PK parameters will be estimated using standard Phoenix WinNonlin methods, details of which may be found in the documentation accompanying the WinNonlin software package. The rules specified in Table 8 will be applied:

Table 8 PK Parameter Estimation Details

| Sampling times | Actual |
|---|---|
| Calculation method | Linear Log Trapezoidal |
| Number of points used for lambda-z | At least 3, not including Cmax |
| Minimum requirements for AUC | At least 3 consecutive measurable concentrations |

Where possible, the terminal elimination rate constant (lambda-z) will be calculated for all participant profiles. The value of lambda-z will be determined by the slope of the regression line of the natural log transformed concentrations vs time.

The WinNonlin determined choice of data points for determination of lambda-z will be reviewed by the pharmacokineticist who may adjust the selection in order to provide a more appropriate fit. The choice of data points for determination of lambda-z for each profile will be confirmed following a documented peer review.

## 9.1.3 Plasma PK Parameter Reporting Specifications

The following parameters will be reported for each Study Part/Study Treatment/Study Day as applicable, according to the rounding specifications provided in Table 5 and Table 6:

#### Part 1

Tmax, Cmax, AUC(0-24), AUC(0-48), AUC(0-last), AUC(0-inf), AUCextrap, T1/2, lambda-z, CL/F, CLr\*, Vz/F, lambda-z lower, lambda-z upper

#### Part 2 – fasted

Tmax, Cmax, AUC(0-24), AUC(0-48), AUC(0-last), AUC(0-inf), AUCextrap, T1/2, lambda-z, CL/F, Vz/F, lambda-z lower, lambda-z upper

#### Part 2 - fed

Tmax, Cmax, AUC(0-24), AUC(0-48), AUC(0-last), AUC(0-inf), AUCextrap, T1/2, lambda-z, CL/F, Vz/F, Frel Cmax, Frel AUC(0-last), Frel AUC(0-inf), lambda-z lower, lambda-z upper

#### Part 3, Day 1

Tmax, Cmax, AUC(0-tau)

## Part 3, Day 3

Tmax, Cmax, AUC(0-tau), T1/2, lambda-z, CL/Ftau, Vz/Ftau, AR Cmax, AR AUC, lambda-z lower, lambda-z upper

The flags/footnotes given in Table 9 will be applied to the PK parameters where relevant and will be shown in the PK parameter listings. Additional flags may be applied based on emerging data.

<sup>\*</sup> Renal clearance will only be calculated in Part 1 should a validated method be developed, and the urine concentrations be required to be reported by Quotient, as an addendum to the CSR

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Table 9 PK Parameter Flags and Footnotes

| Flag | Footnote |
|---|---|
| а | Adjusted rsq of regression (the goodness of fit statistic for the elimination phase) was <0.8 |
| b | Period used for regression analysis was less than 2-fold the calculated half-life |
| С | Extrapolated portion of AUC(0-inf) >20% |
| d | Insufficient post-Cmax data points for estimation of lambda-z |
| е | Entire profile BLQ, no PK parameters could be calculated |
| f | Fewer than 3 consecutive measurable concentrations, AUCs not calculated |
| g | Measurable pre-dose values were observed, however were considered less than 5 % of Cmax (Part 2 only) |

In the event that the adjusted rsq of regression is <0.8 ("a" flag) then lambda-z and parameter estimates derived using lambda-z and AUC(0-inf) will be deemed unreliable and will be flagged and listed but excluded from the summary statistics and formal statistical analysis.

In the event that the time period used for regression analysis is less than 2-fold the calculated half-life ("b" flag) T1/2 will be flagged, listed, and included in summary statistics and formal statistical analysis.

In the event that the extrapolated portion of AUC(0-inf) >20% ("c" flag), then AUC(0-inf) and parameter estimates derived using AUC(0-inf) will be deemed unreliable and will be flagged and listed but excluded from the summary statistics and formal statistical analysis.

In the event that there are insufficient post-Cmax data points (i.e., <3) for estimation of lambda-z ("d" flag) then lambda-z and parameter estimates derived using lambda-z and AUC(0-inf) will be reported as NC.

In the event that there are fewer than 3 consecutive measurable concentrations ("f" flag) then all AUC parameter estimates will be reported as NC.

In the event that measurable pre-dose values less than 5% of Cmax were observed ("g" flag), all parameter estimates for the profiles affected will be listed, flagged and included in summary statistics and formal statistical analysis.

Note: in the event that measurable pre-dose concentrations greater than 5% of Cmax are observed, requirements for additional flags and further action will be agreed with MMV and documented at the same time as the PK population.

#### 9.2 Urine PK Parameter Estimation

Handling of the urine concentration data is not currently planned analysis in the CSR. However, should a validated method be developed and the urine concentrations be required to be reported by Quotient in Part 1, then the following should apply to the processing of the urine data.

In Part 1, Cohort 1C and 1D, the urine PK parameters for MMV367 may be derived for each participant and collection interval by treatment using SAS.

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


#### 9.2.1 Definition of Urine PK Parameters

Urine PK parameter definitions are provided in Table 10.

Table 10 Urine PK Parameter Definitions and Rounding Specifications

| Parameter | Definition | Unit | DP | No. of<br>DP |
|---|---|---|---|---|
| Ae | Amount excreted | mass unit | DP | 2 |
| CumAe | Cumulative amount excreted | mass unit | DP | 2 |
| %Ae | Percentage of dose excreted | % | DP | 2 |
| Cum%Ae | Cumulative percentage of dose excreted | % | DP | 2 |

DP = decimal places

Dose is defined as per Table 7

Urine PK parameters will be calculated as follows:

• When converting urine collection weights to urine volume (if required), the following conversion factor will be used:

$$1.02 g$$
 of urine =  $1 mL$  of urine

This will be calculated in SAS as follows:

Urine weight (g) / 1.02 = Urine volume (mL)

 If MMV367 concentrations in urine are provided in mass unit/g the following conversion will be performed using SAS:

Concentration (mass units/g) \* 1.02 = Concentration (mass units/mL)

Ae will be derived for each collection period:

- CumAe, will be calculated by the incremental summation of the Ae over all
  collection periods. Note: The amount excreted in the pre-dose sample should not
  be included in the calculation of the cumulative amount excreted.
- %Ae will be derived for each collection period:

- Cum%Ae will be calculated by the incremental summation of the %Ae over all
  collection periods. Note: The percentage of dose excreted in the pre-dose sample
  will not be included in the calculation of the cumulative percentage of dose
  excreted.
- Where a participant has failed to void over a particular collection interval the Ae for that collection interval will be set to zero.
- If part of a void over a particular collection interval is missing due to spillage or accidental discarding, the Ae will still be calculated providing other samples have

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


been collected within the interval. Where no other samples are collected within the interval the concentration will be set to missing for the purposes of the calculation urine PK parameters. In both scenarios the data will be flagged to highlight a missing void. Affected participant(s) may be excluded from summary statistics, this will be documented as part of the PK population.

 Imputation of non-numerical values reported in the urine dataset (i.e., concentrations that are BLQ) will be entered as zero for calculation of urine PK parameters.

#### 9.3 Concentration and PK Parameter Summary Tables

Summary statistics (i.e., n, mean, SD, CV%, median, minimum, maximum, geometric mean, geometric SD and geometric CV%) of concentration data will be calculated for each time point and treatment for MMV367 in plasma. The number of BLQ values (n#) per time point will also be presented. Geometric statistics will not be calculated for Day 1, pre-dose concentrations.

Summary statistics (i.e., n, mean, SD, CV%, median, minimum and maximum) of plasma PK parameters will be calculated for MMV367 for each treatment and day (where appropriate). Geometric mean, geometric SD and geometric CV% will be presented for all plasma PK parameters except Tmax.

In Part 1, Cohort 1C and 1D, should a validated method be developed, and the urine concentrations be required to be reported by Quotient in Part 1, urine Ae and CumAe will be summarised using the n, mean, SD, CV%, median, minimum, and maximum) whilst %Ae and Cum%Ae will be summarised using the n, mean, SD, CV%, median, minimum and maximum only.

Non-measurable values reported in the plasma concentration data (i.e., values that are BLQ), will be entered as zero for the determination of summary statistics with the exception of geometric means, geometric SD and geometric CV%, where BLQ values will be imputed as half the lower limit of quantification (LLOQ) value. This also applies to any concentrations that are defined as PK parameters. Data recorded as NR, NS or NC will be handled as missing (i.e., no assumption will be made about the actual concentration).

#### 9.4 Concentration and PK Figures

Mean, spaghetti and individual plasma concentration vs time plots will be produced on both the linear/linear scale and on log10/linear scale. For all plots on a linear/linear scale, pre-dose concentration values reported as BLQ will be set to zero. Post-dose concentration values reported as BLQ will be set to zero, up to the point at which all concentrations fall below the LLOQ, after which they will be presented as missing. For all plots on a log 10/linear scale, pre-dose concentration values reported as BLQ will be presented as missing. Post-dose concentration values reported as BLQ will be set to half the BLQ value, up to the point at which all concentrations fall below the LLOQ, after which they will be presented as missing. Where curves from multiple treatment regimens or subjects are overlaid on the same plot, symbols will be used to identify different subjects/ treatment regimens and a legend will be included on the plots to define the symbols used.

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Mean plasma concentration vs time plots (using nominal times) will be produced for:

#### Part 1

• All treatments on the same plot (1 plot with up to 5 profiles)

#### Part 2

• Fed and Fasted treatments on the same plot (1 plot with 2 profiles)

#### Part 3

- All treatments on the same plot with separate plots for Day 1 and Day 3 (2 plots with up to 3 profiles per plot)
- Day 1 and Day 3 on the same plot, with separate plots for each treatment (up to 3 plots with 2 profiles per plot)

These will be produced as follows:

- Linear/linear scale using arithmetic mean concentrations (error bars ± arithmetic SD)
- Log10/linear scale using geometric mean concentrations (error bars x/÷ geometric SD)

Separate plasma concentration vs time spaghetti plots (using actual sampling time after dosing) will be produced for each treatment (and Day in Part 3) with each plot displaying 1 line per participant.

In Part 2, individual plasma concentration vs time plots (using actual sampling times after dosing) will be produced separately for each individual participant with fed and fasted treatments on the same plot in Part 2. Additionally, in Part 3, individual plasma concentration vs time plots will be produced separately for each participant and each Day, as well as each individual participant and both Days on the same plot.

For the food effect comparison in Part 2, scatter plots of individual plasma PK parameter values for Cmax, AUC(0-last) and AUC(0-inf). The PK parameter estimates will be plotted on the y-axis (linear scale) and regimen on the x-axis. Each participant's individual points will be connected with a line. In addition, the corresponding geometric mean parameter values will be plotted using a different symbol and connected with a thicker line. Separate plots will be produced for each parameter.

#### 9.5 Concentration and PK Listings

The sample collection data (e.g., collection times) for PK samples will be listed. In addition, all concentration data and PK parameters will be listed on a per participant basis. Any flags used will be included as a footnote with the appropriate definition.

#### 9.6 Statistical Analysis of PK Parameters

## 9.6.1 Part 1 and Part 3: Assessment of Dose Proportionality

Formal statistical analysis will be performed on the PK parameters Cmax, AUC(0-last) and AUC(0-inf) in Part 1, and Cmax and AUC(0-tau) in Part 3, including data from up to 5 different dose levels in Part 1 and up to 3 different dose levels, on Day 1 and Day 3 separately in Part 3 to assess dose proportionality. This will be assessed using a power model as follows:

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


$$log (AUC or Cmax) = \mu + \beta \times log(dose)$$

where  $\mu$  and  $\beta$  are the intercept and the slope of the model, respectively. The PK parameters will be undergo a natural log transformation. The model will include the log dose as a fixed effect and log PK parameter as the dependent variable The analysis will be performed using SAS Software procedure PROC MIXED, the method will be specified as Restricted Maximum Likelihood and the denominator degrees of freedom for the fixed effects will be calculated using Kenward and Roger's method.

The model is usually referred to as a power model [1] as after exponentiation:

AUC (or Cmax) = 
$$\alpha \times dose^{\beta}$$

The estimate obtained for  $\beta$  together with its 90% CI will be presented along with the number of subjects and the geometric means.

The following is an example of the SAS Software code that will be used:

Where LVAR is the log transformed PK parameter and LDOSE is the log transformed dose.

Dose proportionality will be assessed against the critical region defined by the formula below [2][3]:

$$1 + \frac{\ln (\theta_L)}{\ln (r)} < \beta < 1 + \frac{\ln (\theta_H)}{\ln (r)}$$

where:  $\theta_L = 0.50$  $\theta_H = 2.00$ 

r = ratio highest dose level/lowest dose level

 $\beta$  = slope of line as a measure of dose proportionality from power model

If the 90% CI for  $\beta$  lie entirely within the critical region defined above, dose proportionality will be concluded over the dose range under analysis. The critical region will be calculated using SAS Software as part of the statistical analysis and presented in the analysis table as a footnote.

In addition, the power model will be used to estimate the increase in the PK parameter resulting from a doubling in the dose i.e.,  $2^{\beta}$  90% CI associated with this estimate will also be provided.

This analysis will be performed if there is quantifiable plasma PK data for a minimum of 3 active dose levels. Dose levels will be included in the analysis if quantifiable plasma PK data is available for a minimum of 3 subjects within the relevant dose level.

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Where dose proportionality cannot be concluded over the full dose range then dose proportionality may be assessed over a reduced dose range to identify if dose proportionality exists over a narrower dose range.

#### 9.6.2 Part 2: Assessment of Food Effect

Formal statistical analysis will be performed on the PK parameters Cmax, AUC(0-last) and AUC(0-inf), to assess the presence of a food effect. The null hypothesis is that there is no difference between fed and fasted treatments.

The PK parameters will undergo a natural logarithmic transformation and will be analysed using mixed effect modelling techniques. The model will include terms for fed/fasted status and period fitted as fixed effects and participant fitted as a random effect.

Only subjects who complete both the fed and fasted periods will be included in the statistical analysis. Furthermore, for AUC(0-inf) only, a participant must have reliable estimates of AUC(0-inf) for both fed and fasted periods to be included in the statistical analysis. If the number of subjects with reliable estimates for both periods is less than 4 (i.e., less than 50% of planned number of evaluable subjects) then no formal statistical analysis of AUC(0-inf) will be performed i.e., descriptive summaries only.

The adjusted means including differences from the fed/fasted comparison and the associated 90% CIs obtained from the model are back transformed on the log scale to obtain adjusted geometric mean ratios (GMRs) and 90% CIs of the ratio. These will be presented together with the p-value from the fed/fasted comparison.

The fixed effects table from the model with F-statistic and p-value for the relevant effects will be presented in a separate table.

The intra-participant variability values will be calculated for all treatments combined and are obtained from the residual term from the SAS Software output. These values are calculated as follows:

```
CVw = 100 x (exp(Mean Square Error) - 1)^{1/2}
```

The analysis will be performed using the SAS Software procedure PROC MIXED, the method will specified as Restricted Maximum Likelihood and the denominator degrees of freedom for the fixed effects will be calculated using Kenward-Roger method [4]. The following is an example of the SAS Software code that will be used:

```
PROC MIXED DATA=<input dataset name> METHOD=REML ORDER=INTERNAL;
    CLASS SUBJIDN FSTATUS APERIODN;
    MODEL LVAR = FSTATUS APERIODN / OUTP=PRED DDFM=KR;
    RANDOM SUBJIDN;
    ESTIMATE <relevant pairwise treatment comparisons> / CL ALPHA=0.10;
    LSMEANS TRTAN / ALPHA=0.10;
    LSMEANS=MEANS ESTIMATES=EST COVPARMS=CVW;
RUN;
```

#### where

- LVAR is the natural log transformed PK parameter of interest
- SUBJIDN is the numeric participant identifier variable
- APERIODN is the numeric period variable

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


FSTATUS is the numeric variable representing fasted or fed status

For each analysis, distributional assumptions underlying the statistical analyses will be assessed by visual inspection of residual plots. Normality will be examined by normal probability (QQ) plots, while homogeneity of variance will be assessed by plotting the residuals against the predicted values for the model. If the distributional assumptions for the parametric approach are not satisfied, then additional sensitivity analyses may be performed including the removal of potential outliers or the use of non-parametric methods to assess the robustness of the original analysis. This will be documented in the CSR together with the reasoning supporting the most appropriate action taken, if applicable. In general terms the results of the original analysis will always be presented in the CSR.

#### 9.6.3 Statistical Figures for Analysis of Pharmacokinetic Data

In Part 1, to complement the dose proportionality assessment the geometric mean values of the PK parameters used to evaluate dose proportionality, along with the geometric SDs from the mean will be presented graphically on a log<sub>10</sub> scale by log<sub>10</sub> (dose level).

Additionally, the individual values for PK parameters used in the evaluation of dose proportionality will also be presented graphically on a log<sub>10</sub> by log<sub>10</sub> (dose level) scale and the power model regression line will be included on these plots.

#### 9.7 Interim Pharmacokinetic Analysis

The details of the planned interim PK analysis are described in this section. However, as the analysis will be performed in real time it may be necessary to change the planned analysis in response to the emerging data.

Summary tables and figures for the interim PK analysis will be presented in an Interim PK Summary Report after being exported from WinNonlin. The formatting of this output will differ slightly from the final PK output which will be produced using SAS to include in the CSR.

The interim PK analysis will be performed on QC checked concentration data for MMV367 in plasma using nominal sampling times and doses. Measures will be taken to maintain the study blind according to Section 5.7.

The following PK parameters will be calculated for the interim analysis:

#### <u> Part 1</u>

Tmax, Cmax, AUC(0-24), AUC(0-48), AUC(0-last), AUC(0-inf), T1/2.

#### Part 3 Day 1:

Tmax, Cmax, AUC(0-tau)

#### Part 3 Day 3:

Tmax, Cmax, AUC(0-tau), T1/2, AR Cmax, AR AUC

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


#### 10 Taste Assessment

For Part 1 only, Taste/Palatability will be assessed using a questionnaire (example provided in Appendix 7 at the time points detailed in Appendix 4. The questionnaire will ask participants to rate the overall acceptability of taste/palatability, with additional questions asked on specific palatability attributes (smell, sweetness, bitterness, flavour, mouth feel/texture, grittiness, and aftertaste), on a 9-point Likert scale. The clinical staff will provide definitions and examples of each aspect that is being rated if required.

Each participant in Part 1 of the study will complete the questionnaire individually and privately, within no more than 10 min, following IMP administration.

## 10.1 Summary Tables for Taste Questionnaire Assessments

Acceptability of taste (overall liking of product) will be summarised (i.e., n, mean, SD, median, minimum and maximum) by treatment.

For each of the taste attributes described above, the number and percentage of subjects who selected each taste rating on the 9-point scale and/or N/A will be summarised by treatment. The safety population will be used as the denominator in the calculation of percentages.

#### 10.2 Listings for Taste Questionnaire Assessments

All taste assessments data will be listed.

#### 10.3 Statistical Figures for Analysis of Taste Questionnaire Data

In Part 1, to complement to assessment of the taste questionnaire data, boxplots of each dose level will be produced separately for each taste attribute and overall acceptability. Dose level will be plotted on the X axis and taste assessment score will be plotted on the Y axis (i.e., 1=Dislike extremely, 2=Dislike very much etc.).

Additionally, bubble plots of each taste attribute and overall acceptability will be produced. Each dose level will be plotted on the X axis, with the assessment score plotted on the Y axis. Each bubble will contain a count of the number of subjects which scored a particular outcome. The size of the bubble will reflect the count (i.e., The bubble associated which the most popular score will be the biggest).

# 11 Safety Assessments

Safety data summaries will be presented by actual treatment and the safety analysis set will be used throughout.

#### 11.1 Extent of Exposure and Treatment Compliance

The number and percentage of subjects dosed with IMP (each day, Part 3 only), will be presented for all placebo, all active, and each active dose level separately in Part 1 and Part 3, and by treatment received in Part 2.

Dosing details (including the date and time of all IMP administrations and any comments) will be listed for all enrolled subjects. Any recorded deviations from the planned dosing regimen will be listed as protocol deviations. Total number of days of exposure and measures of compliance will be included in the listing (Part 3 only).
QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


#### 11.2 Meal Details

For Part 2 only, meal details as recorded on the electronic case report form (eCRF) will be listed for all enrolled subjects. Any recorded deviations from the planned mealtimes will be listed as protocol deviations.

#### 11.3 Adverse Events

Throughout the study, all AEs will be evaluated by the PI and noted in the AE section of the eCRF. An AE is any untoward medical occurrence in a participant that occurs either before dosing (referred to as a pre-dose AE) or once a medicinal product has been administered, including occurrences which are not necessarily caused by or related to that product.

AEs will be coded using the Medical Dictionary for Regulatory Activities MedDRA v25.0 (or more recent version), and reported by SOC and PT.

AEs will be classified into the following categories:

- Pre-dose AEs: AEs recorded at screening or with a start date and time prior to the first dose of IMP
- Treatment-emergent AEs (TEAEs): AEs that commence during/after the first dose
  of IMP or commence before first dose of IMP (i.e., a pre-dose AE or existing
  medical condition) but worsen in intensity during exposure to IMP

For Part 2 only, TEAEs will be assigned to the treatment of the period in which the AE first occurred. Where the severity of an AE intensifies or symptoms change in a subsequent period, this will be defined as a new AE and included under the regimen associated with the subsequent period. Adverse events that occur during the washout period will be assigned to the treatment the participant received during the period immediately before the washout period.

Adverse events will be classified as "mild," "moderate" or "severe" when considering their severity

Adverse events will be classified as "unrelated", or "related" when considering their relationship to IMP. TEAEs classified as "related", will be defined as IMP-related events. Pre-dose AEs will always have the classification of "unrelated"

If the severity or relationship to IMP of a TEAE is missing, the severity/relationship will be tabulated as "missing" in the summary tables

When summary presentation is made by maximum severity, "missing" will be handled as follows:

- If there are other events (i.e., same SOC and PT code) with a maximum severity recorded as "moderate" or "severe" for that participant and regimen, then the maximum observed severity for that participant will be categorised and presented as "moderate" or "severe", respectively
- If there are other events (i.e., same SOC and PT code) with a maximum severity recorded as "mild" for that participant and regimen, then the maximum observed severity for that participant will be categorised and presented as "missing"

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


When summaries are presented by relationship to IMP, "missing" will be handled as follows:

- If there are other events (i.e., same SOC and PT code) with a most closely related association recorded as "related" for that participant and regimen, then the maximum observed relationship for that participant will be categorised and presented as "related", respectively
- If there are other events (i.e., same SOP and PT code) with a most closely related association recorded as "unrelated" for that participant and regimen, then the maximum observed relationship for that participant will be categorised and presented as "missing"

Where the start date of an AE is missing and the stop date is on or after the day of first dose of IMP or both the start and stop dates are missing then a "worst-case" scenario will be assumed i.e., the AE is assumed to have occurred post-dose and is therefore considered treatment-emergent. If a partial start date/time is available then the event will be considered as treatment-emergent unless the partial information suggests otherwise.

### 11.3.1 Summary Tables for Adverse Events

All pre-dose AEs (as defined in Section 11.3 will be excluded from the summary tables but will be listed for all enrolled subjects.

Descriptive statistical methods will be used to summarise the TEAE data.

For each study part, the number and percentage of subjects reporting each TEAE will be presented for both SOC and PT. For summaries by SOC and PT, with the exception of TEAEs by severity and relationship to IMP, the number of subjects and the number of events will be summarised. For summaries by severity and relationship only the number of subjects will be summarised.

For counts of subjects experiencing events the following will apply:

#### Part 1 and Part 3:

- A participant with a TEAE in more than one body system will be counted once in the total number of subjects with TEAEs
- A participant with more than 1 TEAE in the same SOC counts only once at the SOC level
- A participant with more than 1 TEAE in the same PT counts only once at the PT level

#### Part 2:

- A participant experiencing TEAEs in more than one body system, within a period,
   will be counted once in the total number of subjects with TEAEs in that period
- A participant with more than 1 TEAE in the same SOC, within a period, counts only once at the SOC level
- A participant with more than 1 TEAE in the same PT, within a period, counts only once at the PT level

For event counts, all events are included.

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


When it is necessary to calculate percentages, the denominator will be the total number of subjects in the safety analysis set (and period – Part 2 only), and the numerator will be the total number of subjects reporting a TEAE within the relevant category.

Summaries presented for SOC and PT will be presented in descending order of frequency overall i.e., most frequently reported SOC in the study part and then by most frequently reported PT in the study part within each SOC.

## 11.3.1.1 Overall Summary of Adverse Events

The following will be summarised by treatment and overall, in Part 2, and by all placebo, all active, and each dose level in Part 1 and Part 3 for the safety analysis set:

- Number and percentage of subjects reporting at least 1 TEAE
- Number and percentage of subjects reporting severe TEAEs
- Number and percentage of subjects reporting IMP-related TEAEs
- Number and percentage of subjects reporting serious TEAEs
- Number and percentage of subjects reporting TEAEs leading to participant withdrawal
- Number and percentage of subjects reporting TEAEs leading to death
- Total number of TEAEs
- Total number of severe TEAEs
- Total number of IMP-related TEAEs
- Total number of serious TEAEs
- Total number of TEAEs leading to participant withdrawal
- Total number of TEAEs leading to death

#### 11.3.1.2 Summary of Treatment-Emergent Adverse Events

All subjects reporting TEAEs will be summarised by treatment and overall in Part 2, and by all placebo, all active and each dose level in Part 1 and Part 3. Counts will be given for number of subjects and number of events. Subjects experiencing more than 1 TEAE treatment will be counted only once for number of subjects but will be counted more than once for number of events.

Additionally, subjects reporting TEAEs will be summarised for SOC and PT by treatment and overall in Part 2, and by all placebo, all active and each dose level in Part 1 and Part 3. Counts will be given for number of subjects and number of events. Subjects experiencing more than 1 episode of a TEAE within a treatment will be counted only once within each SOC and PT using the most severe episode.

#### 11.3.1.3 Summary of Treatment-Emergent Adverse Events by Severity

All subjects reporting TEAEs will be summarised by severity (i.e., mild, moderate or severe) and by treatment in Part 2, and by all placebo, all active and each dose level in Part 1 and Part 3. Counts will be given for number of subjects, not number of events. Counts will be given by maximum severity (i.e., subjects experiencing more than 1 TEAE within a treatment will be counted only once using the most severe episode).

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Additionally, subjects reporting TEAEs will be summarised for SOC and PT by maximum severity (i.e., mild, moderate or severe) and by treatment in Part 2, and by all placebo, all active and each dose level in Part 1 and Part 3. Counts will be given for total number of subjects, not for events. Counts by maximum severity will be given (i.e., subjects experiencing more than 1 TEAE within a treatment will be counted only once within each SOC and PT using the most severe episode).

#### 11.3.1.4 Summary of Treatment-Emergent Adverse Events by Relationship to IMP

All subjects reporting TEAEs will be summarised by relationship to IMP (i.e., unrelated, or related) and by treatment in Part 2, and by all placebo, all active and each dose level in Part 1 and Part 3. Counts will be given for number of subjects, not number of events. Counts will be given by the closest relationship to IMP (i.e., subjects experiencing more than 1 TEAE within a treatment will be counted only once using the most closely related event).

Additionally, subjects reporting TEAEs will be summarised for SOC and PT by closest relationship to IMP (i.e., unrelated or related) by treatment in Part 2, and by all placebo, all active and each dose level in Part 1 and Part 3. Counts will be given for total number of subjects, not for events. Counts by closest relationship will be given (i.e., subjects experiencing more than 1 TEAE within a treatment will be counted only once within each SOC and PT using the most closely related event).

# 11.3.1.5 Summary of IMP-related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

All subjects reporting IMP-related TEAEs will be summarised by treatment in Part 2, and by all placebo, all active and each dose level in Part 1 and Part 3. Counts will be given for number of subjects and number of events. Subjects experiencing more than 1 IMP-related TEAE within a treatment will be counted only once for number of subjects but will be counted more than once for number of events.

Additionally, subjects reporting IMP related events will be summarised for SOC and PT by treatment in Part 2, and by all placebo, all active and each dose level in Part 1 and Part 3. Counts will be given for number of subjects and number of events. Subjects experiencing more than 1 episode of an IMP-related TEAE within a treatment will be counted only once within each SOC and PT using the most severe episode.

#### 11.3.1.6 Summary of Serious Adverse Events

All subjects reporting treatment-emergent serious AEs (SAEs) will be summarised by treatment in Part 2, and by all placebo, all active and each dose level in Part 1 and Part 3. Counts will be given for number of subjects and number of events. Subjects experiencing more than 1 SAE within a treatment will be counted only once for number of subjects but will be counted more than once for number of events.

Additionally, subjects reporting treatment-emergent SAEs will be summarised for SOC and PT by treatment in Part 2, and by all placebo, all active and each dose level in Part 1 and Part 3. Counts will be given for number of subjects and number of events. Subjects experiencing more than 1 episode of a SAE within a will be counted only once within each SOC and PT using the most severe episode.

#### 11.3.2 Listings for Adverse Events

All pre-dose AEs (as defined in Section 11.3) will be listed including SOC and PT.

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


A separate data listing of all TEAEs will be provided including the SOC and PT. In addition, a listing of all SAEs will be provided.

#### 11.4 Laboratory Evaluations

The details of sample collection for laboratory safety analysis are described in the study protocol.

Where a value is provided by the safety laboratory as either above or below the limit of detection (LOD) this will be set to the respective LOD itself for descriptive summaries. No imputations will be made in the individual listings.

### 11.4.1 Summary Tables for Laboratory Evaluations

For each study part, haematology, coagulation and clinical chemistry data will be summarised (n, mean, SD, median, minimum and maximum) for each laboratory parameter at each time point, including changes from baseline (Admission, Day-1) at each scheduled post-baseline time point by treatment in Part 2, and by all placebo, all active and each dose level in Part 1 and Part 3.

Shift tables from baseline to each scheduled post-baseline time point (with respect to the number and percentage of subjects with values below, within or above the reference range) will be presented by treatment in Part 2, and by all placebo, all active and each dose level in Part 1 and Part 3. Percentages will be based on the number of subjects with measurements at baseline and the relevant post-baseline time point.

For fasting-sensitive laboratory parameters (i.e., glucose) results taken in the non-fasted state (i.e., LBFAST=N) will not be included in summary statistics by time point or be used in derivations of changes from baseline. For tabulations (e.g., shift tables) both fasted and non-fasted results will be pooled and used in the tabulations, using the appropriate fasted or non-fasted reference range. All results (fasted or non-fasted) will be listed with non-fasted data flagged.

Reference ranges for each laboratory parameter will be presented for the relevant parameter in each summary table.

#### 11.4.2 Listings for Laboratory Evaluations

For each study part, the sample collection data (e.g., collection times) for laboratory analysis and urinalysis data will be listed.

All individual participant data, for planned haematology, clinical chemistry and urinalysis data including derivations, such as change from baseline, will be listed. If applicable, data from unscheduled laboratory tests will also be listed and flagged with a "#" to indicate it will not be used in the summary statistics. In these listings, individual data will be flagged with an "H" or an "L" for values that are higher or lower than their reference ranges, respectively.

Separate listings of all haematology, coagulation, clinical chemistry and urinalysis values outside their reference ranges by participant will also be provided. Reference ranges will be supplied by the safety laboratory for haematology and clinical chemistry and per the eCRF for urinalysis (i.e., a positive or negative result) with the exception of the following reference ranges for urinalysis:

• pH: 5.0 to 9.0

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


• Specific gravity: 1.000 to 1.030

#### 11.5 Vital Signs

For each study part, the details of measurement of supine vital signs (i.e., systolic and diastolic BP, and heart rate) and non-supine vital signs (oral temperature and respiratory rate) will be measured at each scheduled timepoint.

Systolic and diastolic BP and heart rate orthostatic measurements will also be taken (1 supine and 1 standing) according to the time schedules presented in Appendix 4 (Part 1), Appendix 5 (Part 2) and Appendix 6 (Part 3). Vital signs parameters will be reported in the order given above, i.e., both summary tables and data listings.

### 11.5.1 Summary Tables for Vital Signs

For each study part, vital signs data (including orthostatic measurements), and change from baseline (Pre-dose, Day 1 (Period 1), Day 8 (Period 2), will be summarised (i.e., n, mean, SD, median, minimum and maximum) at each post-baseline time point by treatment in Part 2, and by all placebo, all active and each dose level in Part 1 and Part 3.

In addition, the number of subjects with 'substantial' increases or decreases or no substantial change from baseline in systolic BP (>20 mmHg), diastolic BP (>10 mmHg) and heart rate (>15 bpm) will be summarised.

Orthostatic hypotension will also be investigated at each time point. The change in systolic BP and diastolic BP between the mean of the duplicate supine measurements and the subsequent standing measurement will be calculated for each subject (i.e., standing BP- Supine BP) and summarised (i.e., mean, SD, median, minimum, maximum and n) at baseline and each post-baseline time point.

In addition, the number of subjects with 'substantial' decreases or no substantial decrease from supine to standing results in systolic BP (>20 mmHg) and diastolic BP (>10 mmHg) will be presented at each time point.

#### 11.5.2 Listings for Vital Signs

For each study part, all individual vital signs data (including orthostatic measurements) and derivations, such as change from baseline, will be listed. Individual data will be flagged with an "H" or an "L" for values that are higher or lower than their reference ranges, respectively, and subjects with 'substantial' increases or decreases from baseline (as defined in Section 11.5.1) in systolic BP, diastolic BP and heart rate will be flagged with an 'l' (increase) or 'D' (decrease), respectively. If applicable, data from unscheduled vital signs assessments will also be listed and flagged with a "#" to indicate it will not be used in the summary statistics.

In addition, a separate listing of all vital signs data outside their reference ranges by participant will also be provided.

The reference ranges (from Quotient SOP "The Interpretation of the Electrocardiogram, Vital Signs and Clinical Laboratory Data During Phase I / II Clinical Trials") defined in Table 11 will be used.

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


**Table 11 Vital Signs Reference Ranges** 

| Parameter | Lower limit | Upper limit |
|-----------------------|----------------|----------------|
| Systolic BP | 90 mmHg | 140 mmHg |
| Diastolic BP | 50 mmHg | 90 mmHg |
| Heart rate | 45 bpm | 100 bpm |
| Oral Body Temperature | 35.5°C | 37.5°C |
| Respiration Rate | 10 breaths/min | 24 breaths/min |

NA=Not applicable

#### 11.6 ECGs

For each study part, the details of measurement of supine ECG parameters (i.e., ventricular rate, RR interval, QT interval, QTcF interval, PR Interval, QRS duration, QRS axis, rhythm, interpretation and clinical significance and findings) are described in the study protocol. ECG parameters will be reported in the order given above, i.e., both summary tables and data listings.

Triplicate 12-lead ECGs (2 min apart) will be obtained after the participant has been in the supine position for a minimum of 5 min.

On Day 1 of Parts 1 and 2, telemetry (continuous ECG monitoring) will commence at least 30 min before dosing until at least 12 h post-dose. As this monitoring is for safety purposes alone no data will be recorded in the source, except the start and stop time. If cardiac monitoring shows a potentially significant abnormality, a clinical assessment of the participant including a 12 lead ECG will be performed and treatment given, if appropriate.

#### 11.6.1 Summary Tables for ECGs

For each study part and time point where triplicate ECGs are taken the arithmetic mean of the triplicate values for each 12-lead ECG measurement will be computed for each participant. These arithmetic means will then be used to compute the summary statistics for the observed values and for the change from baseline values. If 1 of the 3 measurements is missing, the mean of the 2 non-missing measurements will be used. If 2 measurements are missing, the remaining non-missing value will be used.

ECG data, including change from baseline (mean of single 12-lead measurement, Predose, Day 1 of each dosing period where applicable), will be summarised (i.e., n, mean, SD, median, minimum and maximum) at each post-baseline time point by treatment in Part 2 and by all placebo, all active and each active dose in Part 1 and Part 3.

For each study part, the number and percentage of subjects with normal and prolonged QT intervals corrected for heart rate using Bazett's correction (i.e., QTcB) and Fridericia's correction (i.e., QTcF) and increases in QTcB and QTcF intervals from baseline within the categories defined in Table 12 (based on the International Council on Harmonisation [ICH] E14 guideline [5]) will be summarised by time point and overall. Percentages will be based on the number of subjects with measurements at the relevant time point.

Check validity before use

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Table 12 ICH E14 Ranges for QTcB and QTcF Intervals

| Parameter | ICH E14 Range |
|-----------------------------------------------|--------------------|
| QTcF/ QTcB interval | ≤450 msec (normal) |
| | >450msec |
| | >480 msec |
| | >500 msec |
| Increase in QTcF/ QTcB interval from baseline | ≤30 msec |
| | >30 msec |
| | >60 msec |

## 11.6.2 Listings for ECGs

For each study part, all ECG measurements (i.e., single and mean of triplicate readings) including derivations, such as change from baseline, will be listed.

All ECG measurements will be flagged with an "H" or an "L" for values that are higher or lower than their reference ranges, respectively. If applicable, data from unscheduled ECG assessments will also be listed and flagged with a "#" to indicate it will not be used in the summary statistics.

In addition, for the single values obtained from Single 12-lead measurement, and the mean values calculated from the triplicate ECG values, the number of subjects with increase in QTcF interval from baseline (>30 msec) and with 'substantial increases' (>60 msec) will be flagged with 'I' and 'SI', respectively.

A separate listing of all ECG parameters outside their reference range by participant will also be provided. The reference ranges (from Quotient SOP "The Interpretation of the Electrocardiogram, Vital Signs and Clinical Laboratory Data During Phase I / II Clinical Trials", except QT interval which is from the eCRF) defined in Table 13 will be used.

Additionally, for Part 1 and Part 2 only, the telemetry start and stop times, as well as the nature of any potentially significant abnormality will be listed.

Table 13 ECG Reference Ranges

| Parameter | Lower limit | Upper limit |
|-----------------------|-------------|-------------|
| Ventricular Rate (HR) | 45 bpm | 100 bpm |
| QT Interval | 200 msec | 600 msec |
| QTcB/QTcF Interval | NA | 450 msec |
| PR Interval | 120 msec | 210 msec |
| QRS Duration | NA | 120 msec |
| QRS Axis | -30° | 100° |

HR=heart rate NA=Not applicable

#### 11.7 Body Weight

In Part 1 and Part 3, all body weight data will be listed.

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


#### 11.8 Physical Examination

All physical examination and targeted physical examination details and comments on any findings will be listed by participant for all subjects.

## 12 Interim Statistical Analyses

No interim statistical analysis is planned for this study.

# 13 Changes in the Conduct of the Study or Planned Analysis

## 13.1 Changes in the Conduct of the Study

No changes in the conduct of the study had been reported at the time this document was written.

#### 13.2 Changes to the Planned Analyses

No changes to planned analysis.

## 13.3 Any Other Relevant Changes

Not applicable.

## 14 Overall Considerations

#### 14.1 Statistical Programming and Analysis

The Data Sciences Department at Quotient will perform the statistical programming and analysis to produce all analysis datasets and TFLs using the statistical SAS Software v9.4.

In general terms, categorical data will be presented using counts and percentages, while continuous variables will be presented using n, mean, SD, median, minimum and maximum. For PK data additional statistics including CV%, geometric mean, geometric SD and geometric CV% will be presented, as appropriate.

The geometric mean is obtained by applying a natural log transformation to the raw data, calculating the arithmetic mean of the transformed values and then back transforming the arithmetic mean.

The following formula will be used to calculate the geometric SD:

ie, a natural log transformation is applied to the raw data, the arithmetic SD of the transformed values is calculated, and then the arithmetic SD of the transformed values is back transformed.

The following formula will be used to calculate the geometric CV%:

geometric CV% = 
$$100 \times (\exp{SD[(\log(\text{raw data})]}^2 - 1)^{1/2}$$

ie, a natural log transformation is applied to the raw data, the arithmetic SD of the transformed values is calculated. This value is then squared. The square value is back transformed and a value of 1 is subtracted from the back transformed value. A square root is then applied and the resulting value is multiplied by 100.

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


In general summary statistics and statistical analysis results will be presented as detailed in Table 14, unless otherwise stated:

Table 14 Reporting Conventions for Summary Statistics and Statistical Analysis

| | Statistic | Number of decimal places for reporting (i) |
|---|---|---|
| Data Type | | |
| Erogueney | Counts (n) | None |
| Frequency | Percentages (%) | 1 decimal place |
| | n | None |
| | Mean | i + 1 decimal places |
| | Median | i + 1 decimal places |
| | SD | i + 1 decimal places |
| | Min | i decimal places |
| Summary statistic | Max | i decimal places |
| | CV% | 1 decimal place |
| | Geometric n | None |
| | Geometric Mean | i + 1 decimal places |
| | Geometric SD | i + 1 decimal places |
| | Geometric CV% | 1 decimal place |
| | Ratios (%) | 2 decimal places |
| | Confidence intervals (%) | 2 decimal places |
| Statistical analysis | | if <0.001: presented as <0.001 |
| | p-values | if ≥0.001 and <0.099: presented to 3 decimal places |
| | | all other p-values will be presented to 2 decimal places |

i refers to the number of decimal places reported in the eCRF or other appropriate source data for the original data. Where bioanalytical or PK data are received rounded in significant figures rather than decimal places, summary statistics will be supplied to the same precision.

Details of how the individual PK parameters will be presented are detailed in Section 9.1.1. Where data requires rounding, values ending with 1 to 4 will be rounded down and values ending with 5 to 9 will be rounded up.

All data listings will be based on all enrolled subjects (as defined in Section 3.2.3). Details of age and sex will be included on all data listings.

For the assessment of food effect in Part 2, statistical tests relating to PK parameters will be 2-sided and will be performed using a 10% significance level, leading to 90% (2-sided) confidence intervals (CIs).

If any baseline measurements are found to be missing then consideration will be given to imputation using the preceding time point (e.g., screening, admission, if applicable). Unscheduled assessment may be used if appropriate. Details of any such imputations will be documented as part of the safety analysis set.

There will be no other imputations for the safety data with regard to missing values or study discontinuation (i.e., subjects who do not complete the study). Imputation for PK parameter estimation using WinNonlin is described in Section 9.1.2. Imputations for reporting PK data are described in Section 9.1.3.

If partial dates are available for smoking history, prior medications or medical/surgical history, there will be no date imputations. The data listings will only show the date information for the date part that is available, e.g., if only the year part of the date is available then YYYY will be presented in the listing. If the full date information is missing, then this will be presented as missing on the data listing.

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Separate summary TFLs will be produced for Part 1, Part 2 and Part 3 of this study, respectively. The different parts will be identified by a sub-title indicating the relevant part. The text in the remainder of this document refers to both parts, unless specified otherwise. All summary tables within a study part relating to Part 1 or 3, except for the plasma PK concentration and plasma and urine PK parameter summary tables will be presented by all placebo subjects combined (i.e., all placebo subjects pooled over all dose levels), all active doses combined (i.e., all active subjects pooled over all dose levels) and all active dose levels separately. Summary tables relating to Part 2 will be presented by treatment. For the plasma PK concentration and plasma and urine PK parameter summary tables, these will be presented by all treatments separately. Placebo subjects will not be included on the PK concentration and plasma and urine PK parameter summary tables. TFLs of the same type will have the same TFL numbering with the inclusion of a .1 for Part 1 of the study and a .2 for Part 2 of the study etc. If all or part of this study is conducted during the Coronavirus disease 2019 [COVID-19] pandemic and there is evidence that data relating to primary and/or key secondary endpoints may have been affected in a way that may bias results, then sensitivity analyses may be conducted. Requirements for any sensitivity analyses will be documented at the same time as the related population (i.e., safety /PK population) and details of any sensitivity analyses which were carried out would be fully documented in the CSR.

# 14.2 Quality Control of Summary Tables, Figures and Listings and Statistical Analysis

Isolated data errors detected as a result of the QC checks that are deemed significant (i.e., errors that would impact the interpretation of the results in relation to the study objectives) will be corrected as per the data management plan. Systematic data errors will be investigated further. The data will be corrected if necessary, and the appropriate table, figure, and/or listing re-generated and then re-checked.

In addition to QC checks, a documented peer review will be performed of all SAS Software -generated report standard TFLs, including a review of SAS Software code and program log files.

#### 14.2.1 Quality Control - Summary Tables

Manual QC methods (i.e., comparison of results in the table to results calculated by a calculator or spreadsheet) will be used for all analyses and summary tables. All summary tables will be QC'd as follows:

- Where tables are presented by sequence or treatment (Part 2), or dose group (Part 1 and Part 3) (i.e., no time points), QC will alternate between sequence or treatment (Part 2) or dose group (Part 1 and Part 3) to avoid the same sequence or treatment (Part 2) or dose group (Part 1 and Part 3) being QC'd every timeFor tables presented by sequence or treatment (Part 2) or dose group (Part 1 and Part 3) only (i.e., no time points), all summary statistics for 1 sequence or treatment (Part 2) or dose group (Part 1 and Part 3) will be QC'd
- Where tables are presented by treatment, or dose group (Part 1 and Part 3 only) and time point, QC will alternate between treatment, or dose group (Part 1 and Part 3 only) to avoid the same treatment, or dose group (Part 1 and Part 3 only) being QC'd every time
- For tables presented by treatment, or dose group (Part 1 and Part 3 only) and time point, a single treatment, or dose group (Part 1 and Part 3 only) at 1 time point in

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


each table will be QC'd

- Where tables are produced using a macro for multiple parameters, a minimum of 3 tables, using different treatment, or dose group (Part 1 and Part 3 only) or combinations of treatment, or dose group (Part 1 and Part 3 only) and time point as appropriate, will be QC'd
- For AEs, the treatment details will be 100% QC'd against the randomisation schedule for all subjects
- AE summary tables will be 100% checked using the relevant data listing

### 14.2.2 Quality Control - Figures

All figures will be QC'd manually using the corresponding/appropriate summary table or data listing, as follows:

- Across all figures, QC will alternate between treatment to avoid the same dose treatment being QC'd every time
- Where a figure presents data from more than 1 treatment, only 1 treatment will be QC'd. However, all data points for that treatment will be checked
- Where figures are produced using a macro for individual subjects and/or multiple parameters, a minimum of 3 figures will be QC'd
- Mean figures will be QC'd using the corresponding summary table
- Figures showing individual data will be QC'd using the corresponding data listing

## 14.2.3 Quality Control - Data Listings

In Part 2, all data listings will be subjected to a 100% manual QC check against the eCRF or other appropriate source data for a minimum of 2 subjects. If appropriate, the subjects checked will include at least 1 participant who withdrew early from the study.

In Part 1 and Part 3, all data listings will be subjected to a 100% manual check against the eCRF or other appropriate source data for a minimum of 2 subjects. If appropriate, the subjects checked will include at least 1 participant who withdrew early from the study.

The study treatment allocation details on the dosing data listing will be 100% QC checked against the study randomisation schedule.

#### 14.2.4 Quality Control - Statistical Analysis

QC of statistical analyses will be performed by peer review of program code, log and output. This will be performed by a statistician at Quotient who is not responsible for performing the statistical analysis.

#### 15 SAS Data Transfer

The SDTM and ADaM datasets will be transferred to MMV at the following times:

- Prior to database lock (SDTM transfer of safety/eCRF data only)
- On the finalisation of the CSR, with the define.xml

The SDTM and ADaM datasets will be programmed according to a pre-defined set of specifications following Quotient SOP DOC-028861, with reference to SDTM IG 3.2 and ADaM IG 1.1. Quotient will provide metadata files and data will be transferred as SAS Software transport files. No define .xml output will be included.

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


## 16 Programming Conventions

Quotient standards for layout of TFLs and programming conventions will be used as follows:

- Courier new, font size 8
- Landscape
- A4 paper

Tables and listings will be produced as MS Word 2016 (or more recent version) documents and figures will be produced as PDF files. Listings will be sorted by participant ID number and sequence or treatment (Part 2 only) or dose group (Part 1 and Part 3) i.e., all subjects in sequence 1 will be presented first, followed by subjects in sequence 2, etc.

The mock tables (Section 21) and titles of all TFLs and the formatting, labelling, footnotes and cosmetic appearance of tables may be modified, or additional labelling/footnotes may need to be added during analysis and reporting, for clarification purposes. Any such changes will not be regarded as changes to planned analyses.

## 17 Reference List

- [1] Gough K, Hutchison M, Keene O, et al. Assessment of dose proportionality: report from the statisticians in the pharmaceutical industry/pharmacokinetics UK joint working party. *Drug Info J.* 1995; 29(3): 1039–1048
- [2] Smith BP, Vandenhende FR, DeSante KA, et al. Confidence interval criteria for assessment of dose proportionality. *Pharmaceutical Research*. 2000; 17(10): 1278–1283.
- [3] Hummel J, McKendrick S, Brindley C, et al. Exploratory assessment of dose proportionality: review of current approaches and proposal for a practical criterion. *Pharmaceutical Statist.* 2009; 8: 38–49
- [4] Brown, Prescott. Repeated measures data. In: Brown H and Prescott R, 3<sup>rd</sup> edition. *Applied Mixed Models in Medicine*. Chichester, UK: John Wiley & Sons Ltd; 2015: 242–243.
- [5] International Council for Harmonisation (ICH) Topic E 14, The Clinical Evaluation of QT/QTc Interval Prolongation and Proarrhythmic Potential for Non-Antiarrhythmic Drugs Guidelines approved by the Committee for Medicinal Products for Human Use (CHMP) in May 2005 which came into force November
- [6] Beck A, Ward C, Mendelson M, et al. An inventory for measuring depression. *Archives of General Psychiatry*. 1961; 4: 561-571


# 18 Index of Tables

| | UI Tables |
|---|---|
| Table<br>Number | Table Title |
| | Participant Disposition, Populations and Datasets |
| 14.1.1.1 | Participant Disposition by Reason<br>Summary Statistics: All Enrolled Subjects<br>Part 1 |
| 14.1.2.1.2 | Analysis Populations Summary Statistics: All Enrolled Subjects Part 1 |
| 14.1.2.1.3 | Safety Analysis Sets Summary Statistics: Safety Population Part 1 |
| 14.1.2.1.4 | Taste Analysis Set<br>Summary Statistics: All Enrolled Subjects<br>Part 1 |
| 14.1.2.1.5 | PK Analysis Sets<br>Summary Statistics: All Enrolled Subjects<br>Part 1 |
| 14.1.1.2 | Participant Disposition by Reason<br>Summary Statistics: All Enrolled Subjects<br>Part 2 |
| 14.1.2.2.2 | Analysis Populations Summary Statistics: All Enrolled Subjects Part 2 |
| 14.1.2.2.3 | Safety Analysis Sets<br>Summary Statistics: Safety Population<br>Part 2 |
| 14.1.2.2.4 | PK Analysis Sets<br>Summary Statistics: All Enrolled Subjects<br>Part 2 |
| 14.1.1.3 | Participant Disposition by Reason<br>Summary Statistics: All Enrolled Subjects<br>Part 3 |
| 14.1.2.3.2 | Analysis Populations<br>Summary Statistics: All Enrolled Subjects<br>Part 3 |
| 14.1.2.3.3 | Safety Analysis Sets<br>Summary Statistics: All Enrolled Subjects<br>Part 3 |
| 14.1.2.3.4 | PK Analysis Sets<br>Summary Statistics: All Enrolled Subjects<br>Part 3 |

| Table<br>Number | Table Title |
|---|---|
| | Demographic and Baseline Characteristics |
| 14.1.3.1 | Demographic and Baseline Characteristics<br>Summary Statistics: Safety Analysis Set<br>Part 1 |
| 14.1.4.1 | Lifestyle Details: Smoking History and Alcohol Consumption<br>Summary Statistics: Safety Analysis Set<br>Part 1 |
| 14.1.3.2 | Demographic and Baseline Characteristics<br>Summary Statistics: Safety Analysis Set<br>Part 2 |
| 14.1.4.2 | Lifestyle Details: Smoking History and Alcohol Consumption<br>Summary Statistics: Safety Analysis Set<br>Part 2 |
| 14.1.3.3 | Demographic and Baseline Characteristics Summary Statistics: Safety Analysis Set Part 3 |
| 14.1.4.3 | Lifestyle Details: Smoking History and Alcohol Consumption<br>Summary Statistics: Safety Analysis Set<br>Part 3 |
| | Dosing Details |
| 14.1.5.1 | Extent of Exposure<br>Summary Statistics: Safety Analysis Set<br>Part 1 |
| 14.1.5.2 | Extent of Exposure<br>Summary Statistics: Safety Analysis Set<br>Part 2 |
| 14.1.5.3.1 | Extent of Exposure: Subjects Dosed by Day<br>Summary Statistics: Safety Analysis Set<br>Part 3 |
| 14.1.5.3.2 | Extent of Exposure: Total Days of Exposure<br>Summary Statistics: Safety Analysis Set<br>Part 3 |
| 14.1.5.3.3 | Extent of Exposure: Percentage Treatment Compliance<br>Summary Statistics: Safety Analysis Set<br>Part 3 |

| Table<br>Number | Table Title |
|---|---|
| | Urine Pharmacokinetic Concentrations |
| 14.2.1.1.1 | Excretion: MMV367 Ae(Urine) by Collection Period ( <units>) Summary Statistics: PK Analysis Set Part 1</units> |
| 14.2.1.1.2 | Excretion: MMV367 Cumulative Ae(Urine) ( <units>) Summary Statistics: PK Analysis Set Part 1</units> |
| 14.2.1.1.3 | Recovery: MMV367<br>%Ae(Urine) by Collection Period<br>Summary Statistics: PK Analysis Set<br>Part 1 |
| 14.2.1.1.4 | Recovery: MMV367<br>Cumulative %Ae(Urine)<br>Summary Statistics: PK Analysis Set<br>Part 1 |
| | Plasma Pharmacokinetic Concentrations |
| 14.2.1.1.5 | Plasma Pharmacokinetic Concentrations: MMV367<(units)> Summary Statistics: <pk analysis="" pk="" set="" subset=""> Part 1</pk> |
| 14.2.1.2.1 | Plasma Pharmacokinetic Concentrations: MMV367<(units)> Summary Statistics: <pk analysis="" pk="" set="" subset=""> Part 2</pk> |
| 14.2.1.2.3 | Plasma Pharmacokinetic Concentrations: MMV367<(units)> Summary Statistics: <pk analysis="" pk="" set="" subset=""> Part 3</pk> |
| | Plasma Pharmacokinetic Parameters |
| 14.2.2.1.1 | Plasma Pharmacokinetic Parameters: MMV367<br>Summary Statistics: <pk analysis="" pk="" set="" subset=""><br/>Part 1</pk> |
| 14.2.2.1.2 | Plasma Pharmacokinetic Parameters: MMV367<br>Summary Statistics: <pk analysis="" pk="" set="" subset=""><br/>Part 2</pk> |
| 14.2.2.1.3 | Plasma Pharmacokinetic Parameters: MMV367<br>Summary Statistics: <pk analysis="" pk="" set="" subset=""><br/>Part 3</pk> |
| 14.2.2.2.1 | Plasma Pharmacokinetic Parameters: MMV367<br>Statistical Analysis Results – Assessment of Dose Proportionality: <pk<br>Analysis Set/PK Analysis Subset&gt;<br/>Part 1</pk<br> |

| Table<br>Number | Table Title |
|---|---|
| 14.2.2.2.2 | Plasma Pharmacokinetic Parameters: MMV367<br>Statistical Analysis Results – Assessment of Food Effect: <pk analysis<br="">Set/PK Analysis Subset&gt;<br/>Part 2</pk> |
| 14.2.2.2.3 | Plasma Pharmacokinetic Parameters: MMV367<br>Statistical Analysis Results – Assessment of Dose Proportionality: <pk<br>Analysis Set/PK Analysis Subset&gt;<br/>Part 3</pk<br> |
| | Adverse Events |
| 14.3.1.1 | Overall Summary of Treatment-Emergent Adverse Events Summary Statistics: Safety Analysis Set Part 1 |
| 14.3.1.2 | Treatment-Emergent Adverse Events By MedDRA System Organ Class and Preferred Term Summary Statistics: Safety Analysis Set Part 1 |
| 14.3.1.3 | Treatment-Emergent Adverse Events By MedDRA System Organ Class, Preferred Term and Severity Summary Statistics: Safety Analysis Set Part 1 |
| 14.3.1.4 | Treatment-Emergent Adverse Events By MedDRA System Organ Class, Preferred Term and Relationship to IMP Summary Statistics: Safety Analysis Set Part 1 |
| 14.3.1.5 | Treatment-Emergent Adverse Events Related to IMP By MedDRA System Organ Class and Preferred Term Summary Statistics: Safety Analysis Set Part 1 |
| 14.3.1.6 | Serious Adverse Events By MedDRA System Organ Class and Preferred Term Summary Statistics: Safety Analysis Set Part 1 |
| 14.3.2.1 | Overall Summary of Treatment-Emergent Adverse Events<br>Summary Statistics: Safety Analysis Set<br>Part 2 |
| 14.3.2.2 | Treatment-Emergent Adverse Events By MedDRA System Organ Class and Preferred Term Summary Statistics: Safety Analysis Set Part 2 |
| 14.3.2.3 | Treatment-Emergent Adverse Events By MedDRA System Organ Class, Preferred Term and Severity Summary Statistics: Safety Analysis Set Part 2 |

| Table<br>Number | Table Title |
|---|---|
| 14.3.2.4 | Treatment-Emergent Adverse Events By MedDRA System Organ Class, Preferred Term and Relationship to IMP Summary Statistics: Safety Analysis Set Part 2 |
| 14.3.2.5 | Treatment-Emergent Adverse Events Related to IMP By MedDRA System Organ Class and Preferred Term Summary Statistics: Safety Analysis Set Part 2 |
| 14.3.2.6 | Serious Adverse Events By MedDRA System Organ Class and Preferred Term Summary Statistics: Safety Analysis Set Part 2 |
| 14.3.3.1 | Overall Summary of Treatment-Emergent Adverse Events Summary Statistics: Safety Analysis Set Part 3 |
| 14.3.3.2 | Treatment-Emergent Adverse Events By MedDRA System Organ Class and Preferred Term Summary Statistics: Safety Analysis Set Part 3 |
| 14.3.3.3 | Treatment-Emergent Adverse Events By MedDRA System Organ Class, Preferred Term and Severity Summary Statistics: Safety Analysis Set Part 3 |
| 14.3.3.4 | Treatment-Emergent Adverse Events By MedDRA System Organ Class, Preferred Term and Relationship to IMP Summary Statistics: Safety Analysis Set Part 3 |
| 14.3.3.5 | Treatment-Emergent Adverse Events Related to IMP By MedDRA System Organ Class and Preferred Term Summary Statistics: Safety Analysis Set Part 3 |
| 14.3.3.6 | Serious Adverse Events By MedDRA System Organ Class and Preferred Term Summary Statistics: Safety Analysis Set Part 3 |
| | Laboratory Results |
| 14.4.1.1 | Haematology and Coagulation Summary Statistics: Safety Analysis Set Part 1 Parameter <units></units> |

| Table<br>Number | Table Title |
|---|---|
| 14.4.1.2 | Haematology and Coagulation Shift Analysis: Safety Analysis Set Part 1 Parameter <units></units> |
| 14.4.1.3 | Clinical Chemistry Summary Statistics: Safety Analysis Set Part 1 Parameter <units></units> |
| 14.4.1.4 | Clinical Chemistry Shift Analysis: Safety Analysis Set Part 1 Parameter <units></units> |
| 14.4.2.1 | Haematology and Coagulation Summary Statistics: Safety Analysis Set Part 2 Parameter <units></units> |
| 14.4.2.2 | Haematology and Coagulation Shift Analysis: Safety Analysis Set Part 2 Parameter <units></units> |
| 14.4.2.3 | Clinical Chemistry Summary Statistics: Safety Analysis Set Part 2 Parameter <units></units> |
| 14.4.2.4 | Clinical Chemistry Shift Analysis: Safety Analysis Set Part 2 Parameter <units></units> |
| 14.4.3.1 | Haematology and Coagulation Summary Statistics: Safety Analysis Set Parameter <units> Part 3</units> |
| 14.4.3.2 | Haematology and Coagulation Shift Analysis: Safety Analysis Set Part 3 Parameter <units></units> |
| 14.4.3.3 | Clinical Chemistry Summary Statistics: Safety Analysis Set Part 3 Parameter <units></units> |
| 14.4.3.4 | Clinical Chemistry Shift Analysis: Safety Analysis Set Part 3 Parameter <units></units> |

| Table<br>Number | Table Title |
|---|---|
| | Vital Signs and ECG Results |
| 14.5.1.1 | Vital Signs Summary Statistics: Safety Analysis Set Part 1 Parameter <units></units> |
| 14.5.2.1.1 | ECGs Summary Statistics: Safety Analysis Set Single 12-Lead Part 1 Parameter <units></units> |
| 14.5.2.1.2 | ECGs Summary Statistics: Safety Analysis Set Mean of Triplicate 12-Lead Part 1 Parameter <units></units> |
| 14.5.2.1.3 | ECGs<br>QTcB and QTcF Categorical Data<br>Summary Statistics: Safety Analysis Set<br>Part 1 |
| 14.5.1.2 | Vital Signs Summary Statistics: Safety Analysis Set Parameter <units> Part 2</units> |
| 14.5.2.2.1 | ECGs Summary Statistics: Safety Analysis Set Parameter <units> Single 12-Lead Part 2</units> |
| 14.5.2.2.2 | ECGs Summary Statistics: Safety Analysis Set Mean of Triplicate 12-Lead Parameter <units> Part 2</units> |
| 14.5.2.2.3 | ECGs<br>QTcB and QTcF Categorical Data<br>Summary Statistics: Safety Analysis Set<br>Part 2 |
| 14.5.1.3 | Vital Signs Summary Statistics: Safety Analysis Set Part 3 Parameter <units></units> |

| Table<br>Number | Table Title |
|---|---|
| 14.5.2.3.1 | ECGs Summary Statistics: Safety Analysis Set Parameter <units> Single 12-Lead Part 3</units> |
| 14.5.2.3.2 | ECGs Summary Statistics: Safety Analysis Set Parameter <units> Mean of Triplicate 12-Lead Part 3</units> |
| 14.5.2.3.3 | ECGs<br>QTcB and QTcF Categorical Data<br>Summary Statistics: Safety Analysis Set<br>Part 3 |
| | Other |
| 14.6.1.1 | Taste Assessment: Taste Aspects Summary Statistics: Taste Analysis Set Taste Test Aspect: <xxx> Part 1</xxx> |
| 14.6.1.2 | Taste Assessment: Overall Acceptability Summary Statistics: Taste Analysis Set Part 1 |


19 Index of Figures

| 19 Index of Figures | |
|---|---|
| Figure<br>Number | Figure Title |
| | Plasma Pharmacokinetic Concentrations: MMV367 |
| 14.2.3.1.1 | Plasma Pharmacokinetic Concentrations: MMV367 <units> Linear/Linear Scale Arithmetic Mean (± Arithmetic SD) Values: <pk analysis="" pk="" set="" subset=""> Part 1 Programming note: All treatments on the same plot (up to 5 profiles)</pk></units> |
| 14.2.3.1.2 | Plasma Pharmacokinetic Concentrations: MMV367 <units> Log10/Linear Scale Geometric Mean (×/÷Geometric SD) Values: <pk analysis="" pk="" set="" subset=""> Part 1 Programming note: All treatments on the same plot (up to 5 profiles)</pk></units> |
| 14.2.3.1.3 | Plasma Pharmacokinetic Concentrations: MMV367 <units> Linear/Linear Scale Spaghetti Plots of All Individual Values: <pk analysis="" pk="" set="" subset=""> Part 1</pk></units> |
| 14.2.3.1.4 | Plasma Pharmacokinetic Concentrations: MMV367 <units> Log10/Linear Scale Spaghetti Plots of All Individual Values: <pk analysis="" pk="" set="" subset=""> Part 1</pk></units> |
| 14.2.3.2.1 | Plasma Pharmacokinetic Concentrations: MMV367 <units> Linear/Linear Scale Arithmetic Mean (± Arithmetic SD) Values: <pk analysis="" pk="" set="" subset=""> Part 2 Programming note: Fed and Fasted treatments on the same plot (2 profiles)</pk></units> |
| 14.2.3.2.2 | Plasma Pharmacokinetic Concentrations: MMV367 <units> Log10/Linear Scale Geometric Mean (×/÷Geometric SD) Values: <pk analysis="" pk="" set="" subset=""> Part 2 Programming note: Fed and Fasted treatments on the same plot (2 profiles)</pk></units> |
| 14.2.3.2.3 | Plasma Pharmacokinetic Concentrations: MMV367 <units> Linear/Linear Scale Spaghetti Plots of All Individual Values: <pk analysis="" pk="" set="" subset=""> Part 2</pk></units> |

| Figure<br>Number | Figure Title |
|---|---|
| 14.2.3.2.4 | Plasma Pharmacokinetic Concentrations: MMV367 <units> Log10/Linear Scale Spaghetti Plots of All Individual Values: <pk analysis="" pk="" set="" subset=""> Part 2</pk></units> |
| 14.2.3.2.5 | Plasma Pharmacokinetic Concentrations: MMV367 <units> Linear/Linear Scale Individual Values for Participant <xxx>: <pk analysis="" pk="" set="" subset=""> Part 2 Programming note: Fed and Fasted treatments on the same plot (2 profiles</pk></xxx></units> |
| 14.2.3.2.6 | Plasma Pharmacokinetic Concentrations: MMV367 <units> Log10/Linear Scale Individual Values for Participant <xxx>: <pk analysis="" pk="" set="" subset=""> Part 2 Fed and Fasted treatments on the same plot (2 profiles)</pk></xxx></units> |
| 14.2.3.2.7 | Plasma Pharmacokinetic Values < Cmax>: MMV367 < units> Linear/Linear Scale Scatter Plot: < PK Analysis Set/PK Analysis Subset> Part 2 |
| 14.2.3.3.1 | Plasma Pharmacokinetic Concentrations: MMV367 <units> Linear/Linear Scale Arithmetic Mean (± Arithmetic SD) Values: <pk analysis="" pk="" set="" subset=""> Part 3 Programming note: All treatments on the same plot – separate plots for Day 1 and Day 3</pk></units> |
| 14.2.3.3.2 | Plasma Pharmacokinetic Concentrations: MMV367 <units> Log10/Linear Scale Geometric Mean (×/÷Geometric SD) Values: <pk analysis="" pk="" set="" subset=""> Part 3 Programming note: All treatments on the same plot – separate plots for Day 1 and Day 3</pk></units> |
| 14.2.3.3.3 | Plasma Pharmacokinetic Concentrations: MMV367 <units> Linear/Linear Scale Arithmetic Mean (± Arithmetic SD) Values: <pk analysis="" pk="" set="" subset=""> Part 3 Programming note: Day 1 and Day 3 on the same plot— separate plots for treatments</pk></units> |

| Figure<br>Number | Figure Title |
|---|---|
| 14.2.3.3.4 | Plasma Pharmacokinetic Concentrations: MMV367 <units> Log10/Linear Scale Geometric Mean (×/÷Geometric SD) Values: <pk analysis="" pk="" set="" subset=""> Part 3 Programming note: Day 1 and Day 3 on the same plot— separate plots for treatments</pk></units> |
| 14.2.3.3.5 | Plasma Pharmacokinetic Concentrations: MMV367 <units><br/>Linear/Linear Scale<br/>Spaghetti Plots of All Individual Values: <pk analysis="" analysis<br="" pk="" set="">Subset&gt;<br/><day><br/>Part 3</day></pk></units> |
| 14.2.3.3.6 | Plasma Pharmacokinetic Concentrations: MMV367 <units> Log10/Linear Scale Spaghetti Plots of All Individual Values: <pk analysis="" pk="" set="" subset=""> <day> Part 3</day></pk></units> |
| 14.2.3.3.7 | Plasma Pharmacokinetic Concentrations: MMV367 <units> Linear/Linear Scale Individual Values for Participant <xxx>: <pk analysis="" pk="" set="" subset=""> Day 1 Part 3 Programming note: Separate plots for Day 1 and Day 3</pk></xxx></units> |
| 14.2.3.3.8 | Plasma Pharmacokinetic Concentrations: MMV367 <units> Log10/Linear Scale Individual Values for Participant <xxx>: <pk analysis="" pk="" set="" subset=""> Day 1 Part 3 Programming note: Separate plots for Day 1 and Day 3</pk></xxx></units> |
| 14.2.3.3.9 | Plasma Pharmacokinetic Concentrations: MMV367 <units> Linear/Linear Scale Individual Values for Participant <xxx>: <pk analysis="" pk="" set="" subset=""> Day 1 and Day 3 Part 3 Programming note: Both Day 1 and Day 3 on the same plot</pk></xxx></units> |
| 14.2.3.3.10 | Plasma Pharmacokinetic Concentrations: MMV367 <units> Log10/Linear Scale Individual Values for Participant <xxx>: <pk analysis="" pk="" set="" subset=""> Day 1 and Day 3 Part 3 Programming note: Both Day 1 and Day 3 on the same plot</pk></xxx></units> |

| Figure<br>Number | Figure Title |
|---|---|
| | Statistical Figures |
| 14.2.4.1.1 | Plasma Pharmacokinetic Parameters: MMV367<br>Log10/Log10 Scale<br>Geometric Mean (×/÷ Geometric SD) Values by Dose: PK Analysis Set<br>Part 1<br><parameter (units)=""></parameter> |
| 14.2.4.1.2 | Plasma Pharmacokinetic Parameters: MMV367 Log10/Log10 Scale Individual Values by Dose with Fitted Regression Line: PK Analysis Set Part 1 <parameter (units)=""></parameter> |
| 14.2.4.1.3 | Taste Assessment Box Plot of Taste Scores by Dose: Taste Analysis Set Part 1 <taste aspect=""></taste> |
| 14.2.4.1.4 | Taste Assessment Bubble Plot of Taste Scores by Dose: Taste Analysis Set Part 1 <taste aspect=""></taste> |


20 Index of Listings

| 20 Index of | Listings |
|---|---|
| Listing<br>Number | Listing Title |
| | Participant Informed Consent and Completion/Withdrawal |
| 16.2.1.1 | Participant Informed Consent and Completion/Withdrawal Individual Values: All Enrolled Subjects Part 1 |
| 16.2.1.2 | Participant Informed Consent and Completion/Withdrawal Individual Values: All Enrolled Subjects Part 2 |
| 16.2.1.3 | Participant Informed Consent and Completion/Withdrawal Individual Values: All Enrolled Subjects Part 3 |
| | Protocol Deviations and Inclusion/Exclusion Criteria |
| 16.2.2.1.1 | Protocol Deviations<br>Individual Values: All Enrolled Subjects<br>Part 1 |
| 16.2.2.1.2 | Inclusion/Exclusion Criteria Individual Values: All Enrolled Subjects Part 1 |
| 16.2.2.2.1 | Protocol Deviations<br>Individual Values: All Enrolled Subjects<br>Part 2 |
| 16.2.2.2.2 | Inclusion/Exclusion Criteria Individual Values: All Enrolled Subjects Part 2 |
| 16.2.2.3.1 | Protocol Deviations<br>Individual Values: All Enrolled Subjects<br>Part 3 |
| 16.2.2.3.2 | Inclusion/Exclusion Criteria Individual Values: All Enrolled Subjects Part 3 |
| | Analysis Populations and Reasons for Exclusion |
| 16.2.3.1.1 | Analysis Populations and Reasons for Exclusion<br>Individual Values: All Enrolled Subjects<br>Part 1 |
| 16.2.3.1.2 | Analysis Sets and Analysis Subsets and Reasons for Exclusion Individual Values: All Enrolled Subjects Part 1 |
| 16.2.3.2.1 | Analysis Populations and Reasons for Exclusion<br>Individual Values: All Enrolled Subjects<br>Part 2 |

Number: DOC-101489 Version: 2.0 Status: Approved Approved Date: 19 Dec 2022 QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan

| Listing<br>Number | Listing Title |
|---|---|
| 16.2.3.2.2 | Analysis Sets and Analysis Subsets and Reasons for Exclusion Individual Values: All Enrolled Subjects Part 2 |
| 16.2.3.3.1 | Analysis Populations and Reasons for Exclusion Individual Values: All Enrolled Subjects Part 3 |
| 16.2.3.3.2 | Analysis Sets and Analysis Subsets and Reasons for Exclusion Individual Values: All Enrolled Subjects Part 3 |
| | Demographic and Baseline Characteristics |
| 16.2.4.1.1 | Demographics and Baseline Characteristics<br>Individual Values: All Enrolled Subjects<br>Part 1 |
| 16.2.4.1.2 | Lifestyle Details: Smoking History and Alcohol Consumption Individual Values: All Enrolled Subjects Part 1 |
| 16.2.4.1.3 | Medical/Surgical History<br>Individual Values: All Enrolled Subjects<br>Part 1 |
| 16.2.4.1.4 | Prior and Concomitant Medication<br>Individual Values: All Enrolled Subjects<br>Part 1 |
| 16.2.4.1.5 | Carbon Monoxide Breath Test<br>Individual Values: All Enrolled Subjects<br>Part 1 |
| 16.2.4.1.6 | Urine Drug Screen<br>Individual Values: All Enrolled Subjects<br>Part 1 |
| 16.2.4.1.7 | Alcohol Breath and Carbon Monoxide Test<br>Individual Values: All Enrolled Subjects<br>Part 1 |
| 16.2.4.1.8 | SARS-CoV-2 Antigen Test<br>Individual Values: All Enrolled Subjects<br>Part 1 |
| 16.2.4.1.9 | BDI-II Questionnaire<br>Individual Values: All Enrolled Subjects<br>Part 1 |
| 16.2.4.1.10 | Virology<br>Individual Values: All Enrolled Subjects<br>Part 1 |

| Listing<br>Number | Listing Title |
|---|---|
| 16.2.4.1.11 | Creatinine Clearance<br>Individual Values: All Enrolled Subjects<br>Part 1 |
| 16.2.4.1.12 | Follicle Stimulating Hormone<br>Individual Values: All Enrolled Female Subjects<br>Part 1 |
| 16.2.4.1.13 | Serum Pregnancy Test<br>Individual Values: All Enrolled Female Subjects<br>Part 1 |
| 16.2.4.1.14 | Urine Pregnancy Test<br>Individual Values: All Enrolled Female Subjects<br>Part 1 |
| 16.2.4.2.1 | Demographics and Baseline Characteristics<br>Individual Values: All Enrolled Subjects<br>Part 2 |
| 16.2.4.2.2 | Lifestyle Details: Smoking History and Alcohol Consumption Individual Values: All Enrolled Subjects Part 2 |
| 16.2.4.2.3 | Medical/Surgical History<br>Individual Values: All Enrolled Subjects<br>Part 12 |
| 16.2.4.2.4 | Prior and Concomitant Medication<br>Individual Values: All Enrolled Subjects<br>Part 2 |
| 16.2.4.2.5 | Carbon Monoxide Breath Test<br>Individual Values: All Enrolled Subjects<br>Part 2 |
| 16.2.4.2.6 | Urine Drug Screen<br>Individual Values: All Enrolled Subjects<br>Part 2 |
| 16.2.4.2.7 | Alcohol Breath and Carbon Monoxide Test<br>Individual Values: All Enrolled Subjects<br>Part 2 |
| 16.2.4.2.8 | SARS-CoV-2 Antigen Test<br>Individual Values: All Enrolled Subjects<br>Part 2 |
| 16.2.4.2.9 | BDI-II Questionnaire<br>Individual Values: All Enrolled Subjects<br>Part 2 |
| 16.2.4.2.10 | Virology<br>Individual Values: All Enrolled Subjects<br>Part 2 |

| Listing<br>Number | Listing Title |
|---|---|
| 16.2.4.2.11 | Creatinine Clearance<br>Individual Values: All Enrolled Subjects<br>Part 2 |
| 16.2.4.2.12 | Follicle Stimulating Hormone<br>Individual Values: All Enrolled Female Subjects<br>Part 2 |
| 16.2.4.2.13 | Serum Pregnancy Test<br>Individual Values: All Enrolled Female Subjects<br>Part 2 |
| 16.2.4.2.14 | Urine Pregnancy Test<br>Individual Values: All Enrolled Female Subjects<br>Part 2 |
| 16.2.4.2.15 | Body Weight<br>Individual Values: All Enrolled Subjects<br>Part 2 |
| 16.2.4.3.1 | Demographics and Baseline Characteristics<br>Individual Values: All Enrolled Subjects<br>Part 3 |
| 16.2.4.3.2 | Lifestyle Details: Smoking History and Alcohol Consumption Individual Values: All Enrolled Subjects Part 3 |
| 16.2.4.3.3 | Medical/Surgical History<br>Individual Values: All Enrolled Subjects<br>Part 3 |
| 16.2.4.3.4 | Prior and Concomitant Medication<br>Individual Values: All Enrolled Subjects<br>Part 3 |
| 16.2.4.3.5 | Carbon Monoxide Breath Test<br>Individual Values: All Enrolled Subjects<br>Part 3 |
| 16.2.4.3.6 | Urine Drug Screen<br>Individual Values: All Enrolled Subjects<br>Part 3 |
| 16.2.4.3.7 | Alcohol Breath and Carbon Monoxide Test<br>Individual Values: All Enrolled Subjects<br>Part 3 |
| 16.2.4.3.8 | SARS-CoV-2 Antigen Test<br>Individual Values: All Enrolled Subjects<br>Part 3 |
| 16.2.4.3.9 | BDI-II Questionnaire<br>Individual Values: All Enrolled Subjects<br>Part 3 |

Number: DOC-101489 Version: 2.0 Status: Approved Approved Date: 19 Dec 2022 QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan

| Listing<br>Number | Listing Title |
|---|---|
| 16.2.4.3.10 | Virology<br>Individual Values: All Enrolled Subjects<br>Part 3 |
| 16.2.4.3.11 | Creatinine Clearance<br>Individual Values: All Enrolled Subjects<br>Part 3 |
| 16.2.4.3.12 | Follicle Stimulating Hormone<br>Individual Values: All Enrolled Female Subjects<br>Part 3 |
| 16.2.4.3.13 | Serum Pregnancy Test<br>Individual Values: All Enrolled Female Subjects<br>Part 3 |
| 16.2.4.3.14 | Urine Pregnancy Test<br>Individual Values: All Enrolled Female Subjects<br>Part 3 |
| | Dosing Details and Meal Details |
| 16.2.5.1.1.1 | Dosing Details<br>Individual Values: All Enrolled Subjects<br>Part 1 |
| 16.2.5.1.1.2 | Meal Details<br>Individual Values: All Enrolled Subjects<br>Part 1 |
| 16.2.5.1.2.1 | Dosing Details<br>Individual Values: All Enrolled Subjects<br>Part 2 |
| 16.2.5.1.2.2 | Meal Details<br>Individual Values: All Enrolled Subjects<br>Part 2 |
| 16.2.5.1.3.1 | Dosing Details<br>Individual Values: All Enrolled Subjects<br>Part 3 |
| 16.2.5.1.3.2 | Meal Details<br>Individual Values: All Enrolled Subjects<br>Part 3 |
| | Urine Concentration Data |
| 16.2.5.2.1.1 | Urine Collection Details Individual Values: All Enrolled Subjects Part 1 |
| 16.2.5.2.1.2 | Excretion: MMV367 Ae(Urine) ( <units>) Part 1</units> |

| Listing<br>Number | Listing Title |
|---|---|
| 16.2.5.2.1.3 | Excretion: MMV367 Cumulative Ae(Urine) ( <units>) Part 1</units> |
| 16.2.5.2.1.4 | Excretion: MMV367 Cumulative %Ae(Urine) ( <units>) Part 1</units> |
| 16.2.5.2.1.5 | Recovery: MMV367<br>Cumulative %Ae(Urine)<br>Part 1 |
| 16.2.5.2.1.6 | Recovery: MMV367<br>Cumulative Ae(Urine) ( <units>)<br/>Part 1</units> |
| 16.2.5.2.1.7 | Recovery: MMV367<br>Cumulative %Ae(Urine) ( <units>)<br/>Part 1</units> |
| | Plasma Pharmacokinetic Concentration Data |
| 16.2.5.3.1.1 | Blood Sample Collection Details Pharmacokinetic Analysis, Metabolic Profiling and Pharmacogenetic Testing Individual Values: All Enrolled Subjects Part 1 |
| 16.2.5.3.1.2 | Plasma Pharmacokinetic Concentrations: MMV367 <units> Individual Values: All Enrolled Subjects Part 1</units> |
| 16.2.5.3.2.1 | Blood Sample Collection Details Pharmacokinetic Analysis, Metabolic Profiling and Pharmacogenetic Testing Individual Values: All Enrolled Subjects Part 2 |
| 16.2.5.3.2.2 | Plasma Pharmacokinetic Concentrations: MMV367 <units> Individual Values: All Enrolled Subjects Part 2</units> |
| 16.2.5.3.3.1 | Blood Sample Collection Details Pharmacokinetic Analysis, Metabolic Profiling and Pharmacogenetic Testing Individual Values: All Enrolled Subjects Part 3 |
| 16.2.5.3.3.2 | Plasma Pharmacokinetic Concentrations: MMV367 <units> Individual Values: All Enrolled Subjects Part 3</units> |
| | Plasma Pharmacokinetic Parameter Data |
| 16.2.6.1 | Plasma Pharmacokinetic Parameters: MMV367<br>Individual Values: All Enrolled Subjects<br>Part 1 |

| Listing<br>Number | Listing Title |
|---|---|
| 16.2.6.2 | Plasma Pharmacokinetic Parameters: MMV367<br>Individual Values: All Enrolled Subjects<br>Part 2 |
| 16.2.6.3 | Plasma Pharmacokinetic Parameters: MMV367<br>Individual Values: All Enrolled Subjects<br>Part 3 |
| | Adverse Events |
| 16.2.7.1.1 | Pre-dose Adverse Events<br>Individual Values: All Enrolled Subjects<br>Part 1 |
| 16.2.7.1.2 | All Treatment-Emergent Adverse Events Individual Values: All Enrolled Subjects Part 1 |
| 16.2.7.1.3 | Serious Adverse Events<br>Individual Values: All Enrolled Subjects<br>Part 1 |
| 16.2.7.2.1 | Pre-dose Adverse Events<br>Individual Values: All Enrolled Subjects<br>Part 2 |
| 16.2.7.2.2 | All Treatment-Emergent Adverse Events Individual Values: All Enrolled Subjects Part 2 |
| 16.2.7.2.3 | Serious Adverse Events<br>Individual Values: All Enrolled Subjects<br>Part 2 |
| 16.2.7.3.1 | Pre-dose Adverse Events Individual Values: All Enrolled Subjects Part 3 |
| 16.2.7.3.2 | All Treatment-Emergent Adverse Events Individual Values: All Enrolled Subjects Part 3 |
| 16.2.7.3.3 | Serious Adverse Events<br>Individual Values: All Enrolled Subjects<br>Part 3 |
| | Laboratory Data |
| 16.2.8.1.1 | Blood Sample Collection Details for Laboratory Analysis<br>Individual Values: All Enrolled Subjects<br>Part 1 |
| 16.2.8.1.2 | Haematology and Coagulation<br>Individual Values: All Enrolled Subjects<br>Part 1 |

Number: DOC-101489 Version: 2.0 Status: Approved Approved Date: 19 Dec 2022 QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan

| Listing<br>Number | Listing Title |
|---|---|
| 16.2.8.1.3 | Haematology and Coagulation<br>Individual Values Outside the Reference Range: All Enrolled Subjects<br>Part 1 |
| 16.2.8.1.4 | Clinical Chemistry Individual Values: All Enrolled Subjects Part 1 |
| 16.2.8.1.5 | Clinical Chemistry Individual Values Outside the Reference Range: All Enrolled Subjects Part 1 |
| 16.2.8.1.6 | Urinalysis Sample Collection<br>Individual Values: All Enrolled Subjects<br>Part 1 |
| 16.2.8.1.7 | Urinalysis<br>Individual Values: All Enrolled Subjects<br>Part 1 |
| 16.2.8.1.8 | Urinalysis<br>Individual Values Outside the Reference Range: All Enrolled Subjects<br>Part 1 |
| 16.2.8.2.1 | Blood Sample Collection Details for Laboratory Analysis<br>Individual Values: All Enrolled Subjects<br>Part 2 |
| 16.2.8.2.2 | Haematology and Coagulation<br>Individual Values: All Enrolled Subjects<br>Part 2 |
| 16.2.8.2.3 | Haematology and Coagulation<br>Individual Values Outside the Reference Range: All Enrolled Subjects<br>Part 2 |
| 16.2.8.2.4 | Clinical Chemistry Individual Values: All Enrolled Subjects Part 2 |
| 16.2.8.2.5 | Clinical Chemistry Individual Values Outside the Reference Range: All Enrolled Subjects Part 2 |
| 16.2.8.2.6 | Urinalysis Sample Collection<br>Individual Values: All Enrolled Subjects<br>Part 2 |
| 16.2.8.2.7 | Urinalysis<br>Individual Values: All Enrolled Subjects<br>Part 2 |
| 16.2.8.2.8 | Urinalysis<br>Individual Values Outside the Reference Range: All Enrolled Subjects<br>Part 2 |

| Listing<br>Number | Listing Title |
|---|---|
| 16.2.8.3.1 | Blood Sample Collection Details for Laboratory Analysis<br>Individual Values: All Enrolled Subjects<br>Part 3 |
| 16.2.8.3.2 | Haematology and Coagulation<br>Individual Values: All Enrolled Subjects<br>Part 3 |
| 16.2.8.3.3 | Haematology and Coagulation<br>Individual Values Outside the Reference Range: All Enrolled Subjects<br>Part 3 |
| 16.2.8.3.4 | Clinical Chemistry Individual Values: All Enrolled Subjects Part 3 |
| 16.2.8.3.5 | Clinical Chemistry Individual Values Outside the Reference Range: All Enrolled Subjects Part 3 |
| 16.2.8.3.6 | Urinalysis Sample Collection<br>Individual Values: All Enrolled Subjects<br>Part 3 |
| 16.2.8.3.7 | Urinalysis<br>Individual Values: All Enrolled Subjects<br>Part 3 |
| 16.2.8.3.8 | Urinalysis<br>Individual Values Outside the Reference Range: All Enrolled Subjects<br>Part 3 |
| | Vital Signs and ECGs |
| 16.2.9.1.1.1 | Vital Signs<br>Individual Values: All Enrolled Subjects<br>Part 1 |
| 16.2.9.1.1.2 | Vital Signs<br>Individual Values Outside the Reference Range: All Enrolled Subjects<br>Part 1 |
| 16.2.9.1.2.1 | ECGs Individual Values: All Enrolled Subjects Part 1 (Programming note: The order of ECG parameters is to be as per Section 11.6) |
| 16.2.9.1.2.2 | ECGs Mean Values: All Enrolled Subjects Part 1 (Programming note: The order of ECG parameters is to be as per Section 11.6) |

Number: DOC-101489 Version: 2.0 Status: Approved Approved Date: 19 Dec 2022 QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan

| Listing<br>Number | Listing Title |
|---|---|
| 16.2.9.1.2.3 | ECGs<br>Individual Values Outside the Reference Range: All Enrolled Subjects<br>Part 1 |
| 16.2.9.1.2.4 | Telemetry Individual Values Outside the Reference Range: All Enrolled Subjects Part 1 |
| 16.2.9.2.1.1 | Vital Signs<br>Individual Values: All Enrolled Subjects<br>Part 2 |
| 16.2.9.2.1.2 | Vital Signs<br>Individual Values Outside the Reference Range: All Enrolled Subjects<br>Part 2 |
| 16.2.9.2.2.1 | ECGs Individual Values: All Enrolled Subjects Part 2 (Programming note: The order of ECG parameters is to be as per Section 11.6) |
| 16.2.9.2.2.2 | ECGs Mean Values: All Enrolled Subjects Part 2 (Programming note: The order of ECG parameters is to be as per Section 11.6) |
| 16.2.9.2.2.3 | ECGs<br>Individual Values Outside the Reference Range: All Enrolled Subjects<br>Part 2 |
| 16.2.9.2.2.4 | Telemetry Individual Values Outside the Reference Range: All Enrolled Subjects Part 2 |
| 16.2.9.3.1.1 | Vital Signs<br>Individual Values: All Enrolled Subjects<br>Part 3 |
| 16.2.9.3.1.2 | Vital Signs<br>Individual Values Outside the Reference Range: All Enrolled Subjects<br>Part 3 |
| 16.2.9.3.2.1 | ECGs Individual Values: All Enrolled Subjects Part 3 (Programming note: The order of ECG parameters is to be as per Section 11.6) |
| 16.2.9.3.2.2 | ECGs Mean Values: All Enrolled Subjects Part 3 (Programming note: The order of ECG parameters is to be as per Section 11.6) |

| Listing<br>Number | Listing Title |
|---|---|
| 16.2.9.3.2.3 | ECGs<br>Individual Values Outside the Reference Range: All Enrolled Subjects<br>Part 3 |
| | Other Data |
| 16.2.10.1.1 | Physical Examination Data<br>Individual Values: All Enrolled Subjects<br>Part 1 |
| 16.2.10.1.2 | Targeted Physical Examination Data<br>Individual Values: All Enrolled Subjects<br>Part 1 |
| 16.2.10.1.3 | Body Weight Data<br>Individual Values: All Enrolled Subjects<br>Part 1 |
| 16.2.10.1.3 | Taste Assessment Data Individual Values: All Enrolled Subjects <treatment> Part 1</treatment> |
| 16.2.10.2.1 | Physical Examination Data<br>Individual Values: All Enrolled Subjects<br>Part 2 |
| 16.2.10.2.2 | Targeted Physical Examination Data<br>Individual Values: All Enrolled Subjects<br>Part 2 |
| 16.2.10.3.1 | Physical Examination Data<br>Individual Values: All Enrolled Subjects<br>Part 3 |
| 16.2.10.3.2 | Targeted Physical Examination Data<br>Individual Values: All Enrolled Subjects<br>Part 3 |
| 16.2.10.3.3 | Body Weight Data<br>Individual Values: All Enrolled Subjects<br>Part 3 |
Number: DOC-101489 Version: 2.0 Status: Approved Approved Date: 19 Dec 2022 QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan

**Sponsor/Quotient Sciences Confidential** 

# 21 Mock Tables

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture Protocol: MMV\_MMV367\_21\_01

Page x of y

TABLE 14.1.1.1

Participant Disposition by Reason

Summary Statistics: All Enrolled Subjects

Part 1

Active Dose of MMV367

| | ALL PLACEBO (N=XX) n (%) | ALL ACTIVE (N=XX) n (%) | 100 mg<br>(N=XX)<br>n (%) | 300 mg<br>(N=XX)<br>n (%) | |
|---|---|---|---|---|---|
| Subjects randomised | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Subjects dosed | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Subjects completed | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Subjects discontinued | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Reason for discontinuation | | | | | |
| REASON 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| REASON 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| REASON 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| | <b></b> | ••• | ••• | | |
| <all categories="" on="" source=""></all> | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | ••• |

Note: The data in this table are presented in listing x.x

All subjects were planned to receive a single dose of either MMV367 or matching placebo

All Placebo/All Active relate to placebo or active subjects pooled over all cohorts, respectively

A participant may be discontinued for 1 reason only.

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: This table will be continued for all reasons for discontinuation as recorded on the source. If none of the subjects discontinued from the study early then reasons for discontinuation will not be populated in the summary table Percentages are based on the number of subjects enrolled

A similar table will be produced for Part 3, i.e., Table [14.1.1.3]

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture Protocol: MMV\_MMV367\_21\_01

TABLE 14.1.1.2

Participant Disposition by Reason

Summary Statistics: All Enrolled Subjects

Part 2

### Treatment Sequence

| | Fed/Fasted (N=X) n (%) | Fasted/Fed (N=X) n (%) | Overall<br>(N=X)<br>n (%) |
|---|---|---|---|
| Subjects randomised | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects dosed | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects completed | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects discontinued | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Reason for discontinuation | | | |
| REASON 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| REASON 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| REASON 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| <all categories="" on="" source=""></all> | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: The data in this table are presented in listing x.x

All subjects were to receive both treatments (i.e., Regimen 6 and Regimen 7) in a randomised manner over the two separate dosing occasions

A participant may be discontinued for one reason only

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Page x of y

Programming note: This table will be continued for all reasons for discontinuation as recorded on the source. If none of the subjects discontinued from the study early then reasons for discontinuation will not be populated in the summary table Percentages are based on the number of subjects enrolled in the respective sequence

Reporting and Analysis Plan MMV\_MMV367\_21\_01(QSC207031) Final v2.0 15 Dec 2022

This copy was downloaded by Claire \*\*Widso75ouf 128Dec 2022 at 16:25 GMT+00:00 Check validity before use

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture Protocol: MMV\_MMV367\_21\_01

Page x of y

TABLE 14.1.2.1.2 Analysis Populations Summary Statistics: All Enrolled Subjects

Part 1

Active Dose of MMV367

| | ALL PLACEBO (N=XX) n (%) | ALL ACTIVE (N=XX) n (%) | 100 mg<br>(N=XX)<br>n (%) | 300 mg<br>(N=XX)<br>n (%) | |
|---|---|---|---|---|---|
| Subjects in Safety Population Reasons for exclusion from Safety Population | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| <all categories="" from="" source=""></all> | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| | | | | | ••• |
| Subjects in Taste Population Reasons for exclusion from PK Population | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| <all categories="" from="" source=""></all> | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| | | | ••• | | ••• |
| Subjects in PK Population Reasons for exclusion from PD Population | | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| <all categories="" from="" source=""></all> | | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| | | ••• | | | ••• |

Note: The data in this table are presented in listing x.x

All subjects were planned to receive a single dose of either MMV367 or matching placebo

All Placebo/All Active relate to placebo or active subjects pooled over all cohorts, respectively

A participant may be excluded for more than 1 reason

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: Percentages are based on the number of subjects enrolled A similar table will be produced for Part 3, i.e., Table [14.1.2.3.2]

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture Protocol: MMV\_MMV367\_21\_01

Page x of y

TABLE 14.1.2.2.2 Analysis Populations

Summary Statistics: All Enrolled Subjects

Part 2

### Treatment Sequence

| | Fed/Fasted (N=X) n (%) | Fasted/Fed (N=X) n (%) | Overall (N=X) n (%) |
|---|---|---|---|
| Subjects in safety population Reason for exclusion from safety population | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| <pre><all categories="" listing="" on="" source=""></all></pre> | xx (xx.x)<br> | xx (xx.x)<br> | xx (xx.x)<br> |
| Subjects in PK population Reason for exclusion from PK population | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| <pre><all categories="" listing="" on="" source=""></all></pre> | xx (xx.x)<br> | xx (xx.x)<br> | xx (xx.x) |

Note: The data in this table are presented in listing x.x

All subjects were to receive both treatments (i.e., Regimen 6 and Regimen 7) in a randomised manner over the two separate dosing occasions

A participant may be excluded for more than one reason

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: Percentages are based on the number of subjects enrolled in the respective sequence

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture Protocol: MMV MMV367 21 01

Page x of y

TABLE 14.1.2.1.3 Safety Analysis Set

Summary Statistics: Safety Population

Part 1

Active Dose of MMV367

| | ALL PLACEBO<br>(N=XX)<br>n (%) | ALL ACTIVE (N=XX) n (%) | 100 mg<br>(N=XX)<br>n (%) | 300 mg<br>(N=XX)<br>n (%) |
|---|---|---|---|---|
| Subjects in safety analysis set | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Reasons for exclusion from safety analysis set<br><all categories="" from="" source=""></all> | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: The data in this table are presented in listing x.x

All subjects were planned to receive a single dose of either MMV367 or matching placebo

All Placebo/All Active relate to placebo or active subjects pooled over all cohorts, respectively

A participant may be excluded for more than 1 reason

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: A similar table will be produced for the Taste and PK Analysis Sets(and Subsets if applicable), i.e., Tables [14.1.2.1.4] and [14.1.2.1.5]. Each analysis set/subset will be a subset of their respective population and percentages will be based on number of subjects in each population

Similar tables will be produced for Part 3, i.e., Tables [14.1.2.3.3], [14.1.2.3.4]

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture Protocol: MMV MMV367 21 01 Page x of y

TABLE 14.1.2.2.3 Safety Analysis Set

Summary Statistics: Safety Population

Part 2

| | XX mg FAST (N=X) n (%) | XX mg FED (N=X) n (%) | Overall<br>(N=X)<br>n (%) |
|---|---|---|---|
| Subjects in safety analysis set Reasons for exclusion from safety analysis set | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| <pre><all categories="" from="" source=""></all></pre> | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: The data in this table are presented in listing x.x

All subjects were to receive both treatments (i.e., Regimen 6 and Regimen 7) in a randomised manner over the two separate dosing occasions

A participant may be excluded for more than one reason

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: A similar table will be produced for the PK Analysis Set (and Subset[s], if required), i.e., Table [14.1.2.2.4]

Each analysis set/subset will be a subset of their respective population and percentages

Each analysis set/subset will be a subset of their respective population and percentages

will be based on number of subjects in each population

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture Protocol: MMV\_MMV367\_21\_01

Page x of y

TABLE 14.1.3.1

Demographic and Baseline Characteristics Summary Statistics: Safety Analysis Set

Part 1

Active Dose of MMV367

| | | ALL PLACEBO (N=XX) | ALL ACTIVE (N=XX) | 100 mg<br>(N=XX) | 300 mg<br>(N=XX) | |
|---|---|---|---|---|---|---|
| Age (years) | n | xx | xx | xx | XX | |
| | Mean | XX.X | XX.X | XX.X | XX.X | |
| | SD | XX.X | XX.X | XX.X | XX.X | |
| | Median | XX.X | XX.X | XX.X | XX.X | |
| | Min | XX | XX | XX | XX | |
| | Max | XX | XX | XX | XX | |
| Ethnicity n(%) | <all categories="" on="" source=""></all> | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Race n(%) | <all categories="" on="" source=""></all> | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Sex n(%) | Male | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| | Female | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | ••• |
| Height (cm) | | | | | | |
| Weight (kg) | | | <b></b> | <del></del> | | |
| BMI (kg/m^2) | | | | | | |

Note: The data in this table are presented in listing x.x

All subjects were planned to receive a single dose of either MMV367 or matching placebo

All Placebo/All Active relate to placebo or active subjects pooled over all cohorts, respectively

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: This table will continue for all categories of ethnicity and race

Height, Weight and BMI will be summarised using the same descriptive statistics as Age If any values are missing, then a "missing" row will be included in the table, as applicable

A similar table will be produced for Part 3, i.e., Table [14.1.3.3]

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture Protocol: MMV\_MMV367\_21\_01

Page x of y

TABLE 14.1.3.2

Demographic and Baseline Characteristics Summary Statistics: Safety Analysis Set

Part 2

### Treatment Sequence

| | | Fed/Fasted (N=X) | Fasted/Fed (N=X) | Overall (N=X) |
|---|---|---|---|---|
| Age (years) | n<br>Maran | XX | XX | XX |
| | Mean | XX.XX | XX.XX | XX.XX |
| | SD | XX.XX | XX.XX | XX.XX |
| | Median | XX.XX | XX.XX | XX.XX |
| | Min | XX.X | XX.X | XX.X |
| | Max | XX.X | XX.X | XX.X |
| Ethnicity n(%) | <all categories="" on="" source=""></all> | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Race n(%) | <all categories="" on="" source=""></all> | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Sex n(%) | Male | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Female | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Height (cm) | | | | <b></b> |
| Weight (kg) | | | | <b></b> |
| BMI (kg/m^2) | | <del></del> | | |

Note: The data in this table are presented in listing x.x

All subjects were to receive both treatments (i.e., Regimen 6 and Regimen 7) in a randomised manner over the two separate dosing occasions

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: This table will continue for all categories of ethnicity and race

Height, Weight and BMI will be assessed using the same descriptive statistics as Age

If any values are missing, then a "missing" row will be included in the table, as applicable

Reporting and Analysis Plan MMV\_MMV367\_21\_01(QSC207031) Final v2.0 15 Dec 2022

This copy was downloaded by Claire Waigson1 of 128 Dec 2022 at 16:25 GMT+00:00 Check validity before use

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture Protocol: MMV MMV367 21 01 Page x of y

TABLE 14.1.4.1

Lifestyle Details: Smoking History and Alcohol Consumption

Summary Statistics: Safety Analysis Set

Part 1

Active Dose of MMV367

| | | (N= | PLACEBO<br>=XX)<br>(%) | (N | ACTIVE<br>(=XX) | (1) | 00 mg<br>I=XX)<br>1 (%) | (1) | 00 mg<br>N=XX)<br>n (%) | •••• | • • • • |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Does the participant smoke (1) | NO<br>EVIOUSLY | xx | xx (xx.x)<br>(xx.x) | xx | xx (xx.x)<br>(xx.x) | xx | xx (xx.x)<br>(xx.x) | xx | xx (xx.x)<br>(xx.x) | | |
| Alcohol Consumption (2) NO YE | NE<br>S: NOT EXCESSIVE | | (xx.x)<br>(xx.x) | | (xx.x)<br>(xx.x) | | (xx.x)<br>(xx.x) | | (xx.x)<br>(xx.x) | | |

Note: The data in this table are presented in listing x.x

- All subjects were planned to receive a single dose of either MMV367 or matching placebo
- All Placebo/All Active relate to placebo or active subjects pooled over all cohorts, respectively
- (1) Smoked or used e-cigarettes or nicotine replacement products in the last 12 months
- (2) Regular alcohol consumption (>21 units/week in males and >14 units/week in females)
- 1 unit = 1/2 pint beer, 25 mL of 40% spirit, 1.5 to 2 units = 125 mL glass of wine depending on type

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: A similar table will be produced for Part 3, i.e., Table [14.1.4.3]

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture Protocol: MMV\_MMV367\_21\_01

Page x of y

TABLE 14.1.4.2

Lifestyle Details: Smoking History and Alcohol Consumption

Summary Statistics: Safety Analysis Set

Part 2

#### Treatment Sequence

| | | Fed/Fasted (N=X) | | sted/Fed<br>(N=X) | | verall<br>(N=X) |
|---|---|---|---|---|---|---|
| Does the participant smoke? (1) NO PREVIOUSLY | xx | xx (xx.<br>(xx.x) | x)<br>xx | xx (xx.<br>(xx.x) | x) | xx (xx.x)<br>(xx.x) |
| Alcohol Consumption (2) NONE YES: NOT REGULA | | (xx.x)<br>(xx.x) | XX<br>XX | (xx.x)<br>(xx.x) | xx<br>xx | (xx.x)<br>(xx.x) |

Note: The data in this table are presented in listing x.x

- All subjects were to receive both treatments (i.e., Regimen 6 and Regimen 7) in a randomised manner over the two separate dosing occasions
- (1) Smoked or used e-cigarettes or nicotine replacement products in the last 12 months
- (2) Regular alcohol consumption (>21 units/week in males and >14 units/week in females)
- 1 unit = 1/2 pint beer, 25 mL of 40% spirit, 1.5 to 2 units = 125 mL glass of wine depending on type

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM


Medicines for Malaria Venture Protocol: MMV\_MMV367\_21\_01

Page x of y

TABLE 14.1.5.1 Extent of Exposure

Summary Statistics: Safety Analysis Set

Part 1

| Treatment | Subjects Dosed (N=XX) n (%) |
|-------------|-----------------------------|
| ALL PLACEBO | xx (xx.x) |
| ALL ACTIVE | xx (xx.x) |
| 100 mg | xx (xx.x) |

Note: The data in this table are presented in listing x.x

All subjects were planned to receive a single dose of either MMV367 or matching placebo

All Placebo/All Active relate to placebo or active subjects pooled over all cohorts, respectively

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM


Medicines for Malaria Venture Protocol: MMV\_MMV367\_21\_01

Page x of y

TABLE 14.1.5.2 Extent of Exposure

Summary Statistics: Safety Analysis Set

Part 2

Subjects Dosed (N=X)n (%) Treatment XX mg FAST xx (xx.x) XX mg FED xx (xx.x)

Note: The data in this table are presented in listing x.x

All subjects were to receive both treatments (i.e., Regimen 6 and Regimen 7) in a randomised manner over the two separate dosing occasions

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX DDMMMYYYY HH:MM


Medicines for Malaria Venture Protocol: MMV\_MMV367\_21\_01

Page x of y

TABLE 14.1.5.3.1

Extent of Exposure: Subjects Dosed by Day Summary Statistics: Safety Analysis Set

Part 3

| Day | ALL PLACEBO<br>(N=xx)<br>n (%) | XX mg (N=xx) n (%) | XX mg<br>(N=xx)<br>n (%) | XX mg<br>(N=xx)<br>n (%) |
|---|---|---|---|---|
| DAY 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| DAY 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: The data in this table are presented in listing x.x

All subjects were planned to receive a single dose of either MMV367 or matching placebo over 3 days All Placebo/All Active relate to placebo or active subjects pooled over all cohorts, respectively

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture Protocol: MMV\_MMV367\_21\_01

Page x of y

TABLE 14.2.1.1.1 Excretion: MM367

Ae(Urine) by Collection Period <(units)>Summary Statistics: PK Analysis Set

Part 1

MMV367 (N=XX)

| Collection Period | n | Mean | SD | CV% | Median | Min | Max |
|---|---|---|---|---|---|---|---|
| PRE-DOSE | 1717 | xx.xx | | | | xx.x | |
| TIME() - TIME1 | XX | | XX.XX | XX.X | XX.XX | | XX.X |
| | XX | XX.XX | XX.XX | XX.X | XX.XX | XX.X | XX.X |
| TIME1 - TIME2 | XX | XX.XX | XX.XX | XX.X | XX.XX | XX.X | XX.X |
| TIME2 - TIME3 | XX | XX.XX | XX.XX | XX.X | XX.XX | XX.X | XX.X |
| <all intervals="" other="" time=""></all> | XX | XX.XX | XX.XX | XX.X | XX.XX | XX.X | XX.X |

Note: The data in this table are presented in listing x.x

All subjects were planned to receive a single dose of either MMV367 or matching placebo
All Placebo/All Active relate to placebo or active subjects pooled over all cohorts, respectively
Where a participant has failed to void or has a ND concentration over a particular collection interval, the amount

excreted (Ae) has been set to zero

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

(Programming Note: This table will be continued for all collection periods

A similar table will be produced for:

• %Ae(Urine) (Recovery), i.e., Table [14.2.1.1.3]

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture Protocol: MMV\_MMV367\_21\_01

Page x of y

TABLE 14.2.1.1.2 Excretion: MMV367

Cumulative Ae(Urine) <(units)>
Summary Statistics: PK Analysis Set

Part 1

MMV367 (N=XX)

| Collection Period | | Mean | SD | CV% | Median | Min | Max |
|---|---|---|---|---|---|---|---|
| PRE-DOSE | XX | XX.XX | XX.XX | XX.X | XX.XX | XX.X | XX.X |
| TIMEO - TIME1 | XX | XX.XX | XX.XX | XX.X | XX.XX | XX.X | XX.X |
| TIMEO - TIME2 | XX | XX.XX | XX.XX | XX.X | XX.XX | XX.X | XX.X |
| TIMEO - TIME3 | XX | XX.XX | XX.XX | XX.X | XX.XX | XX.X | XX.X |
| ••• | | | | | | | |
| <all intervals="" other="" time=""></all> | XX | XX.XX | XX.XX | XX.X | XX.XX | XX.X | XX.X |

Note: The data in this table are presented in listing x.x

All subjects were planned to receive a single dose of either MMV367 or matching placebo

All Placebo/All Active relate to placebo or active subjects pooled over all cohorts, respectively

PROGRAM PATH: X:\~\QSC205477\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

(Programming note: This table will be continued for all collection periods. If required, as a result of early withdrawal or varying follow-up periods, this table will be produced using the LOCF approach. A similar table will be produced for • Cumulative %Ae(Urine) (Recovery), i.e., Table [14.2.1.1.4]

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture Protocol: MMV MMV367 21 01

Page x of y

TABLE 14.2.1.1.5

Plasma Pharmacokinetic Concentrations: MMV367(<units>)
Summary Statistics: <PK Analysis Set/PK Analysis Subset>

Part 1

| | Arithmetic (1) | | | | | | | | | Geometric (2) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Time Point | n | n# | Mean | SD | CV% | Median | Min | Max | Mean | SD | CV% |
| 100 mg | PRE-DOSE | xx | XX | xx.xx | xx.xx | xx.x | xx.xx | xx.x | XX.X | NC | NC | NC |
| (N=XX) | TIMEPOINT 1 | XX | XX | XX.XX | XX.XX | XX.X | XX.XX | XX.X | XX.X | XX.XX | XX.XX | XX.X |
| | TIMEPOINT 2 | XX | XX | xx.xx | XX.XX | XX.X | XX.XX | XX.X | XX.X | XX.XX | XX.XX | XX.X |
| | | ••• | | | | | | ••• | | | | |
| 300 mg | PRE-DOSE | xx | XX | xx.xx | xx.xx | xx.x | xx.xx | XX.X | XX.X | NC | NC | NC |
| (N=XX) | TIMEPOINT 1 | XX | XX | XX.XX | XX.XX | XX.X | XX.XX | XX.X | XX.X | XX.XX | XX.XX | XX.X |
| | TIMEPOINT 2 | XX | XX | XX.XX | XX.XX | XX.X | XX.XX | XX.X | XX.X | XX.XX | XX.XX | XX.X |
| | | | | ••• | | | | | ••• | | ••• | |

Note: The data in this table are presented in listing x.x

- All subjects were planned to receive a single dose of either MMV367 or matching placebo
- All Placebo/All Active relate to placebo or active subjects pooled over all cohorts, respectively
- n# indicates the number of subjects with a BLQ value recorded at the time point indicated
- (1) For arithmetic summary statistics, concentration values reported as BLQ have been set to zero
- (2) For calculation of geometric summary statistics, values reported as BLQ have been set to  $\frac{1}{2}$  × LLOQ, except for pre-dose values which will not be summarised. The LLOQ value was <value, units>

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: This table will be continued for all treatments and time points

Similar tables will be produced for Part 2 i.e., Table [14.2.1.2.1] and Part 3 i.e., [14.2.1.2.3],

with a column for Visit included before time point column.

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture Protocol: MMV MMV367 21 01

Page x of y

TABLE 14.2.2.1.1

Plasma Pharmacokinetic Parameters: MMV367

Summary Statistics: <PK Analysis Set/PK Analysis Subset>

Part 1

| Treatment | Statistic | Parameter 1 (units) | Parameter 2 (units) | Parameter 3 (units) | All Other PK Parameters (units) |
|---|---|---|---|---|---|
| | | | | | <br><del></del> |
| 100 mg | n | XX | XX | XX | <br>XX |
| (N=XX) | Mean | XX.X | XX.X | XX.X | <br>XX.X |
| | SD | XX.X | XX.X | XX.X | <br>XX.X |
| | CV% | XX.X | XX.X | XX.X | <br>XX.X |
| | Median | XX.X | XX.X | XX.X | <br>xx.x |
| | Min | XX | XX | XX | <br>XX |
| | Max | XX | XX | XX | <br>XX |
| | Geometric Mean | XX.X | XX.X | XX.X | <br>XX.X |
| | Geometric SD | XX.X | XX.X | XX.X | <br>xx.x |
| | Geometric CV% | XX.X | XX.X | XX.X | <br>xx.x |
| 300 mg | | | | | <br> |
| (N=XX) | | | | ••• | <br> |
| | <b></b> | | | | <br> |

Note: The data in this table are presented in listing x.x

The LLOQ value was <value, units

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: This table will be continued for all treatments and PK parameters

Similar tables will be produced for Part 2 i.e., Table [14.2.2.1.2] and Part 3, i.e., Table [14.2.2.1.3]

with a column for Visit included before statistic column.

Check validity before use

All subjects were planned to receive a single dose of either MMV367 or matching placebo

All Placebo/All Active relate to placebo or active subjects pooled over all cohorts, respectively

For concentration parameters, BLQ values will be set to 0 for arithmetic statistics and to ½ x LLQQ for geometric statistics>

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture Protocol: MMV MMV367 21 01

Page x of y

TABLE 14.2.2.2.1

Plasma Pharmacokinetic Parameters: MMV367

Statistical Analysis Results - Assessment of Dose Proportionality: <PK Analysis Set/PK Analysis Subset> Part 1

Active Dose of MMV367

| PK<br>Parameter | | 100 mg<br>(N=XX) | 300 mg<br>(N=XX) | 750mg<br>(N=XX) | 1500mg<br>(N=XX) | 2000mg<br>(N=XX) |
|---|---|---|---|---|---|---|
| Cmax (units) | n | XX | XX | XX | XX | xx |
| | Geometric Mean | XX.X | XX.X | XX.X | XX.X | xx.x |
| | ß (90% CI) | | | X.XX | (x.xx | x.xx) |
| | 2^B (90% CI) | | | X.XX | (x.xx | x.xx) |
| AUC (0-last) (units) | n | XX | XX | XX | XX | XX |
| | Geometric Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | ß (90% CI) | | | X.XX | (x.xx | x.xx) |
| | 2^B (90% CI) | | | X.XX | (x.xx | x.xx) |
| AUC (0-inf) (units) | n | XX | xx | XX | XX | xx |
| | Geometric Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | ß (90% CI) | | | X.XX | (x.xx | x.xx) |
| | 2^B (90% CI) | | | X.XX | (x.xx | x.xx) |

Note: The data in this table are presented in listing x.x

All subjects were planned to receive a single dose of either MMV367 or matching placebo over 3 days All Placebo/All Active relate to placebo or active subjects pooled over all cohorts, respectively

Results obtained from log-transformed PK parameters using a power model

The model includes a term for log dose fitted as a fixed effect

The geometric means presented are the same as the geometric means presented in Table [14.2.x.x]. N = total number of subjects in dose group, n = number of subjects with non-missing, valid data,  $\beta$  (ie the slope parameter) and its 90% CI are a measure of dose proportionality,  $2^{\beta}$  represents the increase in exposure for a 2-fold increase in dose Dose proportionality can be concluded if the 90% CI for  $\beta$  lie entirely within the critical region (x.xx, x.xx)

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Status: Approved Date: 19 Dec 2022 Number: DOC-101489 Version: 2.0

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture Protocol: MMV MMV367 21 01

Page x of y

TABLE 14.2.2.2.2

Plasma Pharmacokinetic Parameters: MMV367

Statistical Analysis Results - Assessment of Food Effect: <PK Analysis Set/PK Analysis Subset>

XX ma FED

Part 2

| | 2: | (N=XX) | _ | | | | | |
|---|---|---|---|---|---|---|---|---|
| Parameter | n | Adj Geo<br>Mean<br>(1) | n | Adj Geo<br>Mean<br>(1) | Ratio (%) | 90% CI<br>(3) | P-value<br>(4) | CVw (%)<br>(5) |
| Cmax (units) | xx | xx.xx | xx | xx.xx | xx.xx | (xx.xx, xx.xx) | 0.xxx | xx.xxx |
| AUC(0-last) (units) | xx | xx.xx | XX | xx.xx | XX.XX | (xx.xx, xx.xx) | 0.xxx | xx.xx |
| AUC(0-inf) (units) | XX | XX.XX | XX | xx.xx | XX.XX | (xx.xx, xx.xx) | 0.xxx | XX.XXX |

Note: The data in this table are presented in listing x.x

XX mg FAST

All subjects were to receive both treatments (i.e., Regimen 6 and Regimen 7) in a randomised manner over the two separate dosing occasions

Results obtained from mixed effects model of natural log transformed PK parameters including terms for fed/fasted Status, and period fitted as fixed effects and participant as a random effect

(1) Adj geo mean = adjusted geometric mean from model (2) Ratio of adj geo means with comparison presented as test/reference (3) CI = confidence interval for ratio of adj geo means (4) p-value from two-sided test (null hypothesis of no difference) (5) CVw = Intra-participant variability

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM


Medicines for Malaria Venture Protocol: MMV\_MMV367\_21\_01

Page x of y

TABLE 14.3.1.1

Overall Summary of Treatment-Emergent Adverse Events

Summary Statistics: Safety Analysis Set

Part 1

Active Dose of MMV367

| | | ALL PLACEBO (N=XX) | | | ALL ACTIVE (N=XX) | | | 100 mg<br>(N=XX) | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Event | | n(%) | E | | n(%) | E | | n (%) | E | |
| TEAEs | xx | (xx.x) | xx | XX | (xx.x) | xx | XX | (xx.x) | xx | |
| Severe TEAEs | xx | (xx.x) | xx | XX | (xx.x) | xx | XX | (xx.x) | XX | ••• |
| IMP-related TEAEs | xx | (xx.x) | xx | XX | (xx.x) | xx | XX | (xx.x) | XX | ••• |
| Serious TEAEs | хх | (xx.x) | XX | XX | (xx.x) | xx | XX | (xx.x) | XX | |
| TEAEs leading to participant withdrawal | | xx (xx.x) | | XX | xx (xx.x) | | XX | xx (xx.x) | ) | XX |
| TEAEs leading to death | XX | (xx.x) | XX | XX | (xx.x) | XX | XX | (xx.x) | XX | |

Note: The data in this table are presented in listing x.x

All subjects were planned to receive a single dose of either MMV367 or matching placebo

All Placebo/All Active relate to placebo or active subjects pooled over all cohorts, respectively

E = Total Number of Events

TEAEs are coded using MedDRA vXX.X

n is the number of subjects reporting at least one event

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: A similar table will be produced for Part 3, i.e., Table [14.3.3.1]


Medicines for Malaria Venture Protocol: MMV\_MMV367\_21\_01

Page x of y

TABLE 14.3.2.1

Overall Summary of Treatment-Emergent Adverse Events

Summary Statistics: Safety Analysis Set

Part 2

| | XX mg FA<br>(N=X) | AST | XX mg FI<br>(N=X) | ED | Overall<br>(N=X) | |
|---|---|---|---|---|---|---|
| Event | n (%) | E | n(%) | E | n (%) | E |
| TEAEs | xx (xx.x) | xx | xx (xx.x) | XX | xx (xx.x) | XX |
| Severe TEAE | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| IMP-related TEAEs | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| Serious TEAE | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| TEAE leading to participant withdrawal | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| TEAE leading to death | xx (xx.x) | xx | xx (xx.x) | XX | xx (xx.x) | XX |

Note: The data in this table are presented in listing x.x

All subjects were to receive both treatments (i.e., Regimen 6 and Regimen 7) in a randomised manner over the two separate dosing occasions

E = Total Number of Events

TEAEs are coded using MedDRA vXX.X

n is the number of subjects reporting at least one event

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture Protocol: MMV MMV367 21 01

Page x of y

TABLE 14.3.1.2

Treatment-Emergent Adverse Events

By MedDRA System Organ Class and Preferred Term

Summary Statistics: Safety Analysis Set

Active Dose of MMV367

| System Organ Class | | ALL PLACEBO (N=XX) | | | 100 m<br>(N=XX | | |
|---|---|---|---|---|---|---|---|
| Preferred Term | n(%) | E | n (%) | E | n (%) | E | ••••• |
| TEAEs | xx (xx.x) | xx | xx (xx.x) | XX | xx (xx.x) | XX | |
| SYSTEM ORGAN CLASS 1 | xx (xx.x) | xx | xx (xx.x) | XX | xx (xx.x) | xx | |
| PREFERRED TERM 1 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | |
| PREFERRED TERM 2 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | |
| etc | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | |
| SYSTEM ORGAN CLASS 2 | xx (xx.x) | XX | xx (xx.x) | xx | xx (xx.x) | xx | |
| PREFERRED TERM 1 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | |
| PREFERRED TERM 2 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | |
| etc | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | |

Note: The data in this table are presented in listing x.x

All subjects were planned to receive a single dose of either MMV367 or matching placebo

All Placebo/All Active relate to placebo or active subjects pooled over all cohorts, respectively

E = Total Number of Events

TEAEs are coded using MedDRA vXX.X and are presented in descending order of frequency

Subjects experiencing more than one TEAE within a treatment are counted only once for number of subjects but will be counted more than once for number of events. Subjects experiencing more than one TEAE within

a treatment are counted only once within each SOC and PT

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: This table will be continued for all SOC and PT

A similar table will be produced for Part 3, i.e., Table [14.3.3.2]

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture Protocol: MMV MMV367 21 01

Page x of y

TABLE 14.3.2.2
Treatment-Emergent Adverse Events
By MedDRA System Organ Class and Preferred Term
Summary Statistics: Safety Analysis Set
Part 2

| | | XX mg | | XX mg FED<br>(N=X) | | | Overall<br>(N=X) | | |
|---|---|---|---|---|---|---|---|---|---|
| | | n(%) | E | | n (%) | E | | n(%) | E |
| TEAEs | xx | (xx.x) | xx | xx | (xx.x) | xx | xx | (xx.x) | xx |
| SYSTEM ORGAN CLASS | 1 xx | (xx.x) | xx | XX | (xx.x) | xx | XX | (xx.x) | XX |
| PREFERRED TERM 1 | L xx | (xx.x) | XX | XX | (xx.x) | XX | XX | (xx.x) | XX |
| PREFERRED TERM 2 | 2 xx | (xx.x) | XX | XX | (xx.x) | XX | XX | (xx.x) | XX |
| etc | | | ••• | | | ••• | | | |
| SYSTEM ORGAN CLASS | 2 xx | (xx.x) | xx | XX | (xx.x) | xx | XX | (xx.x) | XX |
| PREFERRED TERM 1 | L xx | (xx.x) | XX | XX | (xx.x) | XX | XX | (xx.x) | XX |
| PREFERRED TERM 2 | 2 xx | (xx.x) | XX | XX | (xx.x) | XX | XX | (xx.x) | XX |
| etc | | | | | | | | | |

Note: The data in this table are presented in listing x.x

All subjects were to receive both treatments (i.e., Regimen 6 and Regimen 7) in a randomised manner over the two separate dosing occasions

E = Total Number of Events

TEAEs are coded using MedDRA vXX.X and are presented in descending order of frequency Subjects experiencing more than one TEAE within a treatment are counted only once for number of subjects but will be counted more than once for number of events. Subjects experiencing more than one TEAE within a treatment are counted only once within each SOC and PT

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: This table will be continued for all SOC and PT

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture Protocol: MMV MMV367 21 01

Page x of y

TABLE 14.3.1.3

Treatment-Emergent Adverse Events

By MedDRA System Organ Class, Preferred Term and Severity

Summary Statistics: Safety Analysis Set

Part 1

| | | ALL PLACEBO<br>(N=XX) | | | | | |
|---|---|---|---|---|---|---|---|
| System Organ Class<br>Preferred Term | Mild<br>n(%) | Moderate<br>n(%) | Severe<br>n(%) | Mild<br>n(%) | Moderate<br>n(%) | Severe<br>n(%) | ••••• |
| TEAEs | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| SYSTEM ORGAN CLASS 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| PREFERRED TERM 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| PREFERRED TERM 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| etc | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| SYSTEM ORGAN CLASS 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| PREFERRED TERM 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| PREFERRED TERM 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| etc | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | ••• |

Note: The data in this table are presented in listing x.x

All subjects were planned to receive a single dose of either MMV367 or matching placebo

3.7.7 D.7.30000

All Placebo/All Active relate to placebo or active subjects pooled over all cohorts, respectively

TEAEs are coded using MedDRA vXX.X and are presented in descending order of frequency

Counts are given for total number of subjects, not for events

Counts of number of subjects are by maximum severity, ie subjects experiencing more than one TEAE within a treatment are counted only once within that treatment or each SOC and PT using the most severe episode

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: This table will be continued for all SOC and PT

A similar table will be produced for Part 3, i.e., Table [14.3.3.3]

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


XX ma Fed

Medicines for Malaria Venture Protocol: MMV\_MMV367\_21\_01

Page x of y

TABLE 14.3.2.3
Treatment-Emergent Adverse Events
By MedDRA System Organ Class, Preferred Term and Severity
Summary Statistics: Safety Analysis Set

| | | (N=X) | | | | | | (N=X) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Mild<br>n(%) | | Moderate<br>n(%) | | Severe<br>n(%) | | Mild<br>n(%) | | Moderate<br>n(%) | | Severe<br>n(%) | |
| TEAEs | XX | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | XX | (xx.x) | XX | (xx.x) | - |
| SYSTEM ORGAN CLASS 1 | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | |
| PREFERRED TERM 1 | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | |
| PREFERRED TERM 2 | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | |
| etc | | | | | | | | | | | | | |
| SYSTEM ORGAN CLASS 2 | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | |
| PREFERRED TERM 1 | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | |
| PREFERRED TERM 2 | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | |
| etc | | | | | | | | | | | | | |

XX ma FAST

Note: The data in this table are presented in listing x.x

All subjects were to receive both treatments (i.e., Regimen 6 and Regimen 7) in a randomised manner over the two separate dosing occasions

TEAEs are coded using MedDRA vXX.X and are presented in descending order of frequency

Counts are given for total number of subjects, not for events

Counts of number of subjects are by maximum severity, i.e., subjects experiencing more than one TEAE within a treatment are counted only once within that treatment or each SOC and PT using the most severe episode

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: This table will be continued for all SOC and PT

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture Protocol: MMV MMV367 21 01 Page x of y

TABLE 14.3.1.4

Treatment-Emergent Adverse Events

By MedDRA System Organ Class, Preferred Term and Relationship to IMP

Summary Statistics: Safety Analysis Set

Part 1

| | | PLACEBO<br>I=XX) | ALL A<br>(N= | | | | |
|---|---|---|---|---|---|---|---|
| System Organ Class<br>Preferred Term | Unrelated n(%) | Related n(%) | Unrelated n(%) | Related n(%) | Unrelated<br>n(%) | Related n(%) | |
| TEAES | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| SYSTEM ORGAN CLASS 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| PREFERRED TERM 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| PREFERRED TERM 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | ••• |
| etc | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| SYSTEM ORGAN CLASS 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| PREFERRED TERM 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | ••• |
| PREFERRED TERM 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| etc | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |

Note: The data in this table are presented in listing x.x

All subjects were planned to receive a single dose of either MMV367 or matching placebo

All Placebo/All Active relate to placebo or active subjects pooled over all cohorts, respectively

TEAEs are coded using MedDRA vXX.X and are presented in descending order of frequency

Counts are given for total number of subjects, not for events

Counts of number of subjects are by closest relationship, i.e., subjects experiencing more than one TEAE within a treatment are counted only once within that treatment or each SOC and PT using the most closely related event

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: This table will be continued for all SOC and PT

A similar table will be produced for Part 3, i.e., Table [14.3.3.4]

Status: Approved Date: 19 Dec 2022 Number: DOC-101489 Version: 2.0

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture Protocol: MMV MMV367 21 01

Page x of y

TABLE 14.3.2.4

Treatment-Emergent Adverse Events

By MedDRA System Organ Class, Preferred Term and Relationship to IMP

Summary Statistics: Safety Analysis Set

| | XX m<br>(N | g FED<br>XX) | | |
|---|---|---|---|---|
| System Organ Class<br>Preferred Term | Unrelated<br>n(%) | Related n(%) | Unrelated n(%) | Related<br>n(%) |
| TEAEs | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SYSTEM ORGAN CLASS 1 PREFERRED TERM 1 PREFERRED TERM 2 etc | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| SYSTEM ORGAN CLASS 2 PREFERRED TERM 1 PREFERRED TERM 2 etc | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |

Note: The data in this table are presented in listing x.x

All subjects were to receive both treatments (i.e., Regimen 6 and Regimen 7) in a randomised manner over the two separate dosing occasions

TEAEs are coded using MedDRA vXX.X and are presented in descending order of frequency

Counts are given for total number of subjects, not for events

Counts of number of subjects are by closest relationship, ie subjects experiencing more than one TEAE within a treatment are counted only once within that treatment or each SOC and PT using the most closely related event

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: This table will be continued for all SOC and PT

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture Protocol: MMV MMV367 21 01

Page x of y

TABLE 14.3.1.5

Treatment Emergent Adverse Events Related to IMP By MedDRA System Organ Class and Preferred Term Summary Statistics: Safety Analysis Set

Active Dose of MMV367

| System Organ Class | ALL PLAC<br>(N=XX) | | ALL ACTI<br>(N=XX) | | 100 mg<br>(N=XX) | • | |
|---|---|---|---|---|---|---|---|
| Preferred Term | n (%) | Е | n (%) | E | n (%) | E | • |
| TEAEs | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx | |
| SYSTEM ORGAN CLASS 1 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | xx | |
| PREFERRED TERM 1 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | |
| PREFERRED TERM 2 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | |
| etc | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | |
| SYSTEM ORGAN CLASS 2 | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx | |
| PREFERRED TERM 1 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | |
| PREFERRED TERM 2 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | |
| etc | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | |

Note: The data in this table are presented in listing x.x

All subjects were planned to receive a single dose of either MMV367 or matching placebo

All Placebo/All Active relate to placebo or active subjects pooled over all cohorts, respectively

E = Total Number of Events

TEAEs are coded using MedDRA vXX.X and are presented in descending order of frequency

Subjects experiencing more than one TEAE within a treatment are counted only once for number of subjects but will be counted more than once for number of events. Subjects experiencing more than one TEAE within

a treatment are counted only once within each SOC and PT

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: A similar table will be produced for Serious Adverse Events, i.e., Table [14.3.1.6] Similar tables will be produced for Part 3, i.e., Tables [14.3.3.5] and [14.3.3.6]

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture Protocol: MMV MMV367 21 01

TABLE 14.3.2.5

Treatment Emergent Adverse Events Related to IMP By MedDRA System Organ Class and Preferred Term Summary Statistics: Safety Analysis Set

Part 2

| | | | XX mg<br>(N=X | | | XX mg FED<br>(N=X) | |
|---|---|---|---|---|---|---|---|
| | | | n(%) | Е | | n(%) | E |
| TEAEs (1) | | XX | (xx.x) | XX | XX | (xx.x) | XX |
| SYSTEM ORGAN | CLASS 1 | XX | (xx.x) | xx | XX | (xx.x) | XX |
| PREFERRED | TERM 1 | XX | (xx.x) | XX | XX | (xx.x) | XX |
| PREFERRED | TERM 2 | XX | (xx.x) | XX | XX | (xx.x) | XX |
| etc | | | | | | | |
| SYSTEM ORGAN | CLASS 2 | XX | (xx.x) | xx | XX | (xx.x) | XX |
| PREFERRED | TERM 1 | XX | (xx.x) | XX | XX | (xx.x) | XX |
| PREFERRED | TERM 2 | XX | (xx.x) | XX | XX | (xx.x) | XX |
| etc | | | | | | | |

Note: The data in this table are presented in listing x.x

All subjects were to receive both treatments (i.e., Regimen 6 and Regimen 7) in a randomised manner over the two separate dosing occasions

E = Total Number of Events

TEAEs are coded using MedDRA vXX.X and are presented in descending order of frequency Subjects experiencing more than one TEAE within a treatment are counted only once for number of subjects but will be counted more than once for number of events. Subjects experiencing more than one TEAE within a treatment are counted only once within each SOC and PT

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: A similar table will be produced for Serious AEs, i.e., Table [14.3.2.6]

Reporting and Analysis Plan MMV\_MMV367\_21\_01(QSC207031) Final v2.0 15 Dec 2022

This copy was downloaded by Claire Pages of 12 Dec 2022 at 16:25 GMT+00:00 Check validity before use

Page x of y

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture Protocol: MMV MMV367 21 01

Page x of y

TABLE 14.4.1.1

Haematology and Coagulation

Summary Statistics: Safety Analysis Set

Part 1

<Parameter> (<units>) [ref range xxx-xxx (male), xxx-xxx (female)]

| | | | | Re | sult | | | | Cl | hange fr | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Time Point | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max |
| ALL PLACEBO | BASELINE | xx | xx.xx | xx.xx | xx.xx | xx.x | XX.X | | | | | | |
| (N=XX) | TIMEPOINT 1 | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X |
| | TIMEPOINT 2 | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X |
| ALL ACTIVE | BASELINE | XX | xx.xx | xx.xx | XX.XX | XX.X | XX.X | | | | | | |
| (N=XX) | TIMEPOINT 1 | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X |
| | TIMEPOINT 2 | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X |

Note: The data in this table are presented in listing x.x

All subjects were planned to receive a single dose of either MMV367 or matching placebo

All Placebo/All Active relate to placebo or active subjects pooled over all cohorts, respectively BASELINE is defined as Day -1, Admission

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: This table will be continued for all dose levels, time points and parameters

A similar table will be produced for Clinical Chemistry, [14.4.1.3]. Similar tables will be produced for Part 3, with a column for Visit included before time point column, i.e., Tables [14.4.3.1] and [14.4.3.3]

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture Protocol: MMV MMV367 21 01

Page x of y

TABLE 14.4.2.1

Haematology and Coagulation

Summary Statistics: Safety Analysis Set

Part 2

<Parameter> (<units>) [ref range xxx-xxx (male), xxx-xxx (female)]

| | | | | F | kesult | | | Change from Baseline | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Time Point | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max |
| XX mg FAST | BASELINE | XX | xx.xx | xx.xx | xx.xx | xx.x | xx.x | | | | | | |
| (N=X) | TIME POINT 1 | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X |
| | TIME POINT 2 | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X |
| | | | | | | | | | | | ••• | | |
| | <all other="" points="" time=""></all> | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X |
| XX mg FED | BASELINE | XX | xx.xx | xx.xx | xx.xx | xx.x | xx.x | | | | | | |
| (N=X) | TIME POINT 1 | XX | XX.XX | xx.xx | XX.XX | xx.x | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X |
| | TIME POINT 2 | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X |
| | | | | | | ••• | ••• | | ••• | ••• | ••• | | ••• |
| | <all other="" points="" time=""></all> | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X |

Note: The data in this table are presented in listing x.x

All subjects were to receive both treatments (i.e., Regimen 6 and Regimen 7) in a randomised manner over the two separate dosing occasions
BASELINE is defined as Day -1, Admission

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Change from Baseline

Programming note: This table will be continued for all haematology <and coagulation> parameters and all time points
 A similar table will be produced for Clinical Chemistry, i.e., Table [14.4.2.3]

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture Protocol: MMV MMV367 21 01

Page x of y

TABLE 14.4.1.2

Haematology and Coagulation

Shift Analysis: Safety Analysis Set

Part 1

<Parameter> (<units>) [ref range xxx-xxx (male), xxx-xxx (female)]

#### Baseline

| | Time Point | | Below | Within | Above |
|-------------|-------------|----|-----------|-----------|-----------|
| (N=XX) | Assessment | N# | n(%) | n(%) | n(%) |
| ALL DIACEDO | ETMEDOTNE 1 | | | | |
| | TIMEPOINT 1 | XX | | | |
| (N=XX) | Below | | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Within | | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Above | | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ALL ACTIVE | TIMEPOINT 1 | XX | | | |
| (N=XX) | Below | | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Within | | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Above | | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: The data in this table are presented in listing x.x

All subjects were planned to receive a single dose of either MMV367 or matching placebo

All Placebo/All Active relate to placebo or active subjects pooled over all cohorts, respectively

BASELINE is defined as Day -1, Admission

N# is the total number of subjects that have a value at baseline and the relevant time point and is used in the denominator for calculating the percentages of subjects, n indicates the number of subjects with a baseline and a post baseline assessment at the time point indicated. Below/within/above indicate the n (%) of subjects with assessments

below/within/above the normal reference range

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: Continue this table for all dose levels, time points and parameters

A similar table will be produced for Clinical Chemistry, [14.4.1.4]. Similar tables will be produced for Part 3, with a column for Visit included before time point column, i.e., Tables [14.4.3.2] and [14.4.3.4]

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture Protocol: MMV MMV367 21 01

Page x of y

TABLE 14.4.2.2

Haematology and Coagulation

Shift Analysis: Safety Analysis Set

Part 2

<Parameter> (<units>) [ref range xxx-xxx (male), xxx-xxx (female)]

| | | | (N=X)<br>Baseline | | | | (N=X)<br>Baseline | |
|---|---|---|---|---|---|---|---|---|
| Time Point | | Below | Within | Above | = | Below | Within | Above |
| Assessment | N# | n(%) | n (%) | n (%) | N# | n(%) | n (%) | n (%) |
| TIME POINT 1 | xx | | | | xx | | | |
| Below | | xx (xx.x) | xx (xx.x) | xx (xx.x) | | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Within | | xx (xx.x) | xx (xx.x) | xx (xx.x) | | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Above | | xx (xx.x) | xx (xx.x) | xx (xx.x) | | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TIME POINT 2 | XX | | | | XX | | | |
| Below | | xx (xx.x) | xx (xx.x) | xx (xx.x) | | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Within | | xx (xx.x) | xx (xx.x) | xx (xx.x) | | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Above | | xx (xx.x) | xx (xx.x) | xx (xx.x) | | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| <all other="" points="" time=""></all> | | | | | | | | |
| | | | | | | ••• | | |

XX mg FAST

Note: The data in this table are presented in listing x.x

All subjects were to receive both treatments (i.e., Regimen 6 and Regimen 7) in a randomised manner over the two separate dosing occasions

BASELINE is defined as Day -1, Admission of the corresponding study period

N# indicates the number of subjects with a baseline and a post baseline assessment at the time point indicated Below/within/above indicate the n(%)=number(%) of subjects with assessments below/within/above the normal reference range at baseline

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

XX mg FED

Programming note: This table will be continued for all haematology and coagulation parameters and all time points A similar table will be produced for Clinical Chemistry, i.e., Table [14.4.2.4]

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture Protocol: MMV MMV367 21 01 Page x of y

TABLE 14.5.1.1 Vital Signs

Summary Statistics: Safety Analysis Set

Part 1

<Parameter> (<units>) [ref range xxx - xxx (age xx - xx), xxx - xxx (age > xx)]

| | | | | Res | ult | | | | | - | e from<br>line | | | | Substantial<br>Change | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Time Point | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max | DEC | NONE | INC |
| ALL PLACEBO | BASELINE | xx | xx.xx | xx.xx | xx.xx | xx.x | xx.x | | | | | | | | | |
| (N=XX) | TIMEPOINT 1 | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX | XX |
| | TIMEPOINT 2 | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX | XX |
| | | | ••• | | ••• | | | | ••• | | | ••• | | | | |
| ALL ACTIVE | BASELINE | xx | xx.xx | XX.XX | xx.xx | xx.x | XX.X | | | | | | | | | |
| (N=XX) | TIMEPOINT 1 | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX | XX |
| | TIMEPOINT 2 | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX | XX |
| | | | ••• | ••• | | | | | ••• | | | ••• | | | | |

Note: The data in this table are presented in listing x.x

All subjects were planned to receive a single dose of either MMV367 or matching placebo

All Placebo/All Active relate to placebo or active subjects pooled over all cohorts, respectively

BASELINE is defined as Day 1, Pre-dose

Substantial change is defined as:  $> \pm$  20 mmHg Systolic BP,  $> \pm$  10 mmHg Diastolic BP and  $> \pm$  15 bpm HR

DEC: number of subjects with substantial decrease from baseline NONE: number of subjects with no substantial

change from baseline, INC: number of subjects with substantial increase from baseline

PROGRAM PATH: X:\~\OSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: Continue this table for all dose levels, time points and parameters (which will follow the order given in the RAP text)

A similar table will be produced for Part 3, with a column for Visit included before time point
column, i.e., Table [14.5.1.3]

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture
Page x of y
Protocol: MMV MMV367 21 01

TABLE 14.5.1.2 Vital Signs

Summary Statistics: Safety Analysis Set

Part 2

<Parameter> (<units>) [ref range xxx - xxx (age xx - xx), xxx - xxx (age > xx)]

| | | | | R | esult | | | | Change from<br>Baseline | | | | | Substantial<br>Change (1) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Time Point | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max | DEC | NONE | INC |
| XX mg FAST | BASELINE | xx | xx.xx | xx.xx | xx.xx | xx.x | xx.x | | | | | | | | | |
| (N=X) | TIME POINT 1 | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX | XX |
| | TIME POINT 2 | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX | XX |
| | TIME POINT 3 | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX | XX |
| | <all other="" points="" time=""></all> | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | xx.xx | XX.XX | XX.XX | XX.X | XX.X | XX | XX | XX |
| XX mg FED | BASELINE | XX | xx.xx | xx.xx | xx.xx | xx.x | XX.X | | | | | | | | | |
| (N=X) | TIME POINT 1 | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX | XX |
| | TIME POINT 2 | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX | XX |
| | TIME POINT 3 | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX | XX |
| | <all other="" points="" time=""></all> | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX | XX |

Note: The data in this table are presented in listing x.x

All subjects were to receive both treatments (i.e., Regimen 6 and Regimen 7) in a randomised manner

over the two separate dosing occasions

BASELINE is defined as Day 1, Pre-dose of the corresponding study period

Substantial change is defined as:  $> \pm$  20 mmHg Systolic BP,  $> \pm$  10 mmHg Diastolic BP and  $> \pm$  15 bpm HR

DEC: number of subjects with substantial decrease from baseline NONE: number of subjects with no substantial

change from baseline, INC: number of subjects with substantial increase from baseline

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: This table will be continued for all vital signs parameters, which will follow the order given in the RAP text
QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture
Protocol: MMV MMV367 21 01
Page x of y

TABLE 14.5.2.1.1

ECGs

Summary Statistics: Safety Analysis Set

Single 12-Lead

Part 1

<Parameter> (<units>) [<ref range xxx - xxx (age xx - xx), xxx - xxx (age > xx)> / <ref range xxx - xxx (male), xxx-xxx (female)>]

| | | | | Re | sult | | | | Cl | hange fr | om Basel: | ine | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Time Point | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max |
| ALL PLACEBO | BASELINE | XX | xx.xx | xx.xx | xx.xx | XX.X | XX.X | | | | | | |
| (N=XX) | TIMEPOINT 1 | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X |
| | TIMEPOINT 2 | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | xx.x |
| | | | | | | | | | | | ••• | | ••• |
| ALL ACTIVE | BASELINE | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | xx.xx | XX.XX | XX.X | XX.X |
| (N=XX) | TIMEPOINT 1 | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X |
| | TIMEPOINT 2 | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | xx.x |
| | | ••• | ••• | | ••• | | ••• | | ••• | | ••• | ••• | ••• |

Note: The data in this table are presented in listing x.x

All subjects were planned to receive a single dose of either MMV367 or matching placebo

All Placebo/All Active relate to placebo or active subjects pooled over all cohorts, respectively BASELINE is defined as Day 1, mean of 3 Pre-dose measurements

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: This table will be continued for all dose levels, time points and parameters (which will follow the order given in the RAP text)

A similar table will be produced for triplicate readings i.e., Table [14.5.2.1.2]

Similar tables will also be produced for Part 3, with a column for Visit included before time point

column, i.e., Tables [14.5.2.3.1] and [14.5.2.3.2]


Medicines for Malaria Venture Page x of y Protocol: MMV MMV367 21 01

TABLE 14.5.2.2.1

Summary Statistics: Safety Analysis Set

Single 12-Lead

Part 2

<Parameter> (<units>) [<ref range xxx - xxx (age xx - xx), xxx - xxx (age > xx)> / <ref range xxx - xxx (male), xxx-xxx (female)>]

| | | | | Re | esult | | | | ( | Change f | rom Basel: | ine | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Time Point | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max |
| XX mg FAST | BASELINE | xx | XX.XX | xx.xx | xx.xx | xx.x | XX.X | | | | | | |
| (N=X) | TIME POINT 1 | XX | xx.xx | XX.XX | XX.XX | XX.X | xx.x | XX | xx.xx | XX.XX | xx.xx | XX.X | xx.x |
| | TIME POINT 2 | XX | xx.xx | XX.XX | xx.xx | XX.X | XX.X | XX | xx.xx | XX.XX | XX.XX | XX.X | xx.x |
| | TIME POINT 3 | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X |
| | <all other="" points="" time=""></all> | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X |
| XX MG FED | BASELINE | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | | | | | | |
| (N=X) | TIME POINT 1 | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X |
| | TIME POINT 2 | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X |
| | TIME POINT 3 | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X |
| | | | | | | | | | ••• | | | | ••• |
| | <all other="" points="" time=""></all> | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX | XX.XX | XX.XX | XX.XX | XX.X | XX.X |

Note: The data in this table are presented in listing x.x

All subjects were to receive both treatments (i.e., Regimen 6 and Regimen 7) in a randomised manner over the two separate dosing occasions

BASELINE is defined as Day 1, Pre-dose of the corresponding study period

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: This table will be continued for all ECG parameters, which will follow the order given in the RAP text A similar table will be produced for triplicate readings i.e., Table [14.5.2.2.2]

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture Protocol: MMV\_MMV367\_21\_01

Page x of y

TABLE 14.5.2.1.3

ECGs

QTcB and QTcF Categorical Data

Summary Statistics: Safety Analysis Set

Part 1

| | | | | | CcF<br>al (msec) | | ] | QTcF Interval<br>Increase (msed | |
|---|---|---|---|---|---|---|---|---|---|
| Treatment | Time Point | N# | <=450<br>n(%) | 451-480<br>n(%) | 481-500<br>n(%) | >500<br>n(%) | =<30<br>n(%) | 31-60<br>n(%) | >60<br>n(%) |
| ALL PLACEBO | BASELINE | xx | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | | | |
| (N=XX) | TIMEPOINT 1 | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | TIMEPOINT 2 | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ALL ACTIVE | BASELINE | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| (N=XX) | TIMEPOINT 1 | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | TIMEPOINT 2 | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | | | <b></b> | | | | <b></b> | |

Note: The data in this table are presented in listing x.x

All subjects were planned to receive a single dose of either MMV367 or matching placebo

All Placebo/All Active relate to placebo or active subjects pooled over all cohorts, respectively

BASELINE is defined as Day 1, Pre-dose

Categories for QTcF interval and QTcF interval increases are based on ICH E14 guidelines

N# is the total number of subjects at the relevant time point and is used in the denominator for calculating the percentages of subjects, n indicates the number of subjects with observations at the given time point

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: This table will be continued for QTCB

A similar table will be produced for Part 3, with a column for Visit included before time point column, i.e., Table [14.5.2.3.3]

Reporting and Analysis Plan MMV\_MMV367\_21\_01(QSC207031) Final v2.0
15 Dec 2022

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture Protocol: MMV MMV367 21 01

Page x of y

TABLE 14.5.2.2.3

QTcB and QTcF Categorical Data

Summary Statistics: Safety Analysis Set

Part 2

| | | | | Q | TcF | | | QTcF Interval | 1 | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Interv | al (msec) | | ] | Increase (msed | c) | |
| | | | <=450 | 451-480 | 481-500 | >500 | <=30 | 31-60 | >60 | - |
| Treatment | Time Point | N# | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) | |
| XX mg FAST | BASELINE | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | | | | _ |
| (N=X) | TIME POINT 1 | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| | TIME POINT 2 | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| | TIME POINT 3 | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| | | | | | | ••• | | | | |
| | <all other="" points="" time=""></all> | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| XX mg FED | BASELINE | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | | | | |
| (N=X) | TIME POINT 1 | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| | TIME POINT 2 | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| | TIME POINT 3 | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| | | | | | | ••• | ••• | | | |
| | <all other="" points="" time=""></all> | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |

Note: The data in this table are presented in listing x.x

All subjects were to receive both treatments (i.e., Regimen 6 and Regimen 7) in a randomised manner over the two separate dosing occasions

BASELINE is defined as Day 1, Pre-dose of the corresponding study period

Categories for QTcF interval and QTcF interval increases are based on ICH E14 guidelines

 $N^{\#}$  is the number of subjects with a value at baseline and the relevant post-dose time point. It is the denominator for calculating the percentages of subjects, n indicates the number of subjects with observations at the given time point

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX DDMMMYYYY HH:MM

Programming note: This table will be continued for QTcB

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture Protocol: MMV\_MMV367\_21\_01

Page x of y

TABLE 14.6.1.1

Taste Assessments: Taste Aspect

Summary Statistics: Taste Analysis Set

Part 1

<Taste Aspect>

MMV367

| | Dealed Diseales | 100 | 200 |
|---------------|-----------------|-----------|-----------|
| | Pooled Placebo | 100 mg | 300 mg |
| Statistic | (N=XX) | (N=XX) | (N=XX) |
| n | xx | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X |
| Min | XX.X | XX.X | XX.X |
| Max | XX.X | XX.X | XX.X |
| GRADE 1 n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| GRADE 2 n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| GRADE 3 n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| GRADE 4 n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| GRADE 5 n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| GRADE 6 n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| GRADE 7 n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| GRADE 8 n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| GRADE 9 n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: The data in this table are presented in listing x.x

All subjects were planned to receive a single dose of either MMV367 or matching placebo

All Placebo/All Active relate to placebo or active subjects pooled over all cohorts, respectively

Key for grade: 1=Dislike extremely, 2=Dislike very much, 3=Dislike moderately, 4=Dislike slightly, 5=Neither like nor dislike, 6=Like slightly, 7=Like moderately, 8=Like very much, 9=Like extremely

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX

DDMMMYYYY HH:MM

Programming note: This table will be continued for all dose levels.

A separate page will be used for each taste aspect with the relevant subheading

A similar table will be produced for Overall Acceptability, i.e., Table [14.6.1.2]

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Medicines for Malaria Venture Protocol: MMV MMV367 21 01

Page x of y

TABLE 14.6.1.3

Taste Assessments: Taste Aspects including Overall Acceptability

Statistical Analysis Results: Taste Analysis Set

Part 1

Wilcoxon Rank Sum Test: <Taste Aspect>

| | | Test | P | Reference | | | |
|---|---|---|---|---|---|---|---|
| Comparison | n | Median | n | Median | Difference (1) | 90% CI<br>(2) | p-value<br>(3) |
| 100 mg vs<br>Pooled Placebo | XX | xxx | xx | xxx | xxx | (xx.xx, xx.xx) | 0.xxx |
| 300 mg vs<br>Pooled Placebo | XX | xxx | xx | xxx | xxx | (xx.xx, xx.xx) | 0.xxx |
| | | ••• | ••• | | ••• | | |

Note: The data in this table are presented in listing x.x

All subjects were planned to receive a single dose of either MMV367 or matching placebo

All Placebo/All Active relate to placebo or active subjects pooled over all cohorts, respectively

Results obtained from non-parametric Wilcoxon rank sum test

(1) Hodges-Lehmann median difference for test (Regimens 1 to 5 - Pooled Placebo), (2) Confidence interval for Hodges-Lehmann median difference (3) p-value from Wilcoxon rank sum test for the null hypothesis that the Hodges-Lehmann median difference is zero Hodges-Lehmann median difference is not necessarily the same as the difference between medians

PROGRAM PATH: X:\~\QSC207031\~\TFLS\PRODUCTION\TAB-XX DDMMMYYYY HH:MM

Programming note: This table will be continued for all dose level comparisons


Appondix 1 Schodulo of Assessments: Part 1 (Cohorts 1A to 1E)

| Appendix 1 Schedule | | | | • | | | | - 10 M | End of Study |
|---|---|---|---|---|---|---|---|---|---|
| | Screening | Admission | | Re | esident In-cli | nic | | Return Visit <sup>b</sup> | Visitb |
| Study Day | -28 to -2 | -1 | 1 | 2 | 3 | 4 | 5 <sup>a</sup> | 7 | 15 |
| General Assessments | | | | | | | • | | |
| Informed Consent | X | | | | | | | | |
| Medical History | X | Xc | | | | | | | |
| Weight, Height and BMI | X | Xd | | | | | | Xq | Xq |
| Vein Assessment | X | | | | | | | | |
| Carbon Monoxide Breath Test | Х | X | | | | | | | |
| Drug Screen | Х | X | | | | | | | |
| Alcohol Breath Test | X | X | | | | | | | |
| SARS-CoV-2 Antigen <sup>e</sup> | Х | X | | | | | | | |
| Randomisation <sup>f</sup> | | | Х | | | | | | |
| IMP Administration <sup>g</sup> | | | Х | | | | | | |
| Safety Assessments | | | | | | | | | |
| BDI-II Questionnaire | Х | X | | | | | | | |
| Physical Examination | Х | Х | | | | | | | |
| Targeted (symptom driven) Physical Examination <sup>h</sup> | | | Х | Х | Х | Х | Х | Х | Х |
| Safety Labs <sup>i</sup> | Х | Х | | Х | | | Х | X | Х |
| Urinalysis <sup>i</sup> | Х | Х | | Х | | | Х | Х | Х |
| Follicle-stimulating Hormone (FSH) Test <sup>j</sup> | X | | | | | | | | |
| Serum Pregnancy Test <sup>k</sup> | Х | | | | | | | | |
| Urine Pregnancy Testk | | Х | | | | | | X | Х |
| Single 12-Lead ECGs <sup>I</sup> | Х | Х | Х | Х | | | | | Х |
| Triplicate 12-Lead ECGs <sup>I</sup> | | | | | Х | Х | Х | X | |
| Holter Periods <sup>m</sup> | | | Х | Х | | | | | |
| Telemetry <sup>n</sup> | | | Х | | | | | | |
| Vital Signs <sup>o</sup> | Х | Х | Х | Х | Х | Х | Х | X | Х |
| Orthostatic Vital Signs <sup>o</sup> | Х | | Х | Х | | | | X | |
| Adverse Events | < | | | | X | | | | > |
| Prior and Concomitant Medication | < | | | | X- | | | | > |
| PK/Metabolite ID/Pharmacogenetic Asse | essments | | | | | | | | |
| Plasma Samples for MMV367 <sup>p</sup> | | | Х | Х | Х | Х | Х | X | |
| Urine Samples for MMV367pq | | | Х | Х | Х | | | | |

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


| | Screening | Admission | | Re | sident In-cli | nic | | Return Visit <sup>b</sup> | End of Study<br>Visit <sup>b</sup> |
|---|---|---|---|---|---|---|---|---|---|
| Study Day | -28 to -2 | -1 | 1 | 2 | 3 | 4 | <b>5</b> <sup>a</sup> | 7 | 15 |
| Blood Sample for CYP/UGT polymorphism <sup>r</sup> | | | Х | | | | | | |
| Taste/Palatability Assessments | | | | | | | | | |
| Taste/Palatability Questionnaires | | | | | | | | | |

Eligibility will be re-assessed at admission/pre-dose on Day 1.

- <sup>a</sup> Discharge from clinical unit
- b Participants will return for an outpatient visit on Day 7 and an end of study visit on Day 15 (±1 day).
- <sup>c</sup> Update only
- d Weight only
- e It is planned that testing will comprise an antigen test performed at screening and on Day -1 prior to admission to the clinical unit. The definition of the COVID-19 testing time points are participant to change based on the current risk mitigation in place and will be agreed by the study team and documented in the ISF via the Clinical Kick-Off Meeting minutes.
- f Participants will be randomised on the morning of Day 1 prior to dosing
- <sup>9</sup> Participants will receive a single dose of MMV367 or placebo on Day 1
- h Targeted (symptom driven) physical examination of the relevant body system(s) as clinically indicated, as per the investigator's judgement
- Haematology, coagulation and clinical chemistry and urinalysis at each time point, including virology and FSH (post-menopausal female participants only) at screening. See study protocol for safety blood sample time points.
- Post-menopausal female participants only
- <sup>k</sup> All female participants
- <sup>1</sup> See study protocol for single and triplicate 12-lead ECG time points. For triplicate ECGs, participants will be required to rest in the supine position with no external stimuli (e.g. music or television) for 15 min prior to the nominal time point where a triplicate ECG is scheduled.
- m Continuous Holter monitoring will commence at least 1.5 h prior to dosing until at least 24 h post-dose. Participants will be required to rest in the supine position with no external stimuli (e.g. music or television) for 15 min prior to the nominal time point where an ECG extraction is scheduled. See study protocol for Holter extraction time points.
- <sup>n</sup> Telemetry (continuous ECG monitoring) will commence at least 30 min before dosing until at least 12 h post-dose.
- <sup>o</sup> Blood pressure, heart rate and respiratory rate at all time points. Oral temperature will be measured at screening/admission only. See study protocol for vital signs and orthostatic vital signs time points.
- P See study protocol for PK sample time points. Metabolite profiling of MMV367 in plasma and urine will be performed using existing PK samples (pooled residual samples).
- q Urine collection in Cohorts 1C and 1D only.
- <sup>r</sup>Sample will be taken prior to IMP administration (≤2 h before dosing).
- The taste/palatability questionnaire will be completed immediately after IMP administration, see study protocol for details.


Annandiv 2 Schodula of Assassments: Part 2

| | | | | | | | | F | Resider | t in Clinic | | | | | End of Study |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening | Admi-<br>ssion | | | ı | Period | 1 | | | | | Period 2 | | | Visit |
| Study Day | -28 to -2 | -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12ª | 14 <sup>b</sup> |
| General Assessments | | | | | | | | | | | | | | | |
| Informed Consent | Х | | | | | | | | | | | | | | |
| Medical History | Х | Xc | | | | | | | | | | | | | |
| Weight, Height and BMI | Х | $X^d$ | | | | | | | | | | | | | |
| Vein Assessment | Х | | | | | | | | | | | | | | |
| Carbon Monoxide Breath Test | | Χ | | | | | | | | | | | | | |
| Drug Screen | Х | Χ | | | | | | | | | | | | | |
| Alcohol Breath Test | X | Х | | | | | | | | | | | | | |
| SARS-CoV-2 Antigene | X | Х | | | | | | | | | | | | | |
| Randomisation <sup>f</sup> | | | Х | | | | | | | | | | | | |
| IMP Administration <sup>9</sup> | | | Х | | | | | | | Х | | | | | |
| Safety Assessments | | | | • | | | | | | | | • | • | | |
| BDI-II Questionnaire | X | Х | | | | | | | | | | | | | |
| Physical Examination | Х | Х | | | | | | | | | | | | | |
| Targeted (symptom driven)<br>Physical Examination <sup>h</sup> | | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Safety Labs <sup>i</sup> | Х | Х | | Х | | | Х | | Х | | Х | | | Х | Х |
| Urinalysis <sup>i</sup> | Х | Х | | Х | | | Х | | Х | | Х | | | Х | Х |
| Follicle-stimulating Hormone<br>(FSH) Test <sup>j</sup> | Х | | | | | | | | | | | | | | |
| Serum Pregnancy Test <sup>k</sup> | Х | | | | | | | | | | | | | | |
| Urine Pregnancy Test <sup>k</sup> | | Х | | | | | | | | | | | | | Х |
| Single 12-Lead ECGs <sup>I</sup> | Х | Х | Х | X | | | | | | Х | Х | | | | X |
| Triplicate 12-Lead ECGs <sup>I</sup> | | | | | Х | Х | Х | | Х | | | Х | Х | Х | |
| Holter Periods <sup>m</sup> | | | X | Х | | | | | | Х | Х | | | | |
| Telemetry <sup>n</sup> | | | Х | | | | | | | Х | | | | | |
| Vital Signs <sup>o</sup> | Х | Х | Х | Х | Х | Х | Х | | Х | Х | Х | Х | Х | Х | Х |
| Adverse Events | | < | · | | | | | | | | | | | | > |
| Prior and Concomitant<br>Medication | | < | | | | | | | X | | | | | | > |

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


| PK/Pharmacogenetic Assess | sments | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Plasma Samples for MMV367 <sup>p</sup> | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Blood Sample for CYP/UGT polymorphism <sup>q</sup> | | Х | | | | | | | | | | | |

Eligibility will be re-assessed at admission/pre-dose on Day 1.

- <sup>a</sup> Discharge from clinical unit
- <sup>b</sup> Participants will return for an end of study visit on Day 14 (± 1 day).
- <sup>c</sup> Update only
- d Weight only
- e It is planned that testing will comprise an antigen test performed at screening and on Day -1 prior to admission to the clinical unit. The definition of the COVID-19 testing time points are participant to change based on the current risk mitigation in place and will be agreed by the study team and documented in the ISF via the Clinical Kick-Off Meeting minutes.
- f Participants will be randomised on the morning of Period 1, Day 1 prior to dosing
- <sup>9</sup> Participants will receive a single dose of MMV367 on Day 1 and Day 8 in the fed or fasted state
- h Targeted (symptom driven) physical examination of the relevant body system(s) as clinically indicated, as per the investigator's judgement
- <sup>i</sup> Haematology, coagulation, clinical chemistry and urinalysis at each time point, including virology and FSH (post-menopausal female participants only) at screening.
- Post-menopausal female participants only
- <sup>k</sup> All female participants
- <sup>1</sup> See study protocol for single and triplicate 12-lead ECG time points. For triplicate ECGs, participants will be required to rest in the supine position with no external stimuli (e.g. music or television) for 15 min prior to the nominal time point where a triplicate ECG is scheduled.
- m Continuous Holter monitoring will commence at least 1.5 h prior to dosing until at least 24 h post-dose. Participants will be required to rest in the supine position with no external stimuli (e.g. music or television) for 15 min prior to the nominal time point where an ECG extraction is scheduled. See study protocol for Holter extraction time points.
- <sup>n</sup> Telemetry (continuous ECG monitoring) will commence at least 30 min before dosing until at least 12 h post-dose.
- <sup>o</sup> Blood pressure, heart rate and respiratory rate at all time points. Oral temperature will be measured at screening and admission only. See study protocol for vital signs time points.
- <sup>p</sup> See study protocol for PK sample time points.
- <sup>q</sup> Sample will be taken prior to IMP administration (≤2 h before dosing).


Schedule of Assessments: Part 3 (Cohorts 3A to 3C) Annandiv 3

| Appendix 3 Schedu<br>Study Day | Screening | Admission | | | Re | sident lı | n-clinic | | | Return Visit <sup>b</sup> | End of Study<br>Visit <sup>b</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|
| , , | -28 to -2 | -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 <sup>a</sup> | 9 | 17 |
| General Assessments | - | | | | • | | | | | | |
| Informed Consent | X | | | | | | | | | | |
| Medical History | X | Xc | | | | | | | | | |
| Weight, Height and BMI | X | Xd | | | | | | | | Xd | Xd |
| Vein Assessment | X | | | | | | | | | | |
| Carbon Monoxide Breath Test | X | X | | | | | | | | | |
| Drug Screen | X | X | | | | | | | | | |
| Alcohol Breath Test | X | X | | | | | | | | | |
| SARS-CoV-2 Antigen <sup>e</sup> | X | X | | | | | | | | | |
| Randomisation <sup>f</sup> | | | Χ | | | | | | | | |
| IMP Administration <sup>g</sup> | | | Χ | X | Х | | | | | | |
| Safety Assessments | | | | | | | | | | | |
| BDI-II Questionnaire | X | X | | | | | | | | | |
| Physical Examination | Х | X | | | | | | | | | |
| Targeted (symptom driven) Physical Examination <sup>h</sup> | | | X | Х | Х | Х | Х | Х | Х | Х | Х |
| Safety Labs <sup>i</sup> | Х | X | | | Х | | Х | | Х | Х | Х |
| Urinalysis <sup>i</sup> | Х | Х | | | Х | | Х | | Х | X | Х |
| Follicle-stimulating Hormone (FSH)<br>Test <sup>j</sup> | X | | | | | | | | | | |
| Serum Pregnancy Test <sup>k</sup> | Х | | | | | | | | | | |
| Urine Pregnancy Test <sup>k</sup> | | X | | | | | | | | X | Х |
| Single 12-Lead ECGs <sup>I</sup> | X | X | Х | | Х | Х | | | | | Х |
| Triplicate 12-Lead ECGs <sup>I</sup> | | | | Х | | Х | Х | Х | Х | X | |
| Holter Periods <sup>m</sup> | | | Х | Х | Х | Х | | | | | |
| Vital Signs <sup>n</sup> | X | X | Х | Х | Х | Х | Х | Х | Х | X | Х |
| Orthostatic Vital Signs <sup>n</sup> | Х | | Х | Х | Х | Х | | | | Х | |
| Adverse Events | < | | | | | | X | | | | > |
| Prior and Concomitant Medication | < | | | | | | X | | | | > |
| PK/Pharmacogenetic Assessments | | | | | | | | | | | |
| Plasma Samples for MMV367° | | | Х | Х | Х | Х | Х | Х | Х | X | |
| Blood Sample for CYP/UGT polymorphism <sup>p</sup> | | | Х | | | | | | | | |

QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan


Eligibility will be re-assessed at admission/pre-dose on Day 1.

- <sup>a</sup> Discharge from clinical unit
- <sup>b</sup> Participants will return for an outpatient visit on Day 9 and an end of study visit on Day 17 (± 1 day).
- <sup>c</sup> Update only
- d Weight only
- <sup>e</sup> It is planned that testing will comprise an antigen test performed at screening and on Day -1 prior to admission to the clinical unit. The definition of the COVID-19 testing time points are participant to change based on the current risk mitigation in place and will be agreed by the study team and documented in the ISF via the Clinical Kick-Off Meeting minutes.
- f Participants will be randomised on the morning of Day 1 prior to dosing
- <sup>9</sup> Participants will receive a dose of MMV367 or placebo in the morning on Days 1, 2 and 3
- h Targeted (symptom driven) physical examination of the relevant body system(s) as clinically indicated, as per the investigator's judgement
- <sup>1</sup> Haematology, coagulation, clinical chemistry and urinalysis at each time point, including virology and FSH (post-menopausal female participants only) at screening.
- Post-menopausal female participants only
- <sup>k</sup> All female participants
- <sup>1</sup> See study protocol for single and triplicate 12-lead ECG time points. For triplicate ECGs, participants will be required to rest in the supine position with no external stimuli (e.g. music or television) for 15 min prior to the nominal time point where a triplicate ECG is scheduled.
- <sup>m</sup> Continuous Holter monitoring will commence at least 1.5 h prior to dosing until at least 24 h post-dose. Participants will be required to rest in the supine position with no external stimuli (e.g. music or television) for 15 min prior to the nominal time point where an ECG extraction is scheduled. See study protocol for Holter extraction time points.
- <sup>n</sup> Blood pressure, heart rate and respiratory rate at all time points. Oral temperature will be measured at screening and admission only. See study protocol for vital signs and orthostatic vital signs time points.
- ° See study protocol for PK sample time points.
- <sup>p</sup> Sample will be taken prior to IMP administration (≤2 h before dosing).


Part 1 (All Cohorts) Safety and Pharmacokinetic Assessment Time Points (Days 1 to 7) Annendix 4

| ppenaix | 4 Pail I | | Jiioris) Sai | ety and Phann | acokinetic Assess | ment | i ime Poin | us (Day | ys i to |
|---|---|---|---|---|---|---|---|---|---|
| Study Day | Time point | Plasma<br>PK | Urine PK <sup>a</sup> | Safety Labs and<br>Urinalysis | Holter Extractions | Vital<br>Signs <sup>b</sup> | Orthostatic<br>Vital Signs | Single<br>12-lead<br>ECGs | Triplicate<br>12-lead<br>ECGs |
| | -1.5 h | | | | Х | | | Х | |
| | -1 h | | | | Х | | | Х | |
| | Pre-dose<br>(-0.5 h) | х | Х | | Х | Х | х | Х | |
| | 0 h | | | | | | | | |
| | 0.5 h | Х | | | Х | Х | | Х | |
| | 1 h | Х | | | Х | | | Х | |
| 1 | 2 h | Х | 0 to 6 h | | Х | Х | Х | Х | |
| | 3 h | Х | | | X | | | Х | |
| | 4 h | Х | | | Х | Х | Х | Х | |
| | 5 h | Х | | | | | _ | Х | |
| | 6 h | Х | | | Х | Х | | Х | |
| | 8 h | Х | 6 to 12 h | | Х | Х | | Х | |
| | 10 h | | | | | Х | | | |
| | 12 h | Х | 12 to 24 h | | Х | Х | Х | Х | |
| 2 | 24 h | Х | 24 to 48 h | X | Х | Х | Х | Х | |
| 3 | 48 h | Х | 48 to 72 h | | | Х | | | Х |
| 4 | 72 h | Х | | | | Х | | | Х |
| 5 | 96 h | Х | | X | | Х | | | Х |
| 7 | 144 h | Х | | X | | Х | Х | | Х |

a Part 1, Cohorts 1C and 1D only

Allowable windows for PK blood sampling, vital signs assessments and ECGs can be found in: Section 13.1, 14.6 and 14.7 of the study protocol.

<sup>&</sup>lt;sup>b</sup> Blood pressure, heart rate and respiratory rate at all time points.


Annondiy 5 Part 2 Safety and Pharmacokinetic Assessment Time Points (Days 1 to 1/1)

| Appendix 5 | Part 2 Safety and Pharmacokinetic Assessment Time Points (Days 1 to 14) | | | | | | |
|---|---|---|---|---|---|---|---|
| Study Day | Time point | Plasma<br>PK | Safety Labs and<br>Urinalysis | Holter Extractions | Vital Signs <sup>a</sup> | Single<br>12-lead<br>ECGs | Triplicate<br>12-lead<br>ECGs |
| | -1.5 h | | | Х | | Χ | |
| | -1 h | | | X | | Х | |
| | Pre-dose<br>(-0.5 h) | Х | | X | Х | Х | |
| | 0 h | | | | | | |
| | 0.5 h | X | | X | X | Χ | |
| | 1 h | X | | X | | Χ | |
| , | 2 h | X | | X | X | Χ | |
| 1 | 3 h | Х | | X | | Χ | |
| | 4 h | X | | X | X | Χ | |
| | 5 h | Х | | | | | |
| | 6 h | Х | | Х | X | Х | |
| | 7 h | | | | | | |
| | 8 h | Х | | Х | X | Х | |
| | 10 h | | | | X | | |
| | 12 h | Х | | X | X | Х | |
| 2 | 24 h | Х | Х | Х | X | Χ | |
| 3 | 48 h | Х | | | X | | Х |
| 4 | 72 h | Х | | | X | | Х |
| 5 | 96 h | Х | X | | X | | Х |
| 7 | 144 h | Х | Х | | X | | Х |
| | -1.5 h | | | Х | | Х | |
| | -1 h | | | X | | Χ | |
| 8 | Pre-dose<br>(-0.5 h) | Х | | Х | Х | Х | |
| | 0 h | | | | | | |
| | 0.5 h | Х | | X | X | Х | |


| Study Day | Time point | Plasma<br>PK | Safety Labs and<br>Urinalysis | Holter Extractions | Vital Signs <sup>a</sup> | Single<br>12-lead<br>ECGs | Triplicate<br>12-lead<br>ECGs |
|---|---|---|---|---|---|---|---|
| | 1 h | Х | | X | | Χ | |
| | 2 h | Х | | X | Х | Χ | |
| | 3 h | Х | | X | | Х | |
| | 4 h | Х | | X | Х | Х | |
| | 5 h | Х | | | | | |
| | 6 h | Х | | X | Х | Х | |
| | 7 h | | | | | | |
| | 8 h | Х | | X | Х | Х | |
| | 10 h | | | | X | | |
| | 12 h | Х | | X | Х | Χ | |
| 9 | 24 h | Х | Χ | X | X | Χ | |
| 10 | 48 h | Х | | | X | | Х |
| 11 | 72 h | Х | | | X | | Х |
| 12 | 96 h | Х | X | | X | | Х |
| 14 | 144 h | Х | Χ | | X | | Х |

<sup>&</sup>lt;sup>a</sup> Blood pressure, heart rate and respiratory rate at all time points.

Allowable windows for PK blood sampling, vital signs assessments and ECGs can be found in: Sections 13.1, 14.6 and 14.7 of the study protocol.


Annondiv 6 Part 3 Safety and Pharmacokinetic Assessment Time Points (Days 1 to 9)

| Appendi | x 6 Part 3 Sa | afety and Pi | narmacokinet | tic Assessment | t Time Poi | nts (Days 1 | to 9) | |
|---|---|---|---|---|---|---|---|---|
| Study Day | Time point | Plasma PK | Safety Labs and<br>Urinalysis | Holter Extractions | Vital Signs <sup>a</sup> | Orthostatic Vital<br>Signs | Single<br>12-lead<br>ECGs | Triplicate<br>12-lead<br>ECGs |
| | -1.5 h | | | X | | | Х | |
| | -1 h | | | Х | | | Х | |
| | Pre-dose (-0.5 h) | Х | | X | Х | Х | Х | |
| | 0 h | | | | | | | |
| | 0.5 h | Х | | Х | | | | |
| Ī | 1 h | Х | | X | Х | | Х | |
| | 2 h | Х | | X | Х | X | Х | |
| 1 | 3 h | Х | | X | Х | | Х | |
| | 4 h | Х | | X | Х | X | Х | |
| -<br>-<br>-<br>- | 5 h | Х | | | | | | |
| | 6 h | Х | | Х | Х | X | Х | |
| | 8 h | Х | | X | Х | | Х | |
| | 10 h | | | Х | Х | | | |
| | 11 h | | | | | | | |
| | 12 h | Х | | Х | Х | Х | Х | |
| | -1.5 h | | | | | | | Х |
| | -1 h | | | | | | | Х |
| | Pre-dose (-0.5 h)b | Х | | X (Day 1, 24 h) | Х | X (Day 1, 24 h) | | Х |
| | 0 h | | | | | | | |
| | 1 h | | | | | | | |
| , | 2 h | | | | | | | |
| 2 | 3 h | | | | | | | |
| | 4 h | Х | | | Х | | | Х |
| | 5 h | | | | | | | |
| | 6 h | X | | | X | | | Х |
| | 7 h | | | | | | | |
| Ţ. | 8 h | | | | | | | |


| Study Day | Time point | Plasma PK | Safety Labs and<br>Urinalysis | Holter Extractions | Vital Signs <sup>a</sup> | Orthostatic Vital<br>Signs | Single<br>12-lead<br>ECGs | Triplicate<br>12-lead<br>ECGs |
|---|---|---|---|---|---|---|---|---|
| | 9 h | | | | | | | |
| | 10 h | | | | Х | | | |
| | 11 h | | | | | | | |
| | 12 h | Х | | | Х | | | Х |
| | -1.5 h | | | X | | | Х | |
| | -1 h | | | Х | | | Х | |
| | Pre-dose (-0.5 h) <sup>c</sup> | Х | X (Day 1, 48 h) | X (Day 1, 48 h) | Х | Х | Χ | |
| | 0 h | | | | | | | |
| | 0.5 h | Х | | Х | Х | | Χ | |
| | 1 h | Х | | Х | Х | | Х | |
| | 2 h | Х | | Х | Х | X | Х | |
| | 3 h | Х | | Х | Х | | Х | |
| 3 | 4 h | Х | | Х | Х | Х | Х | |
| | 5 h | Х | | | | | | |
| | 6 h | X | | Х | Х | X | Χ | |
| | 7 h | | | | | | | |
| | 8 h | Х | | Х | Х | | Х | |
| | 9 h | | | | | | | |
| | 10 h | | | Х | Х | | | |
| | 11 h | | | Х | | | | |
| | 12 h | Х | | Х | Х | Х | Х | |
| 4 | 24 h | Х | | Х | Х | X | Х | |
| <u> </u> | 36 h | Х | | | Х | | | Х |
| 5 | 48 h | Х | Х | | Х | | | Х |
| 6 | 72 h | Х | | | Х | | | Х |
| 7 | 96 h | Х | Х | | Х | | | Х |
| 9 | 144 h | Х | X | | Х | Х | | Х |

a Blood pressure, heart rate and respiratory rate at all time points. b 24 h post-dose Day 1 sample will be taken pre-dose on Day 2


 $^{\rm c}$  24 h post-dose Day 2 sample will be taken pre-dose on Day 3

Allowable windows for PK blood sampling, vital signs assessments and ECGs can be found in: Sections 13.1, 14.6, 14.7 of the study protocol.


#### **Example Taste/Palatability Questionnaire** Appendix 7

An example of the taste/palatability questionnaire can be found on the next page.

Number: DOC-101489 Version: 2.0 Status: Approved Date: 19 Dec 2022 QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan **Sponsor/Quotient Sciences Confidential Study Part: Test Product: Participant Number: Participant Initials:** Start time: (to be completed within 10 minutes of tasting) Date: **Question 1** All aspects considered (smell, sweetness, bitterness, flavour, mouthfeel/texture, grittiness, and aftertaste), how would you rate your overall liking of this product: NOTE: Tick 1 box below in blue or black pen Dislike Dislike very Dislike Dislike Like Like very Like Neither like Like slightly nor dislike extremely much moderately slightly moderately much extremely Question 2 We want to know how much you like certain aspects of the product: smell, sweetness, bitterness, flavour, mouthfeel/texture, grittiness, and aftertaste. NOTE: Tick 1 box in the row for each aspect Dislike Dislike Like N/A Dislike very Dislike Neither like Like Like very Like slightly nor dislike moderately extremely much moderately slightly much extremely Smell Sweetness **Bitterness** Flavour Mouthfeel/texture

| Aftertaste | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Entered<br>(initials): | into | eCRF | by | Date: | QC ch<br>(initials): | necked l | ру | Date: |
| | | | | | <del>_</del> | | - | |

Grittiness

Number: DOC-101489 Version: 2.0 Status: Approved Approved Date: 19 Dec 2022 QSC207031(MMV\_MMV367\_21\_01) - Reporting and Analysis Plan

# Document Approvals Approved Date: 19 Dec 2022

| Approval Task<br>Verdict: Approve | Claire Wilson, Senior Statistician<br>(Claire.Wilson@quotientsciences.com)<br>Functional / Technical Approval<br>19-Dec-2022 12:57:52 GMT+0000 |
|---|---|
| Approval Task<br>Verdict: Approve | Ewan Thomson, Manager, Statistical Programming (Ewan.Thomson@quotientsciences.com) Functional / Technical Approval 19-Dec-2022 13:36:26 GMT+0000 |
| Approval Task<br>Verdict: Approve | Nand Singh, Medical Director<br>(Nand.Singh@quotientsciences.com)<br>Functional / Technical Approval<br>19-Dec-2022 13:41:03 GMT+0000 |
| Approval Task<br>Verdict: Approve | Gemma Bell, Senior Medical Writer<br>(gemma.bell@quotientsciences.com)<br>Functional / Technical Approval<br>19-Dec-2022 15:45:47 GMT+0000 |
| Approval Task<br>Verdict: Approve | Tom Dove, Pharmacokineticist<br>(Tom.Dove@quotientsciences.com)<br>Functional / Technical Approval<br>19-Dec-2022 16:05:15 GMT+0000 |

Document Author(s): Claire Wilson